# SANOFI

#### NCT02906020

# STATISTICAL ANALYSIS PLAN

Multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of GZ/SAR402671 in patients with early-stage Parkinson's disease carrying a GBA mutation or other prespecified variant

#### GZ/SAR402671-ACT14820

| STATISTICIAN: | | |
|-----------------------------|------------------------|-----|
| Statistical Project Leader: | | |
| DATE OF ISSUE: 15-Dec-2020 | | |
| | Total number of pages: | 178 |

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of Sanofi (or any of its affiliated companies). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated to any unauthorized persons, for any reason, in any form whatsoever without the prior written consent of Sanofi (or the concerned affiliated company); 'affiliated company' means any corporation, partnership or other entity which at the date of communication or afterwards (i) controls directly or indirectly Sanofi, (ii) is directly or indirectly controlled by Sanofi, with 'control' meaning direct or indirect ownership of more than 50% of the capital stock or the voting rights in such corporation, partnership or other entity

According to template: QSD-002643 VERSION 6.0 (06-JUL-2016)

# **TABLE OF CONTENTS**

| STATIS | TICAL ANALYSIS PLAN | 1 |
|---|---|---|
| TABLE | OF CONTENTS | 2 |
| LIST OF | ABBREVIATIONS AND DEFINITION OF TERMS | 6 |
| 1 | OVERVIEW AND INVESTIGATIONAL PLAN | 8 |
| 1.1 | STUDY DESIGN AND RANDOMIZATION | 8 |
| 1.2 | OBJECTIVES | 10 |
| 1.2.1 | Part 1: Dose escalation phase | 10 |
| 1.2.1.1 | Primary objectives | |
| 1.2.1.2 | Secondary objectives | 10 |
| 1.2.1.3 | Exploratory objectives | 10 |
| 1.2.2 | Part 2: Treatment phase | 10 |
| 1.2.2.1 | Primary objectives | 10 |
| 1.2.2.2 | Secondary objectives | |
| 1.2.2.3 | Exploratory objectives | 11 |
| 1.3 | DETERMINATION OF SAMPLE SIZE | 11 |
| 1.3.1 | Part 1: Dose escalation phase | 11 |
| 1.3.2 | Part 2: Treatment phase | 11 |
| 1.4 | STUDY PLAN | 13 |
| 1.5 | MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL | 14 |
| 1.6 | STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN | 15 |
| 2 | STATISTICAL AND ANALYTICAL PROCEDURES | 17 |
| 2.1 | ANALYSIS ENDPOINTS | 17 |
| 2.1.1 | Demographic and baseline characteristics | 17 |
| 2.1.2 | Prior or concomitant medications | 18 |
| 2.1.3 | Efficacy endpoints | 19 |
| 2.1.3.1 | Primary efficacy endpoint(s) | |
| 2.1.3.2 | Secondary efficacy endpoint(s) | |
| 2.1.3.3 | Exploratory efficacy endpoint(s) | |
| 2.1.4 | Safety endpoints | |
| 2.1.4.1 | Adverse events variables | |
| 2.1.4.2 | Deaths | |
| 2.1.4.3 | Laboratory safety variables | 24 |

| 2.1.4.4 2.1.4.5 | Vital signs variables Electrocardiogram variables | 24 |
|---|---|---|
| 2.1.4.6 | Physical examination | |
| 2.1.4.7 | Neurological examination | |
| 2.1.4.8<br>2.1.4.9 | Ophthalmological examination | |
| 2.1.4.9 | Pharmacokinetic variables | |
| 2.1.6 | Pharmacodynamic/genomics endpoints | 26 |
| 2.1.7 | Quality-of-life endpoints | |
| 2.1.7 | Health economic endpoints | |
| 2.2 | DISPOSITION OF PATIENTS | |
| 2.2.1 | Randomization and drug dispensing irregularities | 30 |
| 2.3 | ANALYSIS POPULATIONS | 31 |
| 2.3.1 | Efficacy populations | 32 |
| 2.3.2 | Safety population | 32 |
| 2.3.3 | Pharmacokinetics population | 33 |
| 2.3.4 | Pharmacodynamic population | 34 |
| 2.4 | STATISTICAL METHODS | 34 |
| 2.4.1 | Demographics and baseline characteristics | 34 |
| 2.4.2 | Prior or concomitant medications | 35 |
| 2.4.3 | Extent of investigational medicinal product exposure and compliance | 36 |
| 2.4.3.1 | Extent of investigational medicinal product exposure | 36 |
| 2.4.3.2 | Compliance | 37 |
| 2.4.4 | Analyses of efficacy endpoints | 37 |
| 2.4.4.1 | Analysis of primary efficacy endpoint(s) | 38 |
| 2.4.4.2 | Analyses of secondary efficacy endpoints | |
| 2.4.4.3 | Analyses of exploratory efficacy endpoints | |
| 2.4.4.4 | Multiplicity issues | |
| 2.4.5 | Analyses of safety data | |
| 2.4.5.1 | Analyses of adverse events | |
| 2.4.5.2 | Deaths | |
| 2.4.5.3 | Analyses of laboratory variables | |
| 2.4.5.4 | Analyses of vital sign variables | |
| 2.4.5.5 | Analyses of electrocardiogram variables | |
| 2.4.5.6 | Analyses of physical examination variables | |
| 2.4.5.7 | Analyses neurological examination variables | |
| 2.4.5.8<br>2.4.5.9 | Analyses of ophthalmological examination variables Analyses of depression data | |
| 2.4.6 | Analyses of pharmacokinetic and pharmacodynamic variables | |
| 2.4.6.1 | Analyses of pharmacodynamic variables Analyses of pharmacokinetic variables | |
| 4.4.0.4 | Aliaivaea oi pilaittiacokiitelic valiabiea | ਹ0 |

| 2.4.7 | Analy | /ses of quality of life variables | 58 |
|---|---|---|---|
| 2.5 | DATA | A HANDLING CONVENTIONS | 59 |
| 2.5.1 | Gene | eral conventions | 59 |
| 2.5.2 | Data | handling conventions for secondary efficacy variables | 60 |
| 2.5.3 | Missi | ng data | 60 |
| 2.5.4 | | ows for time points | |
| 2.5.5 | | heduled visits | |
| 2.5.6 | | ng of centers for statistical analyses | |
| 2.5.7 | | stical technical issues | |
| 2.5.8 | Phari | macokinetic analysis | 65 |
| 3 | INTE | RIM ANALYSIS | 66 |
| 3.1 | INTE | RNAL DATA REVIEW PRIOR TO DOSE ESCALATION IN PART 1 | 66 |
| 3.2 | INTE | RNAL DATA REVIEW AT THE END OF PART 1 NON-JAPAN | 66 |
| 3.3 | INTE | RNAL DATA REVIEW AT THE END OF PART 1 JAPAN | 67 |
| 3.4 | ANAI | LYSIS OF PART 1 (NON-JAPAN) AND PART 1 (JAPAN) | 67 |
| 3.5 | GEN | ERAL CONVENTIONS FOR INTERIM ANALYSES | 68 |
| 4 | FINA | L ANALYSIS | 69 |
| 5 | DAT | ABASE LOCK | 70 |
| 6 | SOF | TWARE DOCUMENTATION | 71 |
| 7 | REF | ERENCES | 72 |
| 8 | LIST | OF APPENDICES | 73 |
| APPENI | OIX A | POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES (PCSA) CRITERIA | 74 |
| APPENI | DIX B | LIST OF COMMON GBA MUTATIONS | 79 |
| APPENI | OIX C | MDS-UPDRS SCORING ALGORITHM | 85 |
| APPENI | DIX D | PD-CRS SCORING ALGORITHM | 89 |
| APPENI | DIX E | MOCA SCORING ALGORITHM | 90 |
| APPENI | OIX F | BDI-II SCORING ALGORITHM | 91 |
| APPENI | OIX G | PDQ-39 SCORING ALGORITHM | 95 |
| APPENI | DIX H | EQ-5D-5L SCORING ALGORITHM | 97 |

| Statistical Analysis Plan |
|------------------------------------|
| GZ/SAR402671-ACT14820 - venglustat |

| FALLS EFFICACY SCALE SCORING ALGORITHM | 166 |
|---------------------------------------------------------------|-----|
| HEALTH RELATED PRODUCTIVITY QUESTIONNAIRE - SCORING ALGORITHM | 167 |
| ANALYSIS PROCEDURE FOR INTERNAL DATA REVIEW AND INTERIM | 172 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AE: adverse event, adverse event AESI: adverse event of special interest

ALT: alanine aminotransferase

AREDS: Age-Related Eye Disease Study

ARLNS: Age-Related Eye Disease Study (AREDS) Clinical Lens Grading System

AST: aspartate aminotransferase

ATC: anatomic or therapeutic categories

AUC: area under the plasma concentration versus time curve calculated using the

trapezoidal method over a predefined time period

BMI: body mass index

CGI: clinical global impression

CKD-EPI: chronic kidney disease epidemiology collaboration

Cmax: maximum plasma concentration observed

CSF: cerebrospinal fluid

Ctrough: plasma concentration observed just before treatment administration during

repeated dosing

DaTSCAN: ioflupane I-123 injection DaTSCAN

ECG: electrocardiogram

e-CRF: electronic case report form

EQ-5D: EuroQol Five Dimensions Questionnaire

FES: fall efficacy scale

GBA: β-glucocerebrosidase gene

GCase: glucocerebrosidase

GGT: gamma-glutamyl transferase

GL-1: glucosylceramide HLGT: high level group term HLT: high level term

HRPQ: Health-Related Productivity Questionnaire

IMP: Investigational Medicinal Product

ITT: intent-to-treat

IVRS: interactive voice response system IWRS: interactive web response system

LLT: lowest level term

LOCSII: Lens Opacity Classification System II

LP: lumbar puncture LTFU: long-term follow-up lyso-GL-1: glucosylsphingosine

MDS-UPDRS: Movement Disorder Society-Unified Parkinson's Disease Rating Scale

MedDRA: Medical Dictionary for Regulatory Activities

MoCA: Montreal Cognitive Assessment MRI: magnetic resonance imaging

Statistical Analysis Plan GZ/SAR402671-ACT14820 - venglustat 15-Dec-2020 Version number: 2

NFL: neurofilament light chain

PCSA: potentially clinically significant abnormality

PD: Parkinson Disease

PD-CRS: Parkinson's Disease-Cognitive Rating Scale PDQ-39: Parkinson's Disease Questionnaire – 39 PGIC: Patient Global Impression of Change

PK: pharmacokinetics PT: preferred term

SAE: serious adverse event SAP: statistical analysis plan SD: standard deviation

SDMT: Symbol Digit Modalities Test SMQ: Standardized MedDRA Query

SOC: system organ class

TEAE: treatment-emergent adverse event

TMT-A: Trail Making Tests Part A
TMT-B: Trail Making Tests Part B
ULN: upper limit of normal range

WHO-DD: World Health Organization-Drug Dictionary

## 1 OVERVIEW AND INVESTIGATIONAL PLAN

This Statistical Analysis Plan (SAP) is intended to be a detailed description of the definitions and statistical techniques to be used for the analyses of data collected in ACT14820 study.

The first, second and third versions of this SAP covered the analyses of data collected during Part 1 of the study, and were finalized prior to the analysis of Part 1 non-Japan and Part 1 Japan data, respectively. The forth version covered the analyses of data collected during Part 2 of the study, including the 52-week blinded treatment period (Period 2) and the 104-week duration long-term follow-up (LTFU) period (Period 3).

This SAP was amended following recommendations from the FDA to exclude data collected after treatment discontinuation from the primary analysis and use them in sensitivity analyses.

This amended SAP was finalized prior to the final analysis of Part 2 study to ensure the credibility of the study results by pre-specifying the statistical methods for analyses before unblinding of treatment assignments.

Details of amendments of the SAP are described in Table 2.

#### 1.1 STUDY DESIGN AND RANDOMIZATION

This is a two-part, multicenter, multiple-country, randomized, double-blinded, placebo-controlled study in early-stage Parkinson Disease (PD) patients carrying a GBA mutation. The study will be divided into 2 consecutive parts. Part 1 will be a randomized, double-blinded, placebo-controlled dose escalation study, utilizing a sequential cohort design. Part 1 will allow selection of the dose of GZ/SAR402671 for Part 2, a randomized, double-blind, placebo-controlled, 2-arm study of the efficacy and safety of GZ/SAR402671. Part 1 will be conducted only in selected sites (approximately 20 sites [including 4 Japanese sites]); Part 2 will be conducted at multiple sites (approximately 50). Part 2 will start after the appropriate dose for Part 2 is selected in Part 1.

In Part 1, during the screening/baseline period, from Day -60 to Day -1, patients will provide informed consent and undergo screening assessments to determine trial eligibility and undergo baseline measurements. If all eligibility criteria are met, patients will enter the trial. Part 1 will determine the safety and tolerability of GZ/SAR402671 at 4, 8, and 15 mg in early-stage PD patients carrying a GBA mutation by using a dose escalation scheme (4 weeks to assess safety and tolerability of dose and a minimum of an additional 4 weeks to further assess safety and tolerability and any potential changes in other exploratory endpoints in each dose cohort). There will be 3 sequential cohorts that will be placebo-controlled:

- Cohort 1: 4 patients (or 3 patients in Japan) on GZ/SAR402671 4 mg and 1 patient on placebo
- Cohort 2: 4 patients (or 3 patients in Japan) on GZ/SAR402671 8 mg and 1 patient on placebo

• Cohort 3: 4 patients (or 3 patients in Japan) on GZ/SAR402671 15 mg and 1 patient on placebo

No additional dose escalation of GZ/SAR402671 will occur above the highest proposed dose of 15 mg. All patients must complete the first 4 week course of therapy with subsequent blinded data review by an internal review committee whose purpose is to review blinded data (such as safety, tolerability, and/or relevant clinical endpoints), demonstrating safety/tolerability before dose escalation to the next higher level can occur. Patients will continue to be dosed daily and will be followed every 4 weeks until the completion of Part 1, allowing for additional safety and other exploratory endpoints to be collected. Each cohort will have a 4:1 randomization ratio, and the total sample size will be approximately 15 patients (including 12 on GZ/SAR402671 and 3 on placebo). In Japan, each cohort will have a 3:1 ratio, and the total sample size will be approximately 12 Japanese patients (including 9 on GZ/SAR402671 and 3 on placebo). Therefore, the total sample size in Part 1 will be approximately 27 patients.

At the end of 4 weeks of treatment during the dose escalation part, patients in each cohort will have a lumbar puncture (LP); CSF exposure of GZ/SAR402671 will be measured at 2 time points in Part 1: at pretreatment and Week 4. If there is no CSF exposure at the highest dose level, the study will be stopped.

In Part 2, the GZ/SAR402671 dose will be the highest dose determined to be safe and well tolerated in Part 1. Moreover, CSF exposure must be known. If there is no CSF exposure of GZ/SAR402671, then that dose will not be used in Part 2.

If patients from Part 1 continue to meet eligibility requirements, and are willing to continue in the study, they may enroll in Part 2, but re-randomization will be required; furthermore, they will have to sign another informed consent form. All screening assessments will need to be repeated, except for the genetic screening, magnetic resonance imaging (MRI), LP, and ioflupane I-123 injection DaTSCAN (DaTSCAN), to confirm eligibility of patients from Part 1 to enroll in Part 2.

In Part 2, eligible patients will be stratified based on use of levodopa/PD medication (yes/no), cognitive function (Montreal Cognitive Assessment [MoCA]) score <26 [yes/no]) and severe GBA mutation (yes/no). Patients will be randomized in a 1:1 ratio to receive GZ/SAR402671 or placebo for 52 weeks.

Part 2 will include 4 main periods: the up to 60-day screening period (Period 1), the 52-week blinded treatment period (Period 2), the 104-week duration long-term follow-up (LTFU) period (Period 3), and the 6-week post treatment observation period (Period 4).

#### 1.2 OBJECTIVES

#### 1.2.1 Part 1: Dose escalation phase

## 1.2.1.1 Primary objectives

To determine the safety and tolerability of 4, 8, and 15 mg of GZ/SAR402671, as compared to placebo, when administered orally daily for 4 weeks in early-stage PD patients carrying a GBA mutation or other prespecified sequence variants (from now on both mutation types are referred to as 'GBA mutation'). This will allow selection of the dose for the second part of this study (this does not apply to Japanese patients).

#### 1.2.1.2 Secondary objectives

To assess the PK profile of daily oral dosing of GZ/SAR402671 in plasma when administered at doses of 4, 8, or 15 mg over a 4-week period in early-stage PD patients carrying a GBA mutation.

To assess the exposure of GZ/SAR402671 in CSF when administered at doses of 4, 8, or 15 mg over a 4-week period in early-stage PD patients carrying a GBA mutation.

## 1.2.1.3 Exploratory objectives

To assess the pharmacodynamic response of daily oral dosing of GZ/SAR402671 in plasma and CSF when administered at doses of 4, 8, or 15 mg over a 4-week period, as measured by GL-1 in early-stage PD patients carrying a GBA mutation.

To explore the effect of GZ/SAR402671 on scores from selected scales and questionnaires which will be used in this study over an 8 week period in early-stage PD patients carrying a GBA mutation.

#### 1.2.2 Part 2: Treatment phase

#### 1.2.2.1 Primary objectives

To determine the efficacy of GZ/SAR402671 in patients with early-stage PD carrying a GBA mutation when administered orally daily at the dose selected in Part 1, over a 52-week period, as compared to placebo.

## 1.2.2.2 Secondary objectives

To demonstrate the overall safety and tolerability of GZ/SAR402671 administered orally daily for 52 weeks in early-stage PD patients carrying a GBA mutation as compared to placebo.

To assess the pharmacodynamic response to daily oral dosing of GZ/SAR402671 in plasma and CSF as measured by GL-1 in early-stage PD patients carrying a GBA mutation over a 52-week period.

## 1.2.2.3 Exploratory objectives

To explore the effect of GZ/SAR402671 on scores from selected scales and questionnaires which will be used in this study. Of note, for patients receiving levodopa or other PD medication, assessment of scales and questionnaires will be performed during the OFF state (ie, no PD medication may be taken for at least 12 hours prior to the efficacy assessments) except for the Hoehn & Yahr (H&Y) scale which will be completed in "ON" state only at baseline visit (see inclusion criteria I 05).

To assess the effect of GZ/SAR402671 on neurologic functional status via functional neuroimaging over a 52-week period.

To assess the PK profile of GZ/SAR402671 in plasma and CSF of early-stage PD patients carrying a GBA mutation.

To evaluate the pharmacodynamic response to GZ/SAR402671 in plasma and CSF as measured by glucosylsphingosine (lyso-GL-1) in early-stage PD patients carrying a GBA mutation.

To explore the effect of GZ/SAR402671 on CSF biomarkers related to PD or neurodegeneration, including total  $\alpha$ -synuclein ( $\alpha$ -Syn), neurofilament light chain (NFL), tau, phospho-tau, as well as beta-amyloid (1-40 and 1-42).

#### 1.3 DETERMINATION OF SAMPLE SIZE

#### 1.3.1 Part 1: Dose escalation phase

As Part 1 is an exploratory, dose-escalation study, the sample size is not based on the statistical power calculation. Each cohort (for non-Japanese patients only) will have a 4:1 randomization ratio, and the total sample size will be approximately 15 patients (including 12 on GZ/SAR402671 and 3 on placebo).

For Japanese patients only, each cohort will have a 3:1 randomization ratio, and the total sample size will be approximately 12 Japanese patients (including 9 on GZ/SAR402671 and 3 on placebo). This sample size in Japanese Part 1 is considered based upon empirical and feasibility considerations.

Therefore, the total sample size in Part 1 will be approximately 27 patients.

Patients who do not complete a minimum number of scheduled doses of study drug in Part 1 and withdraw for reasons other than safety may be replaced.

#### 1.3.2 Part 2: Treatment phase

Approximately 216 PD patients carrying a GBA mutation in total will be randomized in a 1:1 ratio to the GZ/SAR402671 or placebo groups. A sample size of 108 patients for the GZ/SAR402671 group and 108 for the placebo group provides at least 80% power to detect a 4.06

points improvement compared to the placebo mean change in MDS-UPDRS Parts II+III score over 52 weeks. This sample size calculation assumes a 2-sided alpha = 0.05, a standard deviation for the change from baseline to Week 52 in MDS-UPDRS Part II+III of 10.01 points (estimated from the Parkinson's Progression Markers Initiative [PPMI] database), and allows for an approximate 10% early terminations/unevaluable patients.

A previous study showed that a 3.25 points difference on MDS-UPDRS Part III represent the minimal clinically important difference (MCID) for detecting an improvement. It was estimated from the PPMI database that the standard deviation for change from baseline to Week 52 in MDS-UPDRS Part III was 8.01 points; therefore the MCID of 3.25 points would represent an effect size of 0.406. Since no study evaluated the MCID for MDS-UPDRS Part II+III, the same effect size of 0.406 was assumed, resulting in an estimated MCID of 4.06 points, using the standard deviation of 10.01 for change from baseline to Week 52 in MDS-UPDRS Part II+III also estimated from the PPMI database.

Of note, the approximate 27 (12 Japanese and 15 non-Japanese) early-stage PD patients carrying a GBA mutation from Part 1 may be re-randomized and participate in all of the assessments in Part 2 of this study; however, they will not contribute to the primary efficacy, safety, PK and pharmacodynamics analyses, and will be described separately.

Calculations were made using nQuery 7.0 Advisor software.

#### 1.4 STUDY PLAN

The following figures present the graphical study design:

safety assessment **Cohort 1** to follow Placebo PO, qd Screening N = 160 days max safety assessment to follow GZ/SAR402671 4 mg, PO, qd enrollment pause N = 4safety assessment Cohort 2 to follow Placebo R PO, qd Screening N = 1 60 days max safety assessment BASELINE: to follow CSF Safety Imaging Efficacy GZ/SAR402671 8 mg, PO, qd N = 4END of 4 WEEKS: safety assessment CSF Safety MDS-UPDRS Cohort 3 to follow Placebo END of every 4 WEEKS R PO, qd until Part 1 completion\*: Screening Safety MDS-UPDRS 60 days max safety assessment : daily dosing of to follow placebo or GZ/SAR402671 will continue until Part 1 completion; max 36 weeks GZ/SAR402671 of study medication exposure 15 mg, PO, qd N = 4

Figure 1 - Graphical study design for Part 1

Abbreviations: CSF: cerebrospinal fluid; LP: lumbar puncture; max: maximum; MDS-UPDRS: Movement Disorder Society-Unified Parkinson's Disease Rating Scale; N: number of subjects; PO: oral; qd: once daily; R: randomization.

<sup>\*\*</sup> The LP may be done during the screening period within 14 days prior to randomization (Day -14 to Day -1) or on the day of randomization (Day 1 predose). Only 1 sample will be collected, during screening or at Day 1.

**Blinded Treatment Period** Long-Term Follow-Up Phase GZ/SAR402671 PO, qd N = 108Period 1 GZ/SAR402671\* PO, qd Screening Clinic Visits every 60 days max 6 months Placebo PO, qd N = 10852 W 13 W 26 W 39 W 156 W 162W End of Period 2 Baseline\* End of Period 3 Visit/ Period 4 Efficacy CSF (all) Efficacy CSF (all) Efficacy Imaging Imaging Efficacy Efficacy

Figure 2 - Graphical study design for Part 2

Abbreviations: R: randomization; W: weeks; max: maximum; CSF: cerebrospinal fluid; pts: patients; LP: lumbar puncture.

- The LP may be done during the screening period within 14 days prior to randomization (Day -14 to Day -1) or on the day of randomization (Day 1 pre-dose). Only one sample will be collected, during screening or at Day 1.
- The dose of GZ/SAR402671 will be determined in Part 1.

Abbreviations: CSF: cerebrospinal fluid; LP: lumbar puncture; max: maximum; N: number of patients; PO: oral; qd: once daily; R = randomized; W = weeks.

Day 1; LP at baseline will not be required to confirm eligibility of patients from Part 1 to enroll in Part 2.

#### 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL

This section summarizes major changes to the protocol statistical section with emphasis on changes after study start (after the first patient was enrolled).

The protocol history table below gives the timing, rationale, and key details of major changes to the protocol statistical section.

<sup>\*</sup> The LP may be done during the screening period within 14 days prior to randomization (Day -14 to Day -1) or on the day of randomization (Day 1 predose). Only 1 sample will be collected, during screening or at

<sup>\*\*</sup> The dose of GZ/SAR402671 will be determined in Part 1.

Table 1 - Protocol amendment statistical changes

| Amendment<br>Number | Rationale | Description of statistical changes |
|---|---|---|
| 1 | Inclusion of a Japanese cohort | Increase in sample size of Part 1 (12 additional Japanese patients) |
| | | Definition of specific Japanese populations for efficacy, safety, PK and pharmacodynamics analyses. |
| | | Separate analyses for Japanese and non-Japanese patients |
| Health Authorities in the United Part 2 will not be included in Part 2 States and Japan Part 2 safety, pharmacokinetics and phart | | Clarification that patients from Part 1 who are re-randomized in Part 2 will not be included in Part 2 analyses (for efficacy, safety, pharmacokinetics and pharmacodynamic analyses). These data will be described separately. |
| 4 | Removal of interim analysis | Interim analysis planned for administrative purposes that are no longer required by the Sponsor. |

## 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

The statistical analysis plan history table below gives the timing, rationale, and key details for major changes to the statistical analysis features in the statistical analysis plan.

15-Dec-2020 Version number: 2

Table 2 - Statistical analysis plan changes

| SAP<br>version<br>number | Date<br>approved | Rationale | Description of statistical changes |
|---|---|---|---|
| 1 | 18-Dec-2017 | Initial version | - |
| 1 | 25-Apr-2018 | Specification of an analysis of Part 1 data after completion of Part 1 (non-Japan) | An analysis of Part 1 (non-Japan) data will be performed when all non-Japanese patients have completed Part 1, and after a two-step database lock (see Section 3.4 and Section 5) |
| 1 30-Nov-2018 | 30-Nov-2018 | Specification of an analysis of Part 1 data after completion of Part 1 (Japan) | An analysis of Part 1 (Japan) data will be performed when all Japanese patients have completed Part 1, and after a two-step database lock (see Section 3.4 and Section 5) |
| | | | Update of the EQ-5D-5L scoring algorithm (see Appendix H) |
| | | Inclusion of the procedure for internal data review as appendix of the SAP (Appendix K) | |
| 1 | 22-Jul-2020 | Specification of analyses of Part 2 data | Description of analyses planned for Part 2 of the study. |
| | Comment from FDA on version 1, received on 16-Oct-2020 and 17-Nov- | Change in primary and secondary estimand (Section 2.4.4.1) | |
| | | 2020, to exclude data collected after treatment discontinuation from the primary analysis and use them in sensitivity analyses. | Exclusion of data collected after premature treatment discontinuation from the primary efficacy analysis (Section 2.4.4.1) |
| | | | Addition of a sensitivity analysis including data collected after treatment discontinuation (Section 2.4.4.1) |
| | Exclusion of data after premature treatment discontinuation from analysis of secondary efficacy endpoints (Section 2.4.4.2) and exploratory efficacy endpoints (Section 2.4.4.3) | | |
| | | Delayed visits due to COVID-19 pandemic situation | Analysis window of Week 52 visit extended to D570 (Section 2.5.4, Table 6) |

# 2 STATISTICAL AND ANALYTICAL PROCEDURES

#### 2.1 ANALYSIS ENDPOINTS

## 2.1.1 Demographic and baseline characteristics

The baseline value is defined as the last available value obtained before or equal to the date and time of the first double-blind Investigation Medicinal Product (IMP) administration. In case of missing time of the first double-blind IMP administration and/or time of assessment, the baseline value is defined as the last available value obtained before or equal to the date of the first double-blind IMP. For patients randomized and not treated, the baseline value is defined as the last available value obtained before or equal to the date and time of randomization.

All baseline safety and efficacy parameters are presented along with the on-treatment summary statistics in the safety and efficacy sections (Section 2.4.5 and Section 2.4.4).

## Demographic characteristics

Demographic variables include:

- Gender (Male, Female)
- Age in years (quantitative and categorical variable : <45, [45 65[, [65 75[ and ≥75 years),</li>
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or other Pacific Island, other)
- Ethnicity (Hispanic, non-Hispanic)
- Weight in kilograms (quantitative and categorical variable:  $<50, \ge 50$  and  $<100, \ge 100$ )
- Body mass index (BMI) in kg/m<sup>2</sup> (quantitative and categorical variable:  $<30, \ge 30$ )

#### Parkinson's disease history

Parkinson's disease history include:

- Time since onset of symptoms (in years)
- Time since diagnosis (in years)
- Predominance of symptom at onset (Tremor, Rigidity / Bradykinesia)
- Family history of Parkinson's disease (yes, no)

Any technical details related to computation, dates, and imputation for missing dates are described in Section 2.5.3.

#### **GBA** mutations

GBA mutations will be categorized as severe GBA mutation or other GBA mutation. The list of most common mutations is provided in Appendix B.

## Medical or surgical history

All medical or surgical history information in the e-CRF will be coded using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Sanofi at the time of database lock.

#### Alcohol Habits

Alcohol habits include:

- Frequency of alcoholic drinks in the last 12 months (Never/Occasional/At least monthly/At least weekly/At least daily)
- Number of standard drinks (1 or 2/Greater than 2, where standard drink means 1 pint/bottle of beer, 1 glass of wine, 1 shot of hard liquor...) per day when drinking alcohol

#### 2.1.2 Prior or concomitant medications

All Parkinson's disease medications that the subject has taken within 3 months prior to screening and any Parkinson's disease medications taken during the study are to be reported in the case report form pages. Other medications that the subject has taken during the study are also to be reported.

All medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD) using the version currently in effect at Sanofi at the time of database lock.

- Prior medications are those medications which the patient used prior to the first doubleblind IMP administration. Prior medications could be discontinued before the first administration of IMP or could be ongoing during the treatment phase
- Concomitant medications are any treatments received by the patient concomitantly with the IMP, ie, from the first IMP intake to the day of last IMP intake + 1 day. A given medication can be classified both as a prior medication and as a concomitant medication.
- Posttreatment medications are those the patients took in the period running from the last IMP intake + 2 days up to the end of follow-up phase

Any technical details related to computation, dates, imputation for missing dates are described in Section 2.5.3.

#### 2.1.3 Efficacy endpoints

#### 2.1.3.1 Primary efficacy endpoint(s)

# Part 1: Dose escalation phase

The primary endpoint in Part 1 is safety of each dose cohort. The following additional endpoints will be evaluated:

- Change in MDS-UPDRS PART II+III score, performed during the OFF state, from baseline to 4 weeks
- Change in MDS-UPDRS PART II+III score, performed during the OFF state, from baseline to 8 weeks
- Change in MDS-UPDRS PART I+II+III, performed during the OFF state, from baseline to 4 weeks
- Change in MDS-UPDRS PART I+II+III, performed during the OFF state, from baseline to 8 weeks

The MDS-UPDRS will be performed by the certified blinded rater for all patients at screening, at Day 1, at Week 4 (Day 1), Week 8, and every 4 weeks thereafter, until completion. No PD medication may be taken for at least 12 hours prior to efficacy assessments.

## Part 2: Treatment phase

The primary endpoint is the change in MDS-UPDRS (PART II+III score), performed during the OFF state, from baseline to Week 52. Of note, Part IA, IB, and II of the MDS-UPDRS do not have separate ON or OFF ratings. The OFF definition provided in this protocol is to ensure uniformity among raters and the score sheets should document the OFF status associated with the Part III assessment.

#### 2.1.3.2 Secondary efficacy endpoint(s)

#### Part 1: Dose escalation phase

Not applicable.

# Part 2: Treatment phase

- Change in PD-CRS (total score) from baseline to Week 52.
- Change in MDS-UPDRS PART I+II+III, performed during the OFF state, from baseline to Week 52.
- Change in H&Y stage from baseline to Week 52.

## 2.1.3.3 Exploratory efficacy endpoint(s)

#### Part 1: Dose escalation phase

The following endpoints will be analyzed for Part 1:

- Change in Montreal cognitive assessment (MoCA) score, from baseline to 8 weeks
- Change in oral Symbol Digit Modalities Test (SDMT) score, from baseline to 8 weeks
- Change in Trail Making Tests Part A (TMT-A), Trail Making Tests Part B (TMT-B) and difference between TMT-B minus TMT-A score, from baseline to 8 weeks
- Clinical global impression (CGI) scale, including illness severity (CGIS), global improvement of change (CGIC), and therapeutic response at 8 weeks
- Patient global impression of change (PGIC) at 8 weeks

# Part 2: Treatment phase

The following exploratory efficacy endpoints will be analyzed for Part 2:

- Change from baseline to Week 26 in biomarkers GL-1 and lyso-GL-1 levels in plasma (percent and absolute change).
- Change from baseline to Week 52 in DaTSCAN assessment scores (percent and absolute change). The Striatal Binding Ratio (SBR) will be calculated for the following brain regions, using the occipital lobe as the reference region:
  - Caudate nucleus: left medial, right medial, left, right
  - Putamen: left medial, right medial, left anterior, right anterior, left, right
  - Corpus striatum: left, right, total
- Time to initiation of levodopa or other PD therapy (for patients not on levodopa/other PD therapy at baseline) or to increased (intensification) dose of levodopa/other PD therapy (for patients on levodopa/other PD therapy at baseline). Initiation or intensification of PD medication will be defined as any of the two following criteria fulfilled:
  - Increase of the dose of a PD medication by at least 50% compared to the dose received at baseline, with maintenance of an increased dose until the end of the 52-week blinded treatment period
  - Initiation of a PD medication not received at baseline, with maintenance of the new PD medication until the end of the 52-week blinded treatment period.

Any technical details are described in Section 2.5.2

• Time to Reduction of levodopa/PD medication (for patients on levodopa/other PD medication at baseline). Reduction of PD medication will be defined as any of the two following criteria fulfilled:

- Decrease of the dose of a PD medication by at least 50% compared to the dose received at baseline, with maintenance of a decreased dose until the end of the 52-week blinded treatment period
- Stop of a PD medication received at baseline, with no re-initiation of the PD medication until the end of the 52-week blinded treatment period.

In addition, if a patient reduced a PD medication but initiated or intensified another PD medication, then the patient will not be considered as having reduced his/her PD therapy. Any technical details are described in Section 2.5.2.

- Change from baseline to Week 52 in GL-1, lyso-GL-1 levels in CSF and plasma (percent and absolute change).
- Change from baseline to Week 52 in GCase activity in CSF and dried blood spot (percent and absolute change).
- Change from baseline to Week 52 in biomarkers related to neurodegeneration in plasma and/or in CSF, such as α -Syn, NFL, tau, phospho-tau, as well as beta amyloid (1-40, and 1-42) (percent and absolute change).
- Change from baseline to Week 52 in MDS-UPDRS (total score), performed during the OFF state.
- Change from baseline to Week 52 in MDS-UPDRS individual subscores (Parts I, II, III, and IV).
- Change from baseline to Week 52 in PD-CRS subscores (the subcortical scale [items 1, 3, 4, 5, 7, 8, 9]) and the cortical scale (items 2 and 6).
- Change from baseline to Week 52 in MoCA score.
- Change from baseline to Week 52 in Symbol Digit Modalities Test (SDMT) oral score.
- Change from baseline to Week 52 in Trail Making Test A (TMT-A) and Trail Making Test B (TMT-B) score including the change in the difference between TMT-B minus TMT-A score.
- Change from baseline to Week 52 in Clinical Global Impression (CGI) scale subscores (such as CGI of Improvement).
- Change from baseline to Week 52 in Falls Efficacy Scale (FES)

A description of the calculation of the score for each scale is available in appendices.

The data collected during the study will be used to develop a Parkinson's disease progression model in early-stage PD patients carrying a GBA mutation. This model will be described in a separate document.

## 2.1.4 Safety endpoints

## Observation period

The observation period will be divided into 4 periods:

- The pre-treatment period is defined as the time from the signed informed consent date up to the first double-blind IMP administration
- The on-treatment period is defined as the time from the first administration of the IMP to the last administration of the IMP + 1 day, including any temporary treatment discontinuation period, if any
- The residual treatment period is defined as the time from the last administration of the IMP + 2 days to the last IMP administration + 6 weeks
  - The treatment-emergent adverse event (TEAE) period will include both the ontreatment and the residual treatment periods
- The posttreatment period is defined as the period of time starting the day after the residual treatment period

## Part 1: Dose escalation phase

Safety endpoints will be assessed by:

- Physical examination
- Neurological examination
- Clinical laboratory evaluations, including hematology, biochemistry, and urinalysis
- Vital signs
- Assessment of adverse events (AEs) and concomitant medication
- Ophthalmological examination. Visual acuity and lens evaluation will be performed according to the Lens Opacity Classification System II (LOCSII) for monitoring potential cataract development and worsening of pre-existing cataract.
- ECG

## Part 2: Treatment phase

Safety endpoints will be assessed by:

- Physical examination.
- Neurological examination.
- Clinical laboratory evaluations, including hematology, biochemistry, and urinalysis.
- Vital signs.
- Assessment of adverse events (AEs) and concomitant medication.

- Ophthalmological examination. Visual acuity and lens evaluation will be performed according to the Lens Opacity Classification System II (LOCSII) for monitoring potential cataract development and worsening of pre-existing cataract.
- ECG

#### 2.1.4.1 Adverse events variables

#### Adverse event observation period

- Pretreatment adverse events are adverse events that developed or worsened or became serious from the signed informed consent date up to first administration of IMP
- TEAEs are adverse events that developed or worsened or became serious during the TEAE period (as defined in Section 2.1.4)
- Posttreatment adverse events are adverse events that developed or worsened or became serious during the posttreatment period

All adverse events (including serious adverse events and adverse events with prespecified monitoring) will be coded to a lower-level term (LLT), preferred term (PT), high-level term (HLT), high-level group term (HLGT), and associated primary system organ class (SOC) using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Sanofi at the time of database lock.

Adverse events (including serious adverse events and adverse events of special interest) will be recorded from the time of signed informed consent until the end of the study.

Adverse events of special interest (AESIs) include the following terms (their complete descriptions are provided in the protocol):

- New or worsening lens opacities and cataracts
- Pregnancy occurring in a female patient entered in the clinical trial or in a female partner
  of a male patient entered in the clinical trial will be recorded as an AESI with immediate
  notification in all cases
- Increase in aminotransferase (ALT)
- Symptomatic overdose (serious or non-serious) with IMP: An overdose (accidental or intentional) with the IMP is an event suspected by the Investigator or spontaneously notified by the patient (not based on systematic pills count) and defined as at least twice the intended dose within the intended therapeutic interval, adjusted according to the tested drug

#### 2.1.4.2 Deaths

The deaths observation periods are per the observation periods defined above.

- Death on-study: deaths occurring during the on-study observation period
- Death occurring during the TEAE period (as defined in Section 2.1.4)
- Death occurring during the post-treatment period

• Death post-study: deaths occurring after the end of the study (including all deaths occurring after the patients' 6-week follow-up visit, until database lock.)

#### 2.1.4.3 Laboratory safety variables

Clinical laboratory data consists of blood analysis, including hematology, biochemistry, and urinalysis. Clinical laboratory values after conversion will be analyzed into standard international units and international units will be used in all listings and tables.

All laboratory data listed in this section, except for CSF cell count, will be measured at a central laboratory.

The following laboratory safety variables will be analyzed:

- Hematology: red blood cell count, hematocrit, hemoglobin, white blood cell count with differential count (neutrophils, eosinophils, basophils, monocytes, and lymphocytes), platelets, prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR)
- Biochemistry:
  - Plasma/serum electrolytes: sodium, potassium, chloride, calcium, bicarbonate
  - Liver function: ALT, AST, gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), total and conjugated bilirubin
  - Renal function: urea, serum creatinine, eGFR (based on CKD-EPI formula)
  - Metabolism: glucose, albumin, total proteins

Technical formulas are described in Section 2.5.1.

#### 2.1.4.4 Vital signs variables

Vital signs include: temperature, systolic and diastolic blood pressure (mmHg), heart rate (beats per minute) and respiratory rate (breaths/min).

## 2.1.4.5 Electrocardiogram variables

Electrocardiogram (ECG) parameters include Heart rate (bpm), PR interval (ms), QRS duration (ms), QTc Bazett duration (ms), QTc Fridericia duration (ms). All ECG recordings will be centrally read by independent experts.

#### 2.1.4.6 Physical examination

Each physical examination will include the following physical observations/measurements: general appearance; heart, skin, respiratory auscultation; head, eyes, ears, nose, and throat, extremities/joints, and abdomen.

Physical examination findings will be assessed as normal or abnormal.

#### 2.1.4.7 Neurological examination

Each neurological examination will include, but not be limited to, assessments of the patient's mental status, cranial nerves, motor system (including muscle atrophy, tone and power), deep tendon reflex, sensation, and cerebellar function.

#### 2.1.4.8 Ophthalmological examination

The full ophthalmological examination will include visual acuity, slit-lamp examination and examination of the cornea, lens, and retina. The examination should include pupil dilation and evaluation of the lens according to the LOCSII. This evaluation should be accompanied by pictures of the lens for evaluation by the examining ophthalmologist. Photos of the lens will be reviewed/assessed by a central reader. Ophthalmological evaluation by the central reader will be assessed according to the Age-Related Eye Disease Study (AREDS) Clinical Lens Grading System (ARLNS) (1).

#### 2.1.4.9 Depression

Depression will be monitored during the study using the Beck depression inventory, second edition (BDI-II). The BDI-II is a 21-question, multiple-choice, self-report inventory. It is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and disinterest in sex.

#### 2.1.5 Pharmacokinetic variables

#### Part 1: Dose escalation phase

Plasma PK parameters in Part 1 will include:

- Day 1 (single dose administration): maximum plasma concentration observed (Cmax), time to reach C<sub>max</sub> (t<sub>max</sub>), and area under the plasma concentration versus time curve calculated using the trapezoidal method over a predefined time period (from time t= 0 to 24 hours [AUC<sub>0-24</sub>], and from t= 0 to 48 hours [AUC<sub>0-48</sub>])
- Week 2: plasma concentration observed just before treatment administration during repeated dosing (C<sub>trough</sub>)
- Week 4: C<sub>trough</sub>, C<sub>max</sub>, t<sub>max</sub>, AUC<sub>0-24</sub>, and apparent total body clearance of a drug at steady state after oral administration (CL<sub>ss</sub>/F; calculated using the following equation: CL<sub>ss</sub>/F = Dose/AUC<sub>τ</sub>, where τ is the dosing interval)
- Week 8: Ctrough

Cerebrospinal fluid PK parameters in Part 1 will include:

- Day -14 to Day 1: predose concentration
- Week 4: Concentration at any time within 2 to 4 hours after administration of GZ/SAR402671

## Part 2: Treatment phase

Plasma PK parameters in Part 2 will include:

- Day 1 (single dose administration): C<sub>max</sub>, t<sub>max</sub>, AUC<sub>0-24</sub>
- Week 2: Ctrough
- Week 26:
  - Ctrough
  - Concentration at any time within 2 to 4 hours after administration of GZ/SAR402671 on visit day.
- Week 52:
  - C<sub>trough</sub>
  - Concentration at any time within 2 to 4 hours after administration of GZ/SAR402671 on visit day.

Cerebrospinal fluid PK parameters include:

- Day -14 to Day 1: pre-dose concentration
- Week 52 (all patients): concentration at any time within 2 to 4 hours after administration of GZ/SAR402671 on visit day.

Depending on the timing of plasma and CSF PK sample collection verses the previous dose, Cmax and Ctrough will be defined as follows:

Cmax: venglustat concentration sample taken between 2-5 hr after previous dose

Ctrough: venglustat concentrations sample taken 24 hr after previous dose or just prior to the next dose

Exploratory GZ/SAR402671 metabolite PK profiling and/or metabolite exposure analysis may be performed on plasma and CSF samples collected during Part 1 and Part 2 of the study.

## 2.1.6 Pharmacodynamic/genomics endpoints

#### Part 1: Dose escalation phase

The following biomarkers in blood, dried blood spot and/or cerebrospinal fluid may be analyzed in samples collected during the study, at the discretion of the Sponsor:

# Blood markers (plasma or serum)

- Glucosylceramide (GL-1)
- Glucosylsphingosine (lyso-GL-1)
- Neurofilament light chain (NFL)
- Total alpha-synuclein (α-Syn)

• Amyloid –beta 1-40, and Amyloid –beta 1-42

Other markers may also be assessed.

## Dried blood spot

• Glucocerebrosidase activity (GCase)

Other markers may also be assessed.

# Cerebrospinal Fluid

- Glucosylceramide (GL-1)
- Glucosylsphingosine (lyso-GL-1)
- Neurofilament light chain (NFL)
- Glucocerebrosidase activity (GCase)
- Total alpha-synuclein (α-Syn)
- Tau and phospho-Tau181
- Amyloid –beta 1-40, and Amyloid –beta 1-42

Other markers may also be assessed.

## Part 2: Treatment phase

## Blood markers (plasma or serum)

- Glucosylceramide (GL-1)
- Glucosylsphingosine (lyso-GL-1)
- Neurofilament light chain (NFL)
- Total alpha-synuclein (α-Syn)
- Amyloid –beta 1-40, and Amyloid –beta 1-42

Other markers may also be assessed.

## Dried blood spot

• Glucocerebrosidase activity (GCase)

Other markers may also be assessed.

## Cerebrospinal Fluid

- Glucosylceramide (GL-1)
- Glucosylsphingosine (lyso-GL-1)
- Neurofilament light chain (NFL)

- Glucocerebrosidase activity (GCase)
- Total alpha-synuclein (α-Syn)
- Tau and phospho-Tau181
- Amyloid –beta 1-40, and Amyloid –beta 1-42

Other markers may also be assessed.

## 2.1.7 Quality-of-life endpoints

## Part 1: Dose escalation phase

The following quality of life endpoints will be analyzed for Part 1:

- Change in Parkinson's disease questionnaire 39 (PDQ-39) score, from baseline to 8 weeks, including the following scores:
  - Mobility
  - Activities of daily living
  - Emotional well-being
  - Stigma
  - Social support
  - Cognition
  - Communication
  - Bodily discomfort
  - PDQ-39 single index (PDQ-39-SI)
- Change in EuroQol five dimensions (EQ-5D-5L) score from baseline to 8 weeks

# Part 2: Treatment phase

The following quality of life endpoints will be analyzed for Part 2:

- Change in Parkinson's disease questionnaire 39 (PDQ-39) score, from baseline to 52 weeks, including the following scores:
  - Mobility;
  - Activities of daily living;
  - Emotional well-being;
  - Stigma;
  - Social support;
  - Cognition;
  - Communication;
  - Bodily discomfort;

- PDQ-39 single index (PDQ-39-SI).
- Change in EuroQol five dimensions (EQ-5D-5L) score from baseline to 52 weeks

A description of the calculation of the score for each scale is available in appendices.

### 2.1.8 Health economic endpoints

#### Part 1: Dose escalation phase

The following health economic endpoints will be analyzed for Part 1:

- Change in Health-related productivity questionnaire (HRPQ) score, from baseline to 8 weeks, including:
  - Hours of lost work due to absenteeism in (a) workplace and (b) household
  - Hours of lost work due to presenteeism in (a) workplace and (b) household
  - Total [absenteeism + presenteeism] hours of lost work in (a) workplace and (b) household
  - % of scheduled work lost due to absenteeism, presenteeism, and total productivity loss in (a) workplace and (b) household

## Part 2: Treatment phase

The following health economic endpoints will be analyzed for Part 2:

- Change in Health-related productivity questionnaire (HRPQ) score, from baseline to 52 weeks, including:
  - hours of lost work due to absenteeism in (a) workplace and (b) household
  - hours of lost work due to presenteeism in (a) workplace and (b) household
  - total [absenteeism + presenteeism] hours of lost work in (a) workplace and (b) household
  - % of scheduled work lost due to absenteeism, presenteeism, and total productivity loss in (a) workplace and (b) household

## 2.2 DISPOSITION OF PATIENTS

This section describes patient disposition for both patient study status and the patient analysis populations.

Screened patients are defined as any patients who signed the informed consent.

Randomized patients consist of all patients with a signed informed consent form who have had a treatment kit number allocated and recorded in the IVRS/IWRS database, regardless of whether the treatment kit was used.

For patient study status, the total number of patients in each of the following categories will be presented in the clinical study report using a flowchart diagram or summary table by treatment arm and overall:

- Screened patients
- Screen failure patients and reasons for screen failure
- Non-randomized but treated patients
- Randomized patients
- Randomized but not treated patients and reason for not being treated
- Randomized and treated patients
- Patients who completed the study treatment period, and patients who did not complete the study treatment period
  - Patients are considered having completed the 52-week blinded treatment period if they received the investigational medicinal product until the day before the Week 52 visit or if the duration of exposure to investigational medicinal product was at least 350 days (52 weeks ± 2 weeks as per protocol)
- Patients who discontinued study treatment by main reason for permanent treatment discontinuation
- Patients who completed the study follow-up period as per protocol and patients who did not complete the study follow-up period as per protocol. For interim analyses, patient ongoing at the cut-off date will also be presented.
- Patients who discontinued study by main reason for study discontinuation
- Vital status (dead or alive) at last study contact

For all categories of patients (except for the screened and non-randomized categories) percentages will be calculated using the number of randomized patients as the denominator. Reasons for treatment discontinuation will be supplied in tables giving numbers and percentages by treatment arm. This summary will be provided by treatment arm.

All critical or major deviations potentially impacting efficacy analyses, randomization, and drug-dispensing irregularities, and other major or critical deviations will be summarized in tables giving numbers and percentages of deviations by treatment group.

Additionally, the analysis populations for efficacy, safety, pharmacokinetics and pharmacodynamics will be summarized in a table.

# 2.2.1 Randomization and drug dispensing irregularities

Randomization and drug-dispensing irregularities occur whenever:

- 1. A randomization is not in accordance with the protocol-defined randomization method, such as
  - a) an ineligible patient is randomized,

- b) a patient is randomized based on an incorrect stratum,
- c) a patient is randomized twice (except for patients from Part 1 who are randomized in Part 2).

OR

- 2. A patient is dispensed an IMP kit not allocated by the protocol-defined randomization, such as
  - a) a patient at any time in the study is dispensed a different treatment kit than as randomized (which may or may not contain the correct-as-randomized IMP),
  - b) a nonrandomized patient is treated with IMP reserved for randomized patients.

Randomization and drug-dispensing irregularities will be monitored throughout the study and reviewed on an ongoing basis.

All randomization and drug-dispensing irregularities will be documented in the clinical study report. If the number of irregularities is large enough to make a tabular summary useful, the irregularities will be categorized and summarized among randomized patients (number and percentages). Nonrandomized, treated patients will be described separately.

Randomization and drug-dispensing irregularities to be prospectively identified include but are not limited to:

#### Randomization and drug allocation irregularities

Kit dispensation without IRT transaction

Erroneous kit dispensation

Kit not available

Randomization by error

Patient randomized twice (except for patients from Part 1 who are randomized in Part 2)

Forced randomization

Stratification error

Patient switched to another site

#### 2.3 ANALYSIS POPULATIONS

Patients treated without being randomized will not be considered randomized and will not be included in any efficacy population.

The randomized population includes any patient who has been allocated to a randomized treatment regardless of whether the treatment kit was used.

For any patient randomized more than once in Part 2 (with two different patient ID), with first randomization being by error, only the data associated with the second patient ID (without randomization code error) will be used in any analysis population.

The safety experience of patients treated and not randomized will be reported separately, and these patients will not be in the safety population.

#### 2.3.1 Efficacy populations

## Part 1: Dose escalation phase

Exploratory efficacy endpoints in Part 1 of the study will be described separately for non-Japanese and Japanese patients:

- The Part 1 non-Japanese ITT population will be defined as all non-Japanese patients randomized in Part 1. Patients will be analyzed in the treatment group to which they were randomized
- The Part 1 Japanese ITT population will be defined as all Japanese patients randomized in Part 1. Patients will be analyzed in the treatment group to which they were randomized

## Part 2: Treatment phase

The Part 2 intent-to-treat (ITT) population will be defined as all randomized patients in Part 2. Patients will be analyzed in the treatment group to which they were randomized

Patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 ITT population and will be described separately. The Part 2 ITT population is the primary analysis population for all efficacy endpoints.

#### 2.3.2 Safety population

The Safety populations considered for safety analyses will be the randomized population who did actually receive at least one dose or part of a dose of the double-blind IMP. Patients will be analyzed according to the treatment actually received.

#### Part 1: Dose escalation phase

Safety data in Part 1 will be described separately for non-Japanese and Japanese patients:

- The Part 1 non-Japanese safety population will be defined as all non-Japanese patients randomized in Part 1 who received at least 1 dose of study medication in Part 1 of the study. All safety analyses in non-Japanese Part 1 of the study will be performed on the Part 1 non-Japanese safety population
- The Part 1 Japanese safety population will be defined as all Japanese patients randomized in Part 1 who received at least 1 dose of study medication in Part 1 of the study. All safety analyses in Japanese Part 1 of the study will be performed on the Part 1 Japanese safety population

## In addition:

• Nonrandomized but treated patients will not be part of the safety population; however, their safety data will be presented separately

- Randomized patients for whom it is unclear whether they took the IMP will be included in the safety population as randomized
- For patients receiving more than 1 study treatment within the same part of the study, the treatment group allocation for as-treated analysis will be the one to which the patient was treated with the longest duration.

## Part 2: Treatment phase

The Part 2 safety population will be defined as all randomized patients in Part 2 who received at least 1 dose of study medication in Part 2 of the study. Patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 safety population, and will be described separately. Safety analyses of the 52-week blinded treatment period of Part 2 of the study will be performed on the Part 2 safety population.

The Part 2 LTFU safety population will be defined as patients who participated to the long-term follow-up period and received at least 1 dose of GZ/SAR402671 after the Week 52 visit. Safety analyses of the long-term follow-up period of Part 2 of the study will be performed on the Part 2 LTFU safety population.

#### In addition:

- Nonrandomized but treated patients will not be part of the safety population; however, their safety data will be presented separately
- Randomized patients for whom it is unclear whether they took the double-blind IMP will be included in the safety population as randomized
- For patients receiving more than 1 double-blind IMP within the same part of the study, the treatment group allocation for as-treated analysis will be the one to which the patient was treated with the longest duration.

#### 2.3.3 Pharmacokinetics population

The PK population will be defined as all patients who received at least 1 dose of GZ/SAR402671 and who have at least one PK assessment.

## Part 1: Dose escalation phase

Pharmacokinetics data in Part 1 will be described separately for non-Japanese and Japanese patients:

- The Part 1 non-Japanese PK populations will be defined as all non-Japanese patients randomized in Part 1 who received at least 1 dose of GZ/SAR402671 and who have at least one PK assessment
- The Part 1 Japanese PK populations will be defined as all Japanese patients randomized in Part 1 who received at least 1 dose of GZ/SAR402671 and who have at least one PK assessment

## Part 2: Treatment phase

The Part 2 PK population will be defined as all patients randomized in Part 2 who received at least 1 dose of GZ/SAR402671 and who have at least one PK assessment.

Patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 PK population, and will be described separately.

## 2.3.4 Pharmacodynamic population

The pharmacodynamic population will be defined as all patients who received at least 1 dose of the double-blind IMP and who have at least one pharmacodynamics assessment.

#### Part 1: Dose escalation phase

Pharmacodynamics data in Part 1 will be described separately for non-Japanese and Japanese patients:

- The Part 1 non-Japanese pharmacodynamics populations will be defined as all non-Japanese patients randomized in Part 1 who received at least 1 dose of double-blind IMP and who have at least one pharmacodynamics assessment
- The Part 1 Japanese pharmacodynamics populations will be defined as all Japanese patients in Part 1 who received at least 1 dose of double-blind IMP and who have at least one pharmacodynamics assessment

#### Part 2: Treatment phase

The Part 2 pharmacodynamics populations will be defined as all patients randomized in Part 2 who received at least 1 dose of GZ/SAR402671 and who have at least one pharmacodynamics assessment.

Patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 pharmacodynamics population, and will be described separately.

#### 2.4 STATISTICAL METHODS

## 2.4.1 Demographics and baseline characteristics

Demographic and baseline characteristics will be presented for the randomized population, separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

Continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, minimum and maximum for each treatment arm. Categorical and ordinal data will be summarized using the number and percentage of patients in each treatment arm.

Parameters will be summarized on the randomized population analyzed in the treatment group to which they were randomized.

Parameters described in Section 2.1.1 will be summarized by treatment group and overall treatment groups using descriptive statistics.

Medical/surgical history will be summarized in each treatment arm by primary SOC, HLT and PT. Events will be sorted by SOC internationally agreed order and decreasing frequency of PT based on the incidence in the overall treatment arm.

P-values on demographic and baseline characteristic data will not be calculated.

#### 2.4.2 Prior or concomitant medications

Prior and concomitant medications will be presented for the randomized population, separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

PD medications will include:

- Dopamine replacement therapies (eg: levodopa/carbidopa)
- Dopamine agonists (eg: pramipexole, ropinerole, bromocriptine)
- Monoamine oxidase B inhibitors (eg: rasagiline)
- Catechol-O-methyltransferase inhibitors (eg: entacapone, tolcapone)
- Anticholinergics (eg: artane, cogentin)

A list of ATC codes to be used in determining PD medications will be provided by the Coding Department.

These medications will be summarized by treatment group, by chemical class and standardized medication name.

Other medications will be summarized by treatment group according to the WHO-DD dictionary, considering the first digit of the anatomic category (ATC) class (anatomic category) and the first 3 digits of the ATC class (therapeutic category). All ATC codes corresponding to a medication will be summarized, and patients will be counted once in each ATC category (anatomic or therapeutic) linked to the medication. Therefore patients may be counted several times for the same medication.

The tables for prior PD medications and prior other medications will be sorted by decreasing frequency of ATC followed by all other therapeutic classes based on the overall incidence across treatment groups. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

The tables for concomitant and post-treatment medications (for PD medications and other medications) will be sorted by decreasing frequency of ATC followed by all other therapeutic classes based on the incidence in the GZ/SAR402671 group (pool of all doses for Part 1). In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

#### 2.4.3 Extent of investigational medicinal product exposure and compliance

The extent of IMP exposure and compliance will be assessed and summarized by actual treatment within the safety population (Section 2.3.2), separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

## 2.4.3.1 Extent of investigational medicinal product exposure

The extent of IMP exposure will be assessed by the duration of IMP exposure.

Within each part of the study, duration of IMP exposure is defined as last dose date – first dose date + 1 day, regardless of unplanned intermittent discontinuations (see Section 2.5.3 for calculation in case of missing or incomplete data).

In Part 2, the duration of exposure to GZ/SAR402671 will be calculated for both patients randomized to the GZ/SAR402671 arm and patients randomized to the placebo arm who received GZ/SAR402671 during the 104-week long term follow-up period.

The duration of exposure to GZ/SAR402671 and the duration of exposure to placebo will be summarized descriptively within each treatment arm, as a quantitative variables (number, mean, SD, median, minimum, and maximum). In addition, duration of treatment exposure will also be summarized cumulatively by numbers and percentages for each of the following categories:

- Part 1:
  - ≥1 day
  - >4 weeks
  - $\geq 8$  weeks
  - $\geq$ 12 weeks
  - ≥24 weeks
  - ≥36 weeks
- Part 2:
  - ≥1 day
  - >4 weeks
  - >8 weeks
  - $\geq$ 13 weeks
  - >26 weeks
  - >39 weeks
  - ≥52 weeks
  - ≥78 weeks
  - ≥104 weeks
  - >130 weeks
- >156 weeks

In addition, the cumulative exposure to treatment (number of patient-years of exposure) will be summarized.

#### 2.4.3.2 Compliance

A given administration will be considered noncompliant if the patient did not take the planned dose of treatment as required by the protocol. No imputation will be made for patients with missing or incomplete data.

Treatment compliance will be defined as the ratio: actual number of capsules taken / (intended daily number of capsules \* duration of treatment exposure) \* 100, where the intended daily number of capsules equals to:

- Part 1:
  - 1 capsule per day for patients in Cohort 1 (4mg or placebo)
  - 2 capsules per day for patients in Cohort 2 (8mg or placebo)
  - 1 capsule per day for patients in Cohort 3 (15mg or placebo)
- Part 2:
  - Double blind treatment period: 1 capsule once per day (15mg or placebo) for 52 weeks
  - Long term follow-up period: 1 capsule once per day (15mg) for additional 104 weeks

Treatment compliance will be summarized descriptively (N, mean, SD, median, min, and max). The percentage of patients with compliance <80% will be summarized.

Cases of overdose are reported in the AE e-CRF pages as AESI if symptomatic or AE if asymptomatic. The reported cases of overdose will be described in the AE analysis (see Section 2.1.4).

## 2.4.4 Analyses of efficacy endpoints

Efficacy endpoints will be presented for the efficacy populations (see Section 2.3.1), separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

In Part 2, efficacy data will be presented separately for the two following periods:

- <u>Analysis of the 52-week blinded treatment period of Part 2</u>. This analysis will present efficacy data from baseline to 52 weeks. Efficacy analyses will compare the two treatment arms:
  - Placebo
  - GZ/SAR402671 15mg

- Analysis of the 156-week treatment period. This analysis will present all efficacy data from baseline to 156 weeks, combining the 52-week blinded treatment period and the 104week long-term follow-up period. Efficacy analyses will compare the two treatment strategies:
  - Delayed start: patients randomized to receive placebo for 52 weeks, then GZ/SAR402671 15mg for 104 weeks.
  - Early start: patients randomized to receive GZ/SAR402671 15mg for 52 weeks, then continued GZ/SAR402671 15mg for 104 weeks.

Details of timing of these two analyses is presented in Section 4.

## 2.4.4.1 Analysis of primary efficacy endpoint(s)

## Part 1: Dose escalation phase

The primary endpoint in Part 1 is safety of each dose cohort. MDS-UPDRS in Part 1 will be analyzed for exploratory purpose (see Section 2.4.4.3).

## Part 2: Treatment phase

All analyses of efficacy endpoints in Part 2 of the study will not include patients from Part 1 who are rerandomized in Part 2. Efficacy data in patients from Part 1 will be described separately, with no formal statistical testing.

#### Estimand

The primary estimand is the difference in mean change from baseline to Week 52 in MDS-UPDRS Part II+III score if all randomized patients had completed the treatment period, regardless of whether or not patients required initiation or intensification of levodopa/PD therapy.

A secondary estimand will be the difference in mean change from baseline to Week 52 in MDS-UPDRS Part II+III score, regardless of whether or not patients completed the treatment period or required initiation or intensification of levodopa/PD therapy.

## Statistical hypotheses

Let  $\mu_0$  and  $\mu_1$  be the population means of the change from baseline to Week 52 in MDS-UPDRS Part II+III score under placebo and GZ/SAR402671, respectively. The primary hypothesis that will be tested is "H0:  $\mu_0 = \mu_1$ " versus "H1:  $\mu_0 \neq \mu_1$ ".

## Primary analysis

In accordance with the primary estimand, the primary analysis will exclude data collected after premature treatment discontinuation. For patients who prematurely discontinued study treatment, any MDS-UPDRS assessed after the date of last administration of the IMP + 7 days

(corresponding to approximately 5 half-lives of GZ/SAR402671) will be excluded from the primary analysis.

Change from baseline in MDS-UPDRS Part II+III score will be analyzed using a mixed effect model with repeated measures (MMRM). All data available at Week 13, Week 26, Week 39 and Week 52 analysis time windows (as defined in Table 6) will be used in the primary analysis. For patients who prematurely discontinued study treatment, data assessed more than 7 days after the date of last administration of the IMP will be excluded from the primary analysis.

The model will include the fixed categorical effects of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), time point (as defined in Table 6), treatment-by-time point interaction, randomization strata-by-time point interaction as well as the continuous fixed covariates of baseline MDS-UPDRS Part II+III score and the baseline-by-time point interaction.

This model will be run using SAS Mixed procedure with an unstructured correlation matrix to model the within-patient errors. Parameters will be estimated using restricted maximum likelihood method. Denominator degrees of freedom will be estimated using Kenward-Roger approximation. This model will provide baseline adjusted least-squares means estimates at Week 52 for both treatment groups with their corresponding standard errors (SEs) and 95% confidence intervals (CI). The difference in baseline adjusted least-squares means will be used to compare the GZ/SAR402671 group to the placebo group, at the 2-sided 0.05 level.

Within group least-squares means and standard errors will be calculated using weights equal to the observed proportion of patients in strata variable levels in the study population (i.e. "population weight") rather than equal weights. Population weights are considered more appropriate than equal coefficients due to expected unbalances in the study population between levels of the randomization stratification factors.

In addition, the relative reduction versus placebo will be calculated as:

Relative reduction (%) = 
$$\left(1 - \frac{\text{LS mean change at Week 52 in GZ/SAR402671 arm}}{\text{LS mean change at Week 52 in placebo arm}}\right) \times 100$$

Relative reduction will be presented with 95% confidence interval using Fieller method. This confidence interval will be calculated provided a significant change is observed in the placebo arm at the 0.05 level. In addition, the posterior probability that GZ/SAR402671 achieves a relative reduction by at least 25% and 50% will be calculated using samples from the asymptotic distribution of LS means from the two treatment arms.

## Sensitivity analysis including data collected after treatment discontinuation

A sensitivity analysis will estimate the difference in mean change from baseline to Week 52 in MDS-UPDRS Part II+III score regardless of whether or not patients completed the treatment period. In this sensitivity analysis, MDS-UPDRS assessed more than 7 days after the last IMP

administration will be included in the analysis. The MMRM model described as primary analysis will be repeated after inclusion of these data.

## Sensitivity analysis with slope-based analysis

The rate of change in MDS-UPDRS Part II+III score from baseline to Week 52 will be estimated using a slope-based analysis assuming linear change from baseline to Week 52. A linear mixed effect model will be fitted, which will include the fixed effect of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), time in years from baseline (as continuous variable), treatment\*time interaction and randomization strata\*time interaction, and will include random intercept and slope. Time (in years) will be calculated as (date of assessment – date of randomization + 1) / 365.25.

Within group mean slope will be obtained from the linear mixed effect and difference in slopes will be presented with the 95% confidence intervals. P-value of the comparison of slopes will be presented for descriptive purpose only.

Relative reduction in slope will be presented with 95% confidence interval. The posterior probability that GZ/SAR402671 achieves a relative reduction in slope by at least 0%, 25% and 50% will be calculated.

## Sensitivity analysis exploring alternative approach regarding missing data

The MMRM model relies on the "missing-at-random" (MAR) assumption. As the possibility for a not-missing-at-random (NMAR) missingness mechanism cannot be excluded, a sensitivity analysis to explore the impact of nonignorable missingness on the primary efficacy analysis will be conducted.

The sensitivity analysis will be based on a pattern-mixture model. Multiple imputations will be generated using a "Copy Increment from Reference" (2) method. Assumptions underlying this method are the following:

- For patients in the GZ/SAR402671 arm who prematurely discontinued the IMP before 52 weeks and had missing data, it will be assumed that after treatment discontinuation, changes in mean profile of the primary endpoint will follow that of the placebo arm, starting from the last observed value. This assumption is considered reasonable in a progressive disease such as PD, where treatment is expected to slow down the progression, but after stopping therapy the disease would continue to progress (3). A schematic representation of the imputation model is provided in Figure 3.
- Missing data in patients from the placebo arm or in patients from the GZ/SAR402671 arm who completed the 52-week treatment period will be imputed assuming they are MAR



Figure 3 - Schematic representation of imputation of missing data – Sensitivity analysis using Copy Increment from Reference (CIR) method

Multiple imputations will be generated using SAS macros developed by James Roger (4). The imputation model will include adjustment for randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no).

Missing values will be imputed 1,000 times to generate 1,000 complete data sets. Each completed dataset will be analyzed using an analysis of covariance (ANCOVA) of change from baseline to Week 52 in MDS-UPDRS Part II+III score, including the fixed categorical effects of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), as well as the continuous fixed covariates of baseline value. The final results will be obtained by combining the least squares means and least squares mean differences from these 1,000 analyses, using Rubin's formula.

Sensitivity analysis exploring alternative approach regarding assessment during the OFF state

In the protocol, instructions were given to assess MDS-UPDRS during the OFF state. Patients should not take their PD medications for at least 12 hours prior to the assessment. Different sensitivity analyses will explore the impact of assessment of MDS-UPDRS performed less than 12 hours after intake of PD medication.

These sensitivity analyses will be performed as following:

- Excluding any MDS-UPDRS assessed less than 12 hours after intake of PD medication (irrespective of clinical state)
- Excluding any MDS-UPDRS assessed less than 6 hours after intake of PD medication (irrespective of clinical state)
- Excluding any MDS-UPDRS assessed less than 12 hours after intake of PD medication and for which the clinical state was recorded as "ON".
- Excluding any MDS-UPDRS assessed less than 6 hours after intake of PD medication and for which the clinical state was recorded as "ON".

The MMRM model described as primary analysis will be repeated after exclusion of these data.

## Sensitivity analyses assessing randomization strata

A sensitivity analysis will estimate the difference in mean change from baseline to Week 52 in MDS-UPDRS Part II+III score after including the actual strata derived from data instead of the strata recorded in IVRS (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no). The purpose of this analysis will be to assess the impact of discrepancies observed between the strata recorded in the IVRS and the ones derived from data. The MMRM model described as primary analysis will be repeated after including the actual strata.

## Secondary analysis

A secondary analysis will describe the number and percentage of patients with MDS-UPDRS Part II+III score improvement, no change or worsening at Week 52 based on minimal clinically important difference threshold values in patients with Hoehn&Yahr 1&2 (5):

- Improvement will be defined as change in MDS-UPDRS Part II+III  $\leq$  -4.3
- Worsening will be defined as change in MDS-UPDRS Part II+III  $\geq 3.9$
- No change will be defined as change in MDS-UPDRS Part II+III > -4.3 and <3.9

Patients without any available assessment at Week 52 will be considered as worsened.

#### Subgroup analyses

The MMRM model described as primary analysis will be repeated in each of the following subgroups as appropriate, the p-values will not be adjusted for multiplicity and will be provided for descriptive purpose only, and forest plots will be provided:

- Sex (Male vs. Female);
- Age ( $\leq 60 \text{ vs.} > 60$ );
- GBA mutations (severe vs. non severe): Severe GBA mutation subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);

- Prior PD medications (yes vs. no): Prior PD medication subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);
- Time since onset of symptoms (<= 6 years vs > 6 years);
- Time since diagnosis (<= 6 years vs > 6 years);
- MDS-UPDRS Part II+III at baseline (<=35 vs. > 35);
- Hoehn and Yahr at baseline (<2 vs. >= 2);
- MoCA score at baseline (< 26 vs. >= 26): MoCA score subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);

Unless otherwise specified (see below), for each subgroup analysis, the MMRM model will include the fixed categorical effects of treatment group, randomization strata as per IVRS, subgroup factor, time point, treatment-by-time point interaction, strata-by-time point interaction, subgroup factor-by-time point interaction, treatment-by-subgroup factor interaction, and treatment-by-subgroup-by-time point interaction, as well as the continuous fixed covariates of baseline value and baseline value-by-time point interaction. Exceptions will be made for the following subgroup analyses:

- For subgroup analyses by GBA mutation, the MMRM will not include the randomization stratum of severe GBA mutation (yes/no)
- For subgroup analyses by prior PD medication, the MMRM will not include the randomization stratum of use of levodopa/PD medication (yes/no)
- For subgroup analysis by MoCA score at baseline, the MMRM will not include the randomization stratum of MoCA score <26 (yes/no)
- For subgroup analysis by MDS-UPDRS Part II+III at baseline (<=35 vs. > 35), the MMRM will not include adjustment for baseline

## 2.4.4.2 Analyses of secondary efficacy endpoints

#### Part 1: Dose escalation phase

Not Applicable.

#### Part 2: Treatment phase

Secondary efficacy endpoints include:

- Change in PD-CRS (total score) from baseline to Week 52.
- Change in MDS-UPDRS Parts I+II+III from baseline to Week 52.
- Change in H&Y stage from baseline to Week 52.

Secondary endpoints will be analyzed using the same MMRM model as for the primary efficacy endpoint. For patients who prematurely discontinued study treatment, data collected more than 7 days after the last IMP administration will be excluded from the analysis of secondary endpoints.

### Subgroup analyses

The MMRM model described as primary analysis will be repeated in each of the following subgroups as appropriate, the p-values will not be adjusted for multiplicity and will be provided for descriptive purpose only, and forest plots will be provided:

- GBA mutations (severe vs. non severe): Severe GBA mutation subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);
- Prior PD medications (yes vs. no): Prior PD medication subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);
- Time since diagnosis (<= 6 years vs > 6 years);
- Hoehn and Yahr at baseline (<2 vs. >= 2);
- MoCA score at baseline (< 26 vs. >= 26): MoCA score subgroup will be defined using actual subgroup (not randomization stratum as per IVRS);

Unless otherwise specified (see below), for each subgroup analysis, the MMRM model will include the fixed categorical effects of treatment group, randomization strata as per IVRS, subgroup factor, time point, treatment-by-time point interaction, strata-by-time point interaction, subgroup factor-by-time point interaction, treatment-by-subgroup factor interaction, and treatment-by-subgroup-by-time point interaction, as well as the continuous fixed covariates of baseline value and baseline value-by-time point interaction. Exceptions will be made for the following subgroup analyses:

- For subgroup analyses by GBA mutation, the MMRM will not include the randomization stratum of severe GBA mutation (yes/no)
- For subgroup analyses by prior PD medication, the MMRM will not include the randomization stratum of use of levodopa/PD medication (yes/no)
- For subgroup analysis by MoCA score at baseline, the MMRM will not include the randomization stratum of MoCA score <26 (yes/no)

Further subgroup analyses may be performed if deemed necessary for interpretation of results.

#### Secondary analysis

A secondary analysis will describe the percentage of patients with MDS-UPDRS Part I+II+III score improvement, no change or worsening at Week 52 based on minimal clinically important difference threshold values in patients with Hoehn&Yahr 1&2 (5):

- Improvement will be defined as a change in MDS-UPDRS Part I+II+III  $\leq$  -5.9
- Worsening will be defined as a change in MDS-UPDRS Part I+II+III ≥ 3.7
- No change will be defined as a change in MDS-UPDRS Part I+II+III > -5.9 and <3.7

Patients without any available assessment at Week 52 will be considered as worsened.

#### 2.4.4.3 Analyses of exploratory efficacy endpoints

## Part 1: Dose escalation phase

Descriptive statistics for values and changes from baseline will be presented by treatment arm for each time point. All measurements will be assigned to analysis windows defined in Section 2.5.4, Table 3 in order to provide an assessment for Week 2 to Week 52 time points. For patients who prematurely discontinued study treatment, data collected more than 7 days after the last IMP administration will be excluded from the analysis of exploratory endpoints.

Continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, Q1, Q3 minimum and maximum for each treatment arm at each time point. Categorical and ordinal data will be summarized using the number and percentage of patients in each treatment arm at each time point.

Summary statistics will be provided for the following endpoints:

- MDS-UPDRS: Part II+III score, Part I+II+III score, as well as each part separately (Part I, Part II, Part III)
- Hoehn & Yahr scale, as a categorical variable:
  - Stage 0: No symptoms
  - Stage 1: Symptoms on one side of the body only
  - Stage 2: Symptoms on both sides of the body. No impairment of balance
  - Stage 3: Balance impairment. Mild to moderate disease. Physically independent
  - Stage 4: Severe disability, but still able to walk or stand unassisted
  - Stage 5: Wheelchair-bound or bedridden unless assisted
- PD-CRS: Total score, as well as sub-scores: PD-CRS Fronto-subcortical score PD-CRS Posterior-cortical score
- MoCA: Total score, as a quantitative and categorical variable:
  - <26
  - >26
- Oral SDMT score
- Trail Making Test: TMT-A, TMT-B and difference between TMT-B score minus TMT-A
- Clinical global impression scale: severity of illness and efficacy index (as a categorical variable)
- Patient Global Impression of Change (as a categorical variable)

## Part 2: Treatment phase

All analyses of exploratory efficacy endpoints will be done on Part 2 of the study and will not include patients from Part 1 who are rerandomized in Part 2. Descriptive statistics for values and

changes from baseline will be presented by treatment arm for each time point, p-values for exploratory endpoints may be provided for descriptive purpose only. All measurements will be assigned to analysis windows defined in Section 2.5.4, Table 6 in order to provide an assessment from baseline to Week 156 time points.

## Continuous endpoints

Percent change from baseline to Week 52 in DaTSCAN assessment scores (SBR) will be analyzed using an ANCOVA. The model will include the fixed categorical effects of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), as well as the continuous fixed covariate of baseline.

For all other continuous exploratory endpoints, descriptive statistics by visit will be provided for each treatment arm. Summary statistics (including number of available data, mean, SD, median, Q1, Q3, minimum and maximum) will be presented for value, change from baseline and percent change from baseline (when applicable). Further analyses using MMRM (if repeated assessments) or ANCOVA (if single assessment) may be performed when appropriate.

### Categorical endpoints

Categorical exploratory endpoints described in Section 2.1.3.3 will be summarized by visit, using the number and percentage of patients in each treatment arm.

## <u>Time-to-event endpoints</u>

Time to first occurrence of event of interest data will be presented in terms of cumulative incidence probabilities of occurrence with 95% CI as well as the number of patients at risk, number of patients censored and number of events at key time points (week 13, week 26, week 39 and week 52) using the Kaplan-Meier method and estimates. For time to event exploratory outcomes, statistical comparisons between treatment arms will be carried out using a log-rank test and presented for exploratory purpose only. In addition, Kaplan-Meier curves and summary statistics and estimates showing number of patients at risk and cumulative incidence of events of interest at key time points (week 13, week 26, week 39 and week 52), and appropriate CI may be provided for each treatment arm.

• Time to first initiation of levodopa or other PD medication (for patients not on levodopa/other PD medication at baseline) or to increased dose of levodopa/other PD medication (for patients on levodopa/other PD medication at baseline) is defined as: the time from the date of randomization to the date of first initiation of levodopa or other PD medication (for patients not on levodopa/other PD medication at baseline) or as the time from date of randomization to the date of first documentation of (intensification dose of levodopa/other PD medication (for patients on levodopa/other PD medication at baseline). If no initiation or intensification of levodopa or other PD medication is documented before the first step final analysis date (when all patients from Part 2 have been randomized and have all their data up to Week 52 collected and validated) or database lock, time to first initiation will be censored at the date of last visit or at the date of randomization + 365

days whichever comes first. Definitions of initiation and intensification of PD medication are detailed in Section 2.1.3.3.

• Time to first reduction or stop of levodopa/PD medication (for patients on levodopa/other PD medication at baseline) defined as: the time from the date of randomization to the date of first documentation of reduction or to the date of stop of levodopa/PD medication (for patients on levodopa/other PD medication at baseline). If no reduction or stop of levodopa or other PD medication is documented before the first step final analysis date (when all patients from Part 2 have been randomized and have all their data up to Week 52 collected and validated) or database lock, time to first reduction will be censored at the date of last visit or at the date of randomization + 365 days whichever comes first. Definitions of reduction and stop of PD medication are detailed in Section 2.1.3.3.

## 2.4.4.4 Multiplicity issues

## Part 1: Dose escalation phase

Not Applicable.

## Part 2: Treatment phase

In order to handle multiple secondary endpoints, the overall type-I error will be controlled by the use of a hierarchical approach. Statistical significance of the primary endpoint at the two-sided 0.05 alpha level is required before drawing inferential conclusions about first secondary endpoint (refer to order of list in Section 2.1.3.2). Inferential conclusions about successive secondary endpoints require statistical significance of the prior one.

This fixed hierarchical approach will ensure a strong control of the overall type-I error rate at the two-sided 0.05 level.

No further adjustments will be made for exploratory endpoints for which p-values will be provided for descriptive purpose only.

#### 2.4.5 Analyses of safety data

Safety analyses will be performed on the safety populations (see Section 2.3.2), separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

In Part 2, safety data will be presented separately for the two following periods:

- <u>Safety analysis of the 52-week blinded treatment period of Part 2</u>. This analysis will present safety data collected up to the Week 52 visit (or end of treatment visit in case of premature treatment discontinuation before Week 52). Safety analyses will present safety data from the two treatment arms:
  - Placebo
  - GZ/SAR402671 15mg

- Safety analysis of the 104-week long-term follow-up period of Part 2. This analysis will present safety data collected from the Week 52 visit to the end of study, excluding the initial 52-week blinded treatment period. Only patients having received GZ/SAR402671 15mg during the long-term follow-up period will be included in this analysis. Safety analyses will present safety data from the following groups:
  - Delayed start: patients having received placebo during the 52-week treatment period, then having received GZ/SAR402671 during the long-term follow-up period.
  - Early start: patients having received GZ/SAR402671 during the 52-week treatment period, then having continued to receive GZ/SAR402671 during the long-term follow-up period.
  - All patients: all patients having received GZ/SAR402671 during the long-term follow-up period
- Safety analysis of the overall GZ/SAR402671 treatment period in Part 2. This analysis will present all safety data collected from the first intake of GZ/SAR402671 in Part 2 to the last intake of GZ/SAR402671 in Part 2 plus 6 weeks. All patients having received GZ/SAR402671 15mg in Part 2 (either during the 52-week blinded treatment period or during the long-term follow-up period) will be included in this analysis. Safety analyses will present safety data from the following group:
  - Overall GZ/SAR402671: patients having received GZ/SAR402671 during the 52-week treatment period and/or during the long-term follow-up period.

Details of timing of these two analyses is presented in Section 4.

#### General common rules

The safety analysis will be conducted according to the Sanofi document BTD-009536 (version applicable at the time of database lock) "Analysis and reporting of safety data from Clinical Trials through the Clinical Study Report."

All safety analyses will be performed using the following common rules:

- Safety data in patients who do not belong to the safety population (eg, exposed but not randomized) will be listed separately.
- The baseline value is defined in Section 2.1.1
- The potentially clinically significant abnormality (PCSA) values are defined as abnormal values considered medically important by the Sponsor according to predefined criteria/thresholds based on literature review and defined by the Sponsor for clinical laboratory tests, vital signs, and ECG (PCSA version dated 24 May 2014 [Appendix A])
- PCSA criteria will determine which patients had at least 1 PCSA during the TEAE period, taking into account all evaluations performed during the TEAE period, including unscheduled or repeated evaluations. The number of all such patients will be the numerator for the on-treatment PCSA percentage

- The treatment-emergent PCSA denominator by arm for a given parameter will be based on the number of patients assessed for that given parameter in the TEAE period by treatment arm on the safety population
- For quantitative safety parameters based on central laboratory/reading measurements, descriptive statistics will be used to summarize results and change from baseline values by time point and treatment arm. Summaries will include the endpoint baseline value, the last on-treatment value and change from baseline, the worst on-treatment value and change from baseline. The last on-treatment value is commonly defined as the last value collected during the treatment period (see Section 2.1.4). The worst on-treatment value is defined as the nadir and /or the peak post-baseline during the treatment period according to the direction (minimum or maximum) of the abnormality as defined in the PCSA list
- All measurements (scheduled or unscheduled) will be re-allocated as given in Section 2.5.4, Table 3 and Table 6 and re-allocated visits measurements will be included in the by-time point summary
- The analysis of the safety variables will be essentially descriptive and no systematic testing is planned

#### 2.4.5.1 Analyses of adverse events

#### **Generalities**

The primary focus of AE reporting will be on TEAE as defined in Section 2.1.4. Pre-treatment and post-treatment adverse events (including SAEs and AESIs) will be described separately.

If an AE date/time of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the AE as pre-treatment, treatment-emergent, or post-treatment. The algorithm for imputing date/time of onset will be conservative and will classify an AE as treatment emergent unless there is definitive information to determine it is pre-treatment or post-treatment. Details on classification of AEs with missing or partial onset dates are provided in Section 2.5.3.

Adverse event incidence tables will present by SOC, HLGT, HLT, and PT, for each treatment arm, the number (n) and percentage (%) of patients experiencing an AE sorting based on results of column all. Multiple occurrences of the same event in the same patient will be counted only once in the tables within a treatment period. The denominator for computation of percentages is the safety population within each treatment arm.

Sorting within tables ensures the same presentation for the set of all AEs within the observation period (pre-treatment, treatment-emergent, and post-treatment). For that purpose, the table of all TEAEs presented by SOC and PT sorted by the internationally agreed SOC order and decreasing frequency of PTs within SOCs will define the presentation order for all other tables unless otherwise specified. Sorting will be based on results of column all.

### Analysis of all TEAEs

The following TEAE summaries will be generated for the safety populations.

- Overview of TEAEs by treatment arm, summarizing number (%) of patients with any
  - TEAE
  - Serious TEAE
  - Treatment-emergent AESI
  - TEAE leading to death
  - TEAE leading to permanent treatment discontinuation
- All TEAEs by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least 1 TEAE sorted by the SOC internationally agreed order. The other levels (HLGT, HLT, and PT) will be presented in alphabetical order. This table will be presented by treatment arm
- All TEAEs by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC. This sorting order will be applied to all other tables, unless otherwise specified. This table will be presented by treatment arm
- Number (%) of patients experiencing common TEAE(s) (PT incidence ≥5% in any treatment group) presented by primary SOC and PT, sorted by the sorting order defined aboved
- All TEAEs related to IMP by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE, sorted by the sorting order defined above. This table will be presented by treatment arm
- All TEAEs by maximal severity, presented by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE by severity (ie, mild, moderate, or severe), sorted by the sorting order defined above. This table will be presented by treatment arm

#### Analysis of all treatment emergent serious adverse event(s)

- All treatment-emergent serious adverse events by primary SOC and PT, showing the number (%) of patients with at least 1 serious TEAE, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC. This table will be presented by treatment arm
- Listings will be provided for all serious adverse events (SAE)s by treatment arm during on-treatment period

#### Analysis of all treatment-emergent adverse event(s) leading to treatment discontinuation

• All TEAEs leading to treatment discontinuation, by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC. This table will be presented by treatment arm

### Analysis of all treatment emergent AESI

• All treatment-emergent AESI by primary SOC and PT, showing the number (%) of patients with at least 1 treatment-emergent AESI, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC. This table will be presented by treatment arm.

## Analysis of pretreatment and posttreatment adverse events

An overview presenting number of patients with any pre-/post-treatment adverse events, serious pre-/post-treatment adverse events, pre-/post-treatment adverse events leading to death, pretreatment adverse events leading to permanent treatment discontinuation, pre-/post-treatment AESI will be displayed by treatment arm. If only few patients (<10% of randomized patients) are concerned, a global listing will be provided.

#### 2.4.5.2 Deaths

The following summaries of deaths will be generated for the safety population by treatment arm.

- Number (%) of patients who died by study period (on-study, on TEAE period, post-study) and reasons for death summarized on the safety population by treatment received
- Deaths in nonrandomized patients or randomized but not treated patients
- TEAEs leading to death (death as an outcome on the AE case report form page as reported by the Investigator) by primary SOC and PT showing number (%) of patients with at least 1 TEAE leading to death, sorted by internationally agreed SOC order and by decreasing incidence of PTs within each SOC. This table will be presented by treatment received
- Listings of deaths will be provided. For deaths in non-randomized patients or randomized and not treated patients, a distinct listing will be provided

#### 2.4.5.3 Analyses of laboratory variables

The summary statistics (including mean, standard deviation, median, Q1, Q3, minimum, and maximum) of all laboratory variables (central laboratory values and changes from baseline) will be calculated for each visit, last and worst value assessed during the treatment period, and presented by treatment group. For selected parameters, mean changes from baseline with the corresponding standard error will be plotted over time (at same time points) in each treatment group.

The incidence of PCSAs at any time during the TEAE period (on-treatment PCSAs) will be summarized by treatment group whatever the baseline level and/or according to the following baseline categories:

- Normal/missing
- Abnormal according to PCSA criterion or criteria

For laboratory parameters for which PCSA criterion is not defined, similar table(s) using the normal range could be provided.

#### Drug-induced liver injury

The liver function tests, namely Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline Phosphatase (ALP) and Total Bilirubin are used to assess possible drug induced liver toxicity. The proportion of patients with PCSA values at any post-baseline visit by baseline status will be displayed by treatment group for each parameter.

A e-DISH graph of distribution of peak values of ALT versus peak values of Total bilirubin will also be presented. Note that the ALT and Total bilirubin values are presented on a logarithmic scale. The graph will be divided into 4 quadrants with a vertical line corresponding to 3xULN for ALT and a horizontal line corresponding to 2xULN for Total bilirubin.

Listing of possible Hy's Law cases identified by treatment group (eg, subjects with any elevated ALT of >3xULN, and associated with an increase in bilirubin >2xULN) will display: ALT, AST, ALP, gamma-glutamyl transferase (GGT), total and conjugated bilirubin, prothrombin time (PT), partial thromboplastin time (PTT) international normalized ratio (INR), serum creatinine and complete blood count.

The normalization by parameter (to ≤1 ULN or return to baseline) of elevated liver function tests will be summarized by categories of elevation defined in the PCSA document (with following categories of normalization: normalized before last IMP dose, normalized after last IMP dose, and never Normalized. Note that a patient will be counted only under the maximum elevation category. Note: patients in the category of 'either elevated ALT or AST' are considered normalized only if both ALT and AST return to <1 ULN or to the baseline value.

The incidence of liver related AEs will be summarized by treatment group. The selection of PT will be based on SMQ Hepatic disorder.

## 2.4.5.4 Analyses of vital sign variables

The summary statistics (including number, mean, median, standard deviation, minimum and maximum) of all vital signs variables (raw data and changes from baseline) will be calculated for each time point or study assessment (baseline, each post-baseline time point, endpoint) by treatment arm. For parameters heart rate, systolic and diastolic blood pressures, the last on-treatment and worst on-treatment value will also be provided.

The incidence of PCSAs at any time during the TEAE period will be summarized by treatment arm irrespective of the baseline level and according to the following baseline status categories:

- Normal/missing
- Abnormal according to PCSA criterion or criteria

Listings will be provided with flags indicating the out of range values as well as PCSA values.

#### 2.4.5.5 Analyses of electrocardiogram variables

The summary statistics (including number, mean, median, standard deviation, minimum and maximum) of all ECG variables (central reading values and changes from baseline) will be calculated for each time point or study assessment (baseline, each post-baseline time point, endpoints) by treatment arm.

The incidence of PCSAs at any time during the TEAE period will be summarized by treatment arm irrespective of the baseline level and according to the following baseline status categories:

- Normal/missing
- Abnormal according to PCSA criterion or criteria

Listings will be provided with flags indicating the out of range values as well as PCSA values.

## 2.4.5.6 Analyses of physical examination variables

Number and percentages of patients with abnormal physical examinations at any time during the TEAE period (see Section 2.1.4) will be summarized. A listing will be provided for patients with abnormal physical examination.

#### 2.4.5.7 Analyses neurological examination variables

Number and percentages of patients with abnormal neurological examination at any time during the TEAE period (see Section 2.1.4) will be summarized. A listing will be provided for patients with abnormal neurological examination.

## 2.4.5.8 Analyses of ophthalmological examination variables

Number and percentages of patients with any abnormal ophthalmological examination on any eye at any time (whether present at screening or not) as well as number and percentages of patients with any new onset of abnormal ophthalmological examination on any eye during the TEAE period (see Section 2.1.4) as per investigator (site ophtalmologiste) assessment will be summarized. A listing will be provided for patients with new onset of abnormal ophthalmological examination on any eye during the TEAE period.

Number and percentages of patients with any definite worsening of lens opacity on any eye as well as number and percentages of patients with any possible worsening of lens opacity on any eye during the TEAE period (see Section 2.1.4) as per central reader assessment will be summarized along with a description of lens opacity grading according to the ARLNS grading system (1). A listing will be provided for patients with worsening (definite or possible) of lens opacity on any eye during the TEAE period.

### 2.4.5.9 Analyses of depression data

Descriptive statistics for values and changes from baseline in BDI-II total score will be presented by treatment arm for each time point during the on-treatment period (see Section 2.1.4). All measurements will be assigned to analysis windows defined in Section 2.5.4, Table 3 in order to provide an assessment for Week 2 to Week 52 time points. BDI-II total score continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, minimum and maximum for each treatment arm.

In addition, the worst (highest) BDI-II total score value during the treatment-emergent period will be categorized and summarized using the number and percentage of patients in each treatment arm within each of the following categories:

- 0-13 (minimal depression)
- 14-19 (mild depression)
- 20-28 (moderate depression)
- 29-63 (severe depression)

In addition, the worst (highest) score during the treatment-emergent period for suicidal thoughts (item 9 of BDI-II) will be summarized using the number and percentage of patients in each treatment arm within each of the following categories:

- I don't have any thoughts of killing myself
- I have thoughts of killing myself but I would not carry them out
- I would like to kill myself
- I would kill myself if I had the chance

In addition, the number of participants with BDI-II worsening from baseline during the treatment emergent period will be summarized.

## 2.4.6 Analyses of pharmacokinetic and pharmacodynamic variables

Pharmacokinetic and pharmacodynamic variables will be presented for the Pharmacokinetics and pharmacodynamic populations respectively (see Section 2.3.3 and Section 2.3.4), separately for Part 1 and Part 2 of the study. In Part 1, data will be presented separately for Japanese and non-Japanese patients.

#### 2.4.6.1 Analyses of pharmacodynamic variables

Pharmacodynamic data will be described separately for Part 1 and Part 2 of the study, and separately for Japanese and non-Japanese patients. Data of patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 and will be presented separately.

#### Part 1: Dose escalation phase

For all pharmacodynamics parameters, raw data and percent change from baseline will be summarized in descriptive statistics by treatment group and scheduled time of measurement for each population separately (Japanese and non-Japanese patients). No formal statistical comparison will be made.

Additionally, graphs over time will be presented plotting mean +/- SD by treatment group for each population separately (Japanese and non-Japanese patients).

## Part 2: Treatment phase

In Part 2, pharmacodynamics data will be presented separately for the two following periods:

- <u>Analysis of the 52-week blinded treatment period of Part 2</u>. This analysis will present pharmacodynamics data from baseline to 52 weeks. Pharmacodynamic analyses will compare the two treatment arms:
  - Placebo
  - GZ/SAR402671 15mg
- Analysis of the 156-week treatment period. This analysis will present all
  pharmacodynamics data from baseline to 156 weeks, combining the 52-week blinded
  treatment period and the 104-week long-term follow-up period. Pharmacodynamic
  analyses will compare the two treatment strategies:
  - Delayed start: patients randomized to receive placebo for 52 weeks, then GZ/SAR402671 15mg for 104 weeks.
  - Early start: patients randomized to receive GZ/SAR402671 15mg for 52 weeks, then continued GZ/SAR402671 15mg for 104 weeks.

Percent change from baseline to Week 26 and Week 52 in plasma GL-1 will be analyzed using a MMRM including data available at Week 2, Week 4, Week 13, Week 26, Week 39 and Week 52 analysis time windows (as defined in Table 6). The model will include the fixed categorical effects of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), time point (as defined in Table 6), treatment-by-time point interaction, randomization strata-by-time point interaction as well as the continuous fixed covariates of baseline and the baseline-by-time point interaction

Percent change from baseline to Week 52 in CSF GL-1 will be analyzed using an Analysis of Covariance (ANCOVA). The model will include the fixed categorical effects of treatment group (GZ/SAR402671 versus placebo), randomization strata (use of levodopa/PD medication: yes/no, MoCA score <26: yes/no and severe GBA mutation: yes/no), as well as the continuous fixed covariate of baseline.

For all other continuous exploratory endpoints, descriptive statistics by visit will be provided for each treatment arm. Summary statistics (including number of available data, mean, SD, median, minimum and maximum) will be presented for value, change from baseline and percent change

from baseline (when applicable). Further analyses using MMRM (if repeated assessments) or ANCOVA (if single assessment) may be performed when appropriate.

## 2.4.6.2 Analyses of pharmacokinetic variables

Pharmacokinetic data will be described separately for Part 1 and Part 2 of the study, Data of patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2.

For Part-1 Dose escalation phase: Pharmacokinetic parameters of GZ/SAR402671 in plasma and in CSF will be summarized by descriptive statistics (such as mean, geometric mean, median, SD, SEM, CV, minimum, and maximum) by visit and and treatment groups. Descriptive statistics could be provided by specific subgroups (e.g Japanese and non-Japanese), as needed. PK samples collected outside of the sampling time window as mentioned in section 2.1.5 (Pharmacokinetic variables) or PK samples collected as unscheduled samples will be classified as "undefined concentrations". No descriptive statistics will be performed on these concentrations. This analysis will be performed under the responsibility of Pharmacokinetics, Dynamics and Metabolism (PKDM), Bridgewater, Sanofi.

For Part-2 Treatment phase: Pharmacokinetic parameters of GZ/SAR402671 in plasma and in CSF will be summarized by descriptive statistics (such as mean, geometric mean, median, SD, SEM, CV, minimum, and maximum) by visit. Descriptive statistics could be provided by specific subgroups (e.g Japanese and non-Japanese), as needed. PK samples collected outside of the sampling time window as mentioned in section 2.1.5 (Pharmacokinetic variables) or PK samples collected as unscheduled samples will be classified as "undefined concentrations". No descriptive statistics will be performed on these concentrations. This analysis will be performed under the responsibility of Pharmacokinetics, Dynamics and Metabolism (PKDM), Bridgewater, Sanofi.

Other statistical analyses described below will be performed under the responsibility of Biostatistics, Sanofi.

#### Part 1: Dose escalation phase

#### Accumulation

For C<sub>max</sub> and AUC<sub>0-24</sub>, accumulation will be assessed with a linear model for each population separately (Japanese and non-Japanese patients),

Log(Ratio of Week 4 versus Day 1) = Dose + Error

with dose as fixed effect using SAS Proc Mixed®.

Accumulation ratio of Week 4 versus Day 1 will be assessed for each population separately (Japanese and non-Japanese patients) and for each dose level separately as well as pooled across dose levels within the model framework. Estimate and 90% confidence interval for the accumulation ratio will be obtained by computing estimate and 90% confidence interval for the logarithm of the accumulation ratio within the linear model framework, and then converting to the accumulation ratio by the antilog transformation.

Listings of individual accumulation ratios will be provided, along with their descriptive statistics.

### Dose proportionality

For each population separately (Japanese and non-Japanese patients) and for  $C_{max}$ ,  $AUC_{0.24}$  and CSF concentration (on Week 4 only), dose proportionality will be assessed on Day 1 and Week 4 separately using the empirical power model (pharmacokinetics parameter =  $\alpha$  x dose $\beta$ ), along with an "estimation" interpretation, according to the recommendations in Gough et al. (1995):

"The empirical power model provides a readily and interpretable measure of the degree of non-proportionality, which can be used both to confirm proportionality and to assess the pharmacokinetic and clinical significance of any departures."

"The analysis of dose proportionality studies, however, requires estimation rather than significance testing in order that the pharmacokinetic and clinical significance of any non-proportionality can be assessed."

The power model will be fit on the log-transformed scale:  $log(parameter) = log(\alpha) + \beta x log(dose)$ . Model lack-of-fit will be assessed by residual plots, and by an F-test of the residual mean square versus the pure error residual mean square. If the model fit is adequate, estimates with 90% confidence intervals for  $\beta$  will be obtained, and further used to obtain estimates and 90% confidence intervals for the pharmacokinetics parameter increase associated with an r-fold (r = 2 and r = high dose / low dose) increase in dose, by exponentiating r to the powers of the  $\beta$  estimate and confidence limits,

$$\mathbf{r}^{b \pm t \times SE(b)}$$

If there is evidence of model lack-of-fit, then attempts could be made to fit the model over a reduced dose range (eg, exclude 1 extreme dose level). Otherwise, a linear model will be used, with fixed term for dose, using logarithms of the relevant pharmacokinetics parameters. Estimates with 90% confidence intervals for the parameter increases associated with pairwise dose increases will be obtained by first computing estimates with confidence intervals for differences between pairwise dose groups in the linear model framework, and then converting to ratios using the antilog transformation.

## Dose effect

The distribution of  $t_{max}$  values will be represented by histogram plots for each dose level.

#### Variance components

For each population separately (Japanese and non-Japanese patients), within-subject and total standard deviations for  $log(C_{max})$  and  $log(AUC_{0-24})$  will be estimated by equating observed and expected means squares within the following linear model framework,

$$log(parameter) = Dose + Day + Day \times Dose + Subject(Dose)$$

with fixed effects for dose, day and day-by-dose interaction, and with subject-within-dose as random effect. 90% confidence intervals will be computed using the simple  $\chi 2$  method for the within-subject SD, and the Graybill-Wang procedure for the total SD.

#### 2.4.7 Analyses of quality of life variables

## Part 1: Dose escalation phase

Descriptive statistics for values and changes from baseline will be presented by treatment arm for each time point. Continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, minimum and maximum for each treatment arm.

Summary statistics will be provided for the following exploratory endpoints:

- PDQ-39 questionnaire, including:
  - Mobility
  - Activities of daily living
  - Emotional well-being
  - Stigma
  - Social support
  - Cognition
  - Communication
  - Bodily discomfort
  - PDQ-39 single index (PDQ-39-SI)
- EQ5D: utility index and overall health status
- HRPQ including:
  - Hours of lost work due to absenteeism in (a) workplace and (b) household
  - Hours of lost work due to presenteeism in (a) workplace and (b) household
  - Total [absenteeism + presenteeism] hours of lost work in (a) workplace and (b) household
  - % of scheduled work lost due to absenteeism, presenteeism, and total productivity loss in (a) workplace and (b) household

#### Part 2: Treatment phase

Data of patients from Part 1 who are rerandomized in Part 2 will not be included in Part 2 and will be presented separately.

Quality of life endpoints described in Section 2.1.3.3 will be analyzed using descriptive statistics for values and changes from baseline will be presented by treatment arm for each time point. Continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, minimum and maximum for each treatment arm.

#### 2.5 DATA HANDLING CONVENTIONS

#### 2.5.1 General conventions

The following formulas will be used for computation of parameters.

## Demographic formulas

• BMI = 
$$\frac{\text{weight(kg)}}{\text{height(m)}^2}$$

#### Parkinson's disease history

- Time since onset of symptoms (in years):
  - If complete date of onset of symptoms available: (date of informed consent date of onset of symptoms)/365.25
  - If only year and month of onset of symptoms available: (year/month part of date of informed consent year/month part of date of onset of symptoms)/12
  - If only year of onset of symptoms available: (year part of date of informed consent year part of date of onset of symptoms)
- Time since diagnosis (in years)
  - If complete date of diagnosis available: (date of informed consent date of diagnosis)/365.25
  - If only year and month of diagnosis available: (year/month part of date of informed consent year/month part of date of diagnosis)/12
  - If only year of diagnosis available: (year part of date of informed consent year part of date of diagnosis)

## ECG formulas

• Bazett (QTcB (eçums)): 
$$\frac{QT \text{ (ms)}}{\sqrt{60/HR(bpm)}}$$

• Fridericia (QTcF (ms)): 
$$QT (ms)$$

$$\sqrt[3]{60/HR(bpm)}$$

## Renal function formulas

eGFR value will be derived using the CKD-EPI formula (6):

eGFR (mL/min/1.73m<sup>2</sup>) = 
$$141 \times \min(\text{Scr/}\kappa, 1)^{\alpha} \times \max(\text{Scr/}\kappa, 1)^{-1.209} \times 0.993^{\text{Age}} \times 1.018$$
 [if female] × 1.159 [if black]

where:

- Scr is serum creatinine in mg/dL (serum creatinine in µmol/L should be divided by 88.4)
- $\kappa$  is 0.7 for females and 0.9 for males
- $\alpha$  is -0.329 for females and -0.411 for males
- min indicates the minimum of Scr/κ or 1
- max indicates the maximum of Scr/κ or 1
- For calculation of eGFR in Asian population of patients (except Japanese patients), the Asian-modified CKD-EPI (aCKD-EPI) equation will be used (7):
  - Female and SCr  $\leq$  0.7: 151 × (SCr / 0.7)<sup>-0.328</sup> × (0.993) <sup>Age</sup>
  - Female and SCr > 0.7:  $151 \times (SCr / 0.7)^{-1.210} \times (0.993)^{Age}$
  - Male and SCr  $\leq$  0.9: 149 × (SCr / 0.9)<sup>-0.412</sup> × (0.993) Age
  - Male and SCr > 0.9:  $149 \times (SCr / 0.9)^{-1.210} \times (0.993)^{Age}$
- For calculation of eGFR in Japanese patients, CKD-EPI Study equation multiplied by a Japanese coefficient of 0.813 will be used (8).

#### 2.5.2 Data handling conventions for secondary efficacy variables

## Handling of PD medications

- Dose of a PD medication at baseline will be defined as the dose received the day of randomization in Part 2
- In case of overlap between dates of intake of two or more PD medications with the same WHO-DD standardized medication name, the sum of doses will be calculated during the overlapping period
- Increase or decrease of the dose compared to the dose received at baseline will be determined by comparing the doses of PD medications with the same WHO-DD standardized medication name.

## 2.5.3 Missing data

For categorical variables, patients with missing data are not included in calculations of percentages unless otherwise specified. When relevant, the number of patients with missing data is presented.

## Handling of computation of treatment duration if investigational medicinal product end of treatment date is missing

For the calculation of the treatment duration, the date of the last dose of IMP is equal to the date of last administration reported on the end-of-treatment case report form page. If this date is missing, the exposure duration should be left as missing.

The last dose intake should be clearly identified in the case report form and should not be approximated by the last returned package date.

#### Handling of medication missing/partial dates

No imputation of medication start/end dates or times will be performed. If a medication date or time is missing or partially missing and it cannot be determined whether it was taken prior or concomitantly, it will be considered a prior, concomitant, and posttreatment medication.

#### Handling of adverse events with missing or partial date/time of onset

Missing or partial AE onset dates and times will be imputed so that if the partial AE onset date/time information does not indicate that the AE started prior to treatment or after the TEAE period, the AE will be classified as treatment-emergent. No imputation of AE end dates/times will be performed. These data imputations are for categorization purpose only and will not be used in listings. No imputation is planned for date/time of AE resolution.

## Handling of adverse events when date and time of first investigational medicinal product administration is missing

When the date and time of the first IMP administration is missing, all AEs that occurred on or after the day of randomization should be considered as TEAEs. The exposure duration should be kept as missing.

The last dose intake should be clearly identified in the case report form and should not be approximated by the last returned package date.

# Handling of missing assessment of relationship of adverse events to investigational medicinal product

If the assessment of the relationship to IMP is missing, then the relationship to IMP has to be assumed and the adverse event considered as such in the frequency tables of possibly related adverse events, but no imputation should be done at the data level.

#### Handling of missing severity of adverse events

If the severity is missing for 1 of the treatment-emergent occurrences of an AE, the maximal severity on the remaining occurrences will be considered. If the severity is missing for all the occurrences, a "missing" category will be added in the summary table.

#### Handling of potentially clinically significant abnormalities

If a patient has a missing baseline he will be grouped in the category "normal/missing at baseline."

For PCSAs with 2 conditions, one based on a change from baseline value or a normal range and the other on a threshold value, with the first condition being missing, the PCSA will be based only on the second condition.

For a PCSA defined on a threshold and/or a normal range, this PCSA will be derived using this threshold if the normal range is missing; eg, for eosinophils the PCSA is >0.5 GIGA/L or >ULN if ULN  $\geq$ 0.5 GIGA/L. When ULN is missing, the value 0.5 should be used.

Measurements flagged as invalid by the laboratory will not be summarized or taken into account in the computation of PCSA values.

#### 2.5.4 Windows for time points

Data analyzed by time point (including efficacy, laboratory safety data, ECG, vital signs, quality of life and PK concentration) will be summarized using the analysis windows given in Table 3, Table 4, Table 5, Table 6 and Table 7). These analysis windows will be applicable for all analyses, and they are defined to provide more homogeneous data for time point-specific analyses.

For efficacy and quality of life endpoints, D1 will be defined as the day of randomization. For safety endpoints, D1 will be defined as the day of first IMP intake. In Part1, in case of treatment interruption of at least 7 days (corresponding to approximately 5 half-lives) between the day of first IMP intake and subsequent IMP intakes, D1 will be defined as the day of IMP resumption after treatment interruption (both for efficacy and safety endpoints).

Table 3 - Analysis windows definition for Part 1 - All endpoints except ECG and PK

| Time point | Targeted study day | Analysis window in study days |
|---------------------|--------------------|-------------------------------|
| Week 0 / Day 2 | D2 | D2 |
| Week 0 / Day 3 | D3 | D3 |
| Week 2 | D15 | D8 to D21 |
| Week 4 <sup>a</sup> | D29 | D22 to D42 |
| Week 8 | D57 | D43 to D70 |
| Week 12 | D85 | D71 to D98 |
| Week 16 | D113 | D99 to D126 |
| Week 20 | D141 | D127 to D154 |
| Week 24 | D169 | D155 to D182 |
| Week 28 | D197 | D183 to D210 |
| Week 32 | D225 | D211 to D238 |
| Week 36 | D253 | D239 to D266 |
| Week 40 | D281 | D267 to D294 |
| Week 44 | D309 | D295 to D322 |
| Week 48 | D337 | D323 to D350 |
| Week 52 | D365 | D351 to D378 |

a For vital signs, any data collected between D22 and D42 will be further assigned to analysis window "Week 4 / Day 1" or "Week 4 / Day 2" as per eCRF page.

Table 4 - Analysis windows definition for Part 1 - ECG

| Time point | Target study day | Analysis window |
|---|---|---|
| Day 1 / Pre-dose | Day 1 / Pre-dose | Before Week 0/Day 1 dose |
| Day 1 / 2 hours post dose | Day 1 / 2 hours post dose | 1h to 2h59 after Week 0/Day 1 dose |
| Day 1 / 4 hours post dose | Day 1 / 4 hours post dose | 3h to 4h59 post-dose after Week 0/Day 1 dose |
| Day 1 / 6 hours post dose | Day 1 / 6 hours post dose | 5h to 8h post-dose Week 0/Day 1 dose |
| Week 4 | D29 | D22 to D42 |
| Week 28 | D197 | D183 to D210 |

Table 5 - Analysis windows definition for Part 1 - PK concentration

| Time point | Target study day | Analysis window |
|---|---|---|
| Day 1 / Pre-dose | Day 1 / Pre-dose | Before Week 0/Day 1 dose |
| Day 1 / 1 hour post dose | Day 1 / 1 hour post dose | 0h50 to 1h10 after Week 0/Day 1 dose |
| Day 1 / 2 hours post dose | Day 1 / 2 hours post dose | 1h45 to 2h15 after Week 0/Day 1 dose |
| Day 1 / 4 hours post dose | Day 1 / 4 hours post dose | 3h30 to 4h30 after Week 0/Day 1 dose |
| Day 1 / 8 hours post dose | Day 1 / 8 hours post dose | 7h00 to 9h00 after Week 0/Day 1 dose |
| Day 2 / 24 hours post dose | Day 2 / 24 hours post dose | 23h00 to 25h00 after Week 0/Day 1 dose |
| Day 3 / 48 hours post dose | Day 3 / 48 hours post dose | 46h00 to 50h00 after Week 0/Day 1 dose and before Week 0/Day 3 dose |
| Week 2 / Pre-dose | D15 / Pre-dose | Week 2 - Before Week 2 dose |
| Week 4 / Pre-dose | D29 / Pre-dose | Week 4 - Before Week 4 / Day 1 dose |
| Week 4 / 1 hour post dose | D29 / 1 hour post dose | Week 4/Day 1 - 0h50 to 1h10 after Week 4/Day<br>1 dose |
| Week 4 / 2 hours post dose | D29 / 2 hours post dose | Week 4/Day 1 - 1h45 to 2h15 after Week 4/Day<br>1 dose |
| Week 4 / 4 hours post dose | D29 / 4 hours post dose | Week 4/Day 1 - 3h30 to 4h30 after Week 4/Day<br>1 dose |
| Week 4 / 8 hours post dose | D29 / 8 hours post dose | Week 4/Day 1 - 7h00 to 9h00 after Week 4/Day 1 dose |
| Week 4 / 24 hours post dose | D29 / 24 hours post dose | Week 4/Day 2 - 23h00 to 25h00after Week<br>4/Day 1 dose |
| Week 8 / Pre-dose | D57 / Pre-dose | Week 8 - Before Week 8 dose |

Table 6 - Analysis windows definition for Part 2 - All endpoints except PK

| Time point | Targeted study day | Analysis window in study<br>days |
|----------------|--------------------|----------------------------------|
| Week 0 / Day 2 | D2 | D2 |
| Week 2 | D15 | D8 to D21 |
| Week 4 | D29 | D22 to D60 |
| Week 13 | D92 | D61 to D137 |
| Week 26 | D183 | D138 to D228 |
| Week 39 | D274 | D229 to D319 |
| Week 52 | D365 | D320 to D570 <sup>a</sup> |
| Week 78 | D547 | D457 to D638 <sup>a</sup> |
| Week 104 | D730 | D639 to D820 |
| Week 130 | D911 | D821 to D1002 |
| Week 156 | D1095 | D1003 to D1184 |

a In case a measurement can be assigned to both Week 52 and Week 78 time-points, the measurement will be assigned to the time-point corresponding to the visit where the measurement was

Table 7 - Analysis windows definition for Part 2 - PK concentration

| Time point | Target study day | Analysis window |
|---|---|---|
| Day 1 / Pre-dose | Day 1 / Pre-dose | Before Week 0/Day 1 dose |
| Day 1 / 1 hour post dose | Day 1 / 1 hour post dose | 0h50 to 1h10 after Week 0/Day 1 dose |
| Day 1 / 2 hours post dose | Day 1 / 2 hours post dose | 1h45 to 2h15 after Week 0/Day 1 dose |
| Day 1 / 4 hours post dose | Day 1 / 4 hours post dose | 3h30 to 4h30 after Week 0/Day 1 dose |
| Day 1 / 8 hours post dose | Day 1 / 8 hours post dose | 7h00 to 9h00 after Week 0/Day 1 dose |
| Day 2 / 24 hours post dose | Day 2 / 24 hours post dose | 23h00 to 25h00 after Week 0/Day 1 dose |
| Week 2 / Pre-dose | D15 / Pre-dose | Week 2 - Before Week 2 dose |
| Week 26 / Pre-dose | D183 / Pre-dose | Week 26 - Before Week 26 / Day 1 dose |
| Week 26 / within 2 to 4 hours post dose | D183 / within 2 to 4 hours post dose | Week 26/Day 1 - 1h45 to 4h30 after Week<br>26/Day 1 dose |
| Week 52 / Pre-dose | D365 / Pre-dose | Week 52 - Before Week 52 / Day 1 dose |
| Week 52 / within 2 to 4 hours post dose | D365 / within 2 to 4 hours post dose | Week 52/Day 1 - 1h45 to 4h30 after Week<br>52/Day 1 dose |

If multiple valid values of a variable exist within an analysis window, the value collected at the scheduled visit will be used if within the analysis window. Otherwise the nearest from the targeted study day or time will be selected. If the difference is a tie, the value after the targeted study day or time will be used

For all endpoints except ECG at Day 1 and PK, if multiple valid values of a variable exist within a same day, then the first value of the day will be selected when time is available, else the scheduled visit will be selected.

#### 2.5.5 Unscheduled visits

For all analyses, unscheduled visit measurements may be used to provide a measurement for a time point, a baseline, if appropriate according to their definitions.

### 2.5.6 Pooling of centers for statistical analyses

Not Applicable.

#### 2.5.7 Statistical technical issues

Not Applicable.

## 2.5.8 Pharmacokinetic analysis

For ease of presentation, mean values will be arithmetic mean unless specified. Concentration values below the plasma assay limit will be treated as zero in calculating mean values. Mean values below LLOQ will be reported as LLOQ in the tables and not plotted in the figures if after C<sub>max</sub>. Mean calculations and their associated statistics will be generated from unrounded numbers and may differ slightly from those values that would be determined using the rounded numbers displayed in the tables. Values expressed in all tables will be for ease of presentation and will not be meant to imply accuracy to more than 3 significant figures.

AUC values extrapolated by more than 30% will be excluded from any pharmacokinetic statistical analysis.

Plasma concentrations and pharmacokinetic parameters of GZ402671 will be summarized by arithmetic mean, geometric mean, SD, SEM, coefficient of variation (CV (%)), minimum, median, maximum, and number of observations by treatment group using PKDMS (in-house software) Version 3.1 with Phoenix WinNonlin Professional, Version 8.1.

## 3 INTERIM ANALYSIS

Different data review and interim analyses will be performed during the conduct of Part 1 of the study.

#### 3.1 INTERNAL DATA REVIEW PRIOR TO DOSE ESCALATION IN PART 1

An internal review committee will perform safety data review after the completion of 4 weeks of dosing in all patients from non-Japanese Cohort 1 prior to dosing of the subsequent cohort; the same process will be repeated after the completion of 4 weeks of dosing in all non-Japanese patients in Cohort 2. Review of blinded safety data from Japanese patients in Cohort 1 and Cohort 2 will follow the same process and will be performed separately. Specifically, the internal review committee will review the AE/SAE data and other available individual patient safety data from all the patients in each cohort in a blinded fashion. No additional dose escalations will occur above the highest proposed dose of 15mg. No dose escalation may occur until the last patient in a given cohort has completed 4 weeks of administration of IMP.

#### 3.2 INTERNAL DATA REVIEW AT THE END OF PART 1 NON-JAPAN

An internal review committee (IRC) will review in an un-blinded fashion the following aggregated data from Part 1 in non-Japanese patients before Part 2 can occur:

- Safety:
  - AEs
  - laboratory results
  - ECG
  - Vital signs
  - Examinations (neurological, ophthalmologic, physical)
- Pharmacodynamics:
  - CSF GL-1
- Pharmacokinetic:
  - CSF parameters: Week 4 concentration at any time within 2 to 4 hours after administration of GZ/SAR402671)
  - (Optional) Plasma parameters: C<sub>trough</sub>, C<sub>max</sub>, AUC<sub>0-24</sub>

Only descriptive statistics for the above safety, pharmacodynamics and PK parameters will be prepared and reviewed by the IRC.

This committee will also select the dose for Part 2. The analysis and review for non-Japanese patients will be performed when all non-Japanese patients in Part 1 have completed 4 weeks of dosing and will not wait for patients in Japan to complete Part 1 in order to proceed to Part 2.

To protect the overall integrity of this study, specific steps will be taken to maintain the blind of the study to all those involved in the conduct of the study and/or the data review. These steps are described in Appendix K.

#### 3.3 INTERNAL DATA REVIEW AT THE END OF PART 1 JAPAN

The internal review committee will review blinded TEAE/SAEs and other available individual patient safety data from all the Japanese patients before Part 2 can start in Japan. This committee will also assess PK similarity between Japanese and non-Japanese patients. PK similarity between Japanese and non Japanese will be determined based on PK data available by the time all patients have completed 4 weeks of treatment. The data review will occur when all Japanese patients from Part1 have completed the first 4 week course of therapy.

PK similarity between Japanese and non-Japanese patients will be assessed by an independent unblinded pharmacokineticist:

- Venglustat Plasma PK parameters (Day 1 and week 4) Cmax and AUC0-24 and/or AUC0-48 as applicable will be determined using non compartmental analysis of observed plasma concentrations and nominal time data. The mean (and range) values of these parameters will be compared with the corresponding values obtained previously for Part-1 ROW data
- Venglustat CSF concentrations (mean and range at week 4) will be determined for Japanese patients and compared with the corresponding values obtained previously for Part-1 ROW data

Additional details are provided in Appendix K.

## 3.4 ANALYSIS OF PART 1 (NON-JAPAN) AND PART 1 (JAPAN)

An analysis of Part 1 (non-Japan) data will be conducted when all non-Japanese patients from part 1 have completed Part 1 of the study, and have their data collected and validated. This analysis will be done after a two-step database lock (see Section 5).

An analysis of Part 1 (Japan) data will be conducted when all Japanese patients from part 1 have completed Part 1 of the study, and have their data collected and validated. This analysis will be done after a two-step database lock (see Section 5).

These analyses will provide safety, PK, pharmacodynamics and efficacy data from Part 1 for the purpose of publication.

This analysis of Part 1 will have no impact on the statistical analysis of Part 2, since patients from Part 1 will not be included in the primary analysis of Part 2. In addition, patients from Part 1 who may also participate to Part 2 will be re-randomized when entering in Part 2, and will be described separately.

#### 3.5 GENERAL CONVENTIONS FOR INTERIM ANALYSES

Analyses methods and conventions described in the other sections of this SAP will be applied for all data reviews and interim analyses as applicable. The following additional rules will apply for data reviews and interim analyses:

- Patients without end of treatment visit performed at the time of the cut-off date will be considered as ongoing and exposed up to the cut-off date. Therefore:
  - Patients who did not complete treatment period nor prematurely discontinued the study treatment at cut-off date will be analyzed as "ongoing" in the disposition summary
  - Their TEAE period, treatment period and on-study observation period will end at the cut-off date
  - Their treatment duration will be derived by considering date of cut-off as last IMP dose date
- Analyses of compliance will be performed up to the last IMP dose reported in the e-CRF up to the cut-off date
- AEs occurring, worsening or becoming serious after the cut-off date will not be included in the analyses. However, any available outcome of an adverse event starting prior to the cut-off date will be taken into account, including outcomes posterior to the cut-off date
- Any safety assessment (including physical examination, neurological examination, ophthalmological examination, clinical laboratory evaluations, vital signs, ECG) performed after the cut-off date will not be included in the analyses
- Medications, treatment discontinuations/completions and deaths occurring after the cut-off date will not be included in the analyses
- Post-treatment period, post-study period are not applicable for ongoing patients. Analyses of post-treatment AEs, post-study deaths and post-treatment medications will be performed for patients who either completed or prematurely discontinued the treatment before or at the cut-off date
- Patients will be considered alive at the cut-off date, unless death before the cut-off date has been reported

## 4 FINAL ANALYSIS

The final analysis will be conducted in two steps:

- First step: analysis of the 52-week blinded treatment period of Part 2 of the study:
  - The analysis of the 52-week double-blind treatment period of Part 2 of the study will be conducted when all patients from Part 2 have been randomized and have all their data up to Week 52 collected and validated, and will consist in the final analysis of the primary, secondary, and exploratory endpoints up to Week 52. The cut-off date for this first step analysis will be defined as the date the last patient from Part 2 completes the Week 52 visit of the double-blind treatment period. Efficacy data collected after the Week 52 visit will not be included in this analysis. The safety analysis will be performed on all safety data collected and validated at the cut-off date of the first step analysis, including safety data collected after the Week 52 visit, but before the cut-off date. This analysis will be conducted after a partial database lock and treatment unblinding.
- Second step: analysis up to Week 156 of Part 2 of the study:
  - The second analysis will be conducted at the end of the study and will consist of the final analysis up to Week 156. This analysis will be conducted after the final database lock.

## 5 DATABASE LOCK

A snapshot of the database will be provided for internal data review (see Section 3.2). Data will continue to be added, updated or deleted after the internal data review.

A two-step database lock will be done for the analysis of Part 1 (non-Japan) described in Section 3.4:

- The first database lock will include all eCRF data as well as external data available at the time of this first database lock (including laboratory data, ECG data, PK data, pharmacodynamics data) on all patients in Part 1 (non-Japan). This database lock is planned to be done approximately 9 weeks after the last patient last visit in Part 1 (non-Japan)
- A second database lock will include the remaining external data (including slit lamp, DNA, imaging) that will not be available in the first database lock

Treatment will be unblinded for analysis safety, efficacy, PK and pharmacodynamics data after the first database lock.

A two-step database lock will be done for the analysis of Part 1 (Japan) described in Section 3.4:

- The first database lock will include all eCRF data as well as external data available at the time of this first database lock (including laboratory data, ECG data, PK data, pharmacodynamics data) on all patients in Part 1 (Japan). This database lock is planned to be done approximately
  - 9 weeks after the last patient last visit in Part 1 (Japan)
- A second database lock will include the remaining external data (including slit lamp, DNA, imaging) that will not be available in the first database lock

Treatment will be unblinded for analysis safety, efficacy, PK and pharmacodynamics data after the first database lock.

A two-step database lock will be done for the analysis of Part 2:

- A partial database lock and treatment unblinding will be done when all patients from Part 2 have been randomized and have all their data up to Week 52 collected and validated in order to perform the analysis of the 52-week blinded treatment period of Part 2. The cutoff date for this first step analysis will be defined as the date the last patient from Part 2 completes the Week 52 visit of the double-blind treatment period.
- A final database lock will be done when all patients from Part 2 have been randomized and have all their data up to Week 156 collected and validated in order to perform the final analysis of the end of the study.

## **6 SOFTWARE DOCUMENTATION**

All summaries and statistical analyses will be generated using SAS version 9.4 or higher.

## 7 REFERENCES

- 1. Chew E, Kim J, Sperduto R, Datiles III B, Coleman H, Thompson D et al. Evaluation of the Age-Related Eye Disease Study Clinical Lens Grading System AREDS Report No. 31. Ophthalmology. 2010;117(11): 2112–9.
- 2. O'Kelly M, Ratitch B. Clinical Trials with Missing Data: A Guide for Practitioners. Chichester: John Wiley & Sons. 2014. Chapter 7, Section 7.3.5.
- 3. Kenward MG. Controlled multiple imputation methods for sensitivity analyses in longitudinal clinical trials with dropout and protocol deviation. Clin. Invest. 2015;5(3), 311–320.
- 4. Roger J. Gaussian Repeated Measures with conjugate priors fitted using proc MCMC in SAS, available at https://missingdata.lshtm.ac.uk/2017/04/05/gaussian-repeated-measures-with-conjugate-priors-fitted-using-proc-mcmc-in-sas, accessed 17 July 2018.
- 5. Makkos A, Kovács M, Aschermann Z, et al. Are the MDS-UPDRS-Based Composite Scores Clinically Applicable?. Mov Disord. 2018;33(5):835-839.
- 6. Levey AS, Steven LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, et al. A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009;150(9):604-12.
- 7. Hongwei Ji et al. GFRs from Asian-modified CKD-EPI and Chinese-modified CKD-EPI equations were associated better with hypertensive target organ damage in the communitydwelling elderly Chinese: the Northern Shanghai Study. Clin Interv Aging. 2017;12:1297-308.
- 8. Horio M, Imai E, Yasuda Y, Watanabe T, Matsuo S, et al. Modification of the CKD epidemiology collaboration (CKD-EPI) equation for Japanese: accuracy and use for population estimates. Am J Kidney Dis. 2010;56(1):32-8.
- 9. Goetz CG, Luo S, Wang L, Tilley BC, LaPerre NR, Stebbins GT. Handling Missing Values in the MDS-UPDRS. Mov Disord. 2015;30(12):1632-8.
- 10. Kammerman LA, Cappelleri J, Bartlett J. Patient-Reported Outcomes. Wiley StatsRef: Statistics Reference Online 2017. DOI: 10.1002/9781118445112.stat07929; Sloan JA, Dueck AC, Erikson PA et al. Analysis and Interpretation of Results Based on Patient-Reported Outcomes. Value in Health. 2007;10(2):S106-S115.
#### 8 LIST OF APPENDICES

Appendix A: Potentially clinically significant abnormalities (PCSA) criteria

Appendix B: List of common GBA mutations

Appendix C: MDS-UPDRS scoring algorithm

Appendix D: PD-CRS scoring algorithm

Appendix E: MoCA scoring algorithm

Appendix F: BDI-II scoring algorithm

Appendix G: PDQ-39 scoring algorithm

Appendix H: EQ-5D scoring algorithm

Appendix I: Falls Efficacy Scale scoring algorithm

Appendix J: Health Related Productivity Questionnaire - scoring algorithm

Appendix K: Analysis procedure for internal data review and interim analysis

### Appendix A Potentially clinically significant abnormalities (PCSA) criteria

#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

for Phase 2/3 studies (oncology excepted) (From BTD-009536 - Version 3.0 -24-MAY-2014)

| Parameter | PCSA | Comments |
|---|---|---|
| Clinical Chemis | try | |
| ALT | By distribution analysis : >3 ULN >5 ULN >10 ULN >20 ULN | Enzymes activities must be expressed in ULN, not in IU/L. Concept paper on DILI – FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. Categories are cumulative. First row is mandatory. Rows following one mentioning zero can be deleted. |
| AST | By distribution analysis : >3 ULN >5 ULN >10 ULN >20 ULN | Enzymes activities must be expressed in ULN, not in IU/L. Concept paper on DILI – FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. Categories are cumulative. First row is mandatory. Rows following one mentioning zero can be deleted. |
| Alkaline<br>Phosphatase | >1.5 ULN | Enzymes activities must be expressed in ULN, not in IU/L. Concept paper on DILI – FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. |
| Total Bilirubin | >1.5 ULN<br>>2 ULN | Must be expressed in ULN, not in µmol/L or mg/L. Categories are cumulative. Concept paper on DILI – FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. |
| Conjugated Biliru | ıbin >35% Total Bilirubin and TBILI>1.5 ULN | Conjugated bilirubin dosed on a case-by-case basis. |
| ALT and Total<br>Bilirubin | ALT>3 ULN and TBILI>2 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. To be counted within a same treatment phase, whatever the interval between measurement. |

for Phase 2/3 studies (oncology excepted)

(From BTD-009536 - Version 3.0 -24-MAY-2014)

| Parameter | PCSA | Comments |
|---|---|---|
| СРК | >3 ULN | FDA Feb 2005. |
| | >10 ULN | Am J Cardiol April 2006. |
| | | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| CLcr (mL/min) | <15 (end stage renal disease) | FDA draft Guidance 2010 |
| (Estimated | ≥15 - <30 (severe decrease in GFR) | Pharmacokinetics in patients with impaired renal |
| based on the | 2 ≥30 - < 60 (moderate decrease in GFR) | function-study design, data analysis, and impact on dosing and labeling |
| Cockcroft-Gault | ≥60 - <90 (mild decrease in GFR) | |
| equation) | ≥ 90 (normal GFR) | |
| eGFR | <15 (end stage renal disease) | FDA draft Guidance 2010 |
| (mL/min/1.73m2)<br>(Estimate of GFR | ≥15 - <30 (severe decrease in GFR) | Pharmacokinetics in patients with impaired renal function-study design, data analysis, and impact on |
| based on an MDRD | ≥30 - < 60 (moderate decrease in GFR) | dosing and labeling |
| equation) | ≥60 - <90 (mild decrease in GFR)<br>≥ 90 (normal GFR) | |
| 0 " " | , | |
| Creatinine | ≥150 µmol/L (Adults) | Benichou C., 1994. |
| | ≥30% change from baseline<br>≥100% change from baseline | |
| | 2 100 % Change norn baseline | |
| Uric Acid | > 400 ···· = 1// | Harrison- Principles of internal Medicine 17th Ed., 2008. |
| Hyperuricemia | >408 μmol/L<br><120 μmol/L | |
| Hypouricemia | · | |
| Blood Urea<br>Nitrogen | ≥17 mmol/L | |
| Chloride | <80 mmol/L | |
| | >115 mmol/L | |
| Sodium | ≤129 mmol/L | |
| | ≥160 mmol/L | |
| Potassium | <3 mmol/L | FDA Feb 2005. |
| | ≥5.5 mmol/L | |
| Total Cholesterol | ≥7.74 mmol/L | Threshold for therapeutic intervention. |
| Triglycerides | ≥4.6 mmol/L | Threshold for therapeutic intervention. |
| Lipasemia | ≥3 ULN | |
| Amylasemia | ≥3 ULN | |

for Phase 2/3 studies (oncology excepted) (From BTD-009536 - Version 3.0 -24-MAY-2014)

| Parameter | PCSA | Comments |
|---|---|---|
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | ADA Jan 2008. |
| HbA1c | >8% | |
| Albumin | ≤25 g/L | |
| CRP | >2 ULN or >10 mg/L (if ULN not provided) | FDA Sept 2005. |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L (Black) | Increase in WBC: not relevant. |
| | ≥16.0 Giga/L | To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-induced |
| | | blood cytopenias, 1991. |
| | | FDA criteria. |
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17th Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female) | Criteria based upon decrease from baseline are more |
| | ≥185 g/L (Male); ≥165 g/L (Female) | relevant than based on absolute value. Other categories for decrease from baseline can be used |
| | Decrease from Baseline ≥20 g/L | (≥30 g/L, ≥40 g/L, ≥50 g/L). |
| | • | |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female) | |
| | ≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | |
| RBC | ≥6 Tera/L | Unless specifically required for particular drug development, the analysis is redundant with that of Hb. |
| | | Otherwise, consider FDA criteria. |
| | 100 0: " | |
| Platelets | <100 Giga/L | International Consensus meeting on drug-induced blood cytopenias, 1991. |
| | ≥700 Giga/L | 2.000 of opolitios, 100 i. |

for Phase 2/3 studies (oncology excepted)

(From BTD-009536 - Version 3.0 -24-MAY-2014)

| Parameter | PCSA | Comments |
|---|---|---|
| Urinalysis | | |
| pH | ≤4.6 | |
| | ≥8 | |
| Vital signs | | |
| HR | ≤50 bpm and decrease from baseline ≥20 bpm<br>≥120 bpm and increase from baseline≥20 bpm | To be applied for all positions (including missing) except STANDING. |
| SBP | ≤95 mmHg and decrease from baseline ≥20mmHg<br>≥160 mmHg and increase from baseline ≥20 mmHg | To be applied for all positions (including missing) except STANDING. |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg<br>≥110 mmHg and increase from baseline ≥10 mmHg | To be applied for all positions (including missing) except STANDING. |
| Orthostatic<br>Hypotension<br>Orthostatic SDB<br>Orthostatic DBP | ≤-20 mmHg<br>≤-10 mmHg | |
| Weight | ≥5% increase from baseline<br>≥5% decrease from baseline | FDA Feb 2007. |

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 - Version 3.0 -24-MAY-2014)

| Parameter | PCSA | Comments |
|---|---|---|
| ECG | | Ref.: ICH E14 guidance (2005) and E14 Q&A (2012), and Cardiac Safety Research Consortium White Paper on PR and QRS (Nada et al. Am Heart J. 2013; 165(4) : 489-500) |
| HR | <50 bpm<br><50 bpm and decrease from baseline ≥20 bpm<br><40 bpm<br><40 bpm and decrease from baseline ≥20 bpm<br><30 bpm<br><30 bpm and decrease from baseline ≥20 bpm | Categories are cumulative |
| | >90 bpm >90 bpm and increase from baseline ≥20bpm >100 bpm >100 bpm and increase from baseline ≥20bpm >120 bpm >120 bpm and increase from baseline ≥20 bpm | Categories are cumulative |
| PR | >200 ms >200 ms and increase from baseline ≥25% > 220 ms >220 ms and increase from baseline ≥25% > 240 ms > 240 ms > 240 ms and increase from baseline ≥25% | Categories are cumulative |
| QRS | >110 ms<br>>110 msec and increase from baseline ≥25%<br>>120 ms<br>>120 ms and increase from baseline ≥25% | Categories are cumulative |
| QT | >500 ms | |
| QTc | Absolute values (ms) | To be applied to any kind of QT correction formula. Absolute values categories are cumulative |
| | >450 ms<br>>480 ms<br>>500 ms | QTc >480 ms and $\Delta$ QTc>60 ms are the 2 PCSA categories to be identified in individual subjects/patients listings. |
| | Increase from baseline Increase from baseline ]30-60] ms Increase from baseline >60 ms | |

### Appendix B List of common GBA mutations

Note: If the patient has a GBA mutation that is not on the list, a consult will always be required to determine the eligibility of the patient and severity of the novel variant.

| Category | Allele Name | cDNA nucleotide substitution | Amino Acid substitution |
|---|---|---|---|
| Severe GBA Mutations | Frameshifts | 1 | 1 |
| | 122CC | 122insC | Arg41ProfsX6 |
| | 148-149insGTAT | 148-149insGTAT | Tyr50CysfsX15 |
| | 203Cdel | 203delC | Pro68ArgfsX23 |
| | 329–333del CAGAA | 329–333del CAGAA | Not determined |
| | 330delA | 330delA | Glu111AsnfsX7 |
| | 413delC | 413delC | Pro138LeufsX62 |
| | 493insA | 493insA | Not determined |
| | 500insT | 500insT | Ser168LeufsX12 |
| | 532delC | 532delC | Not determined |
| | 534delT | 534delT | Asp179MetfsX21 |
| | 595-596delCT | 595_596delCT | Leu199AspfsX62 |
| | 72delC | 72delC | Leu25SerfsX66 |
| | V214Stop | 741delC | Trp248GlyfsX6 |
| | 84GG | 84dupG | Leu29AlafsX18 |
| | 898delG | 898delG | Ala300ProfsX4 |
| | 914Cdel | 914delC | Pro305LeufsX31 |
| | 953delT | 953delT | Leu318ProfsX18 |
| | Tyr343Stop | 1029delT | Tyr343X |
| | 1093-1094insG | 1093dupG | Glu365GlyfsX71 |
| | 1098insA | 1098dupA | His367ThrfsX69 |
| | 1122-1123insTG | 1121_1122dupTG | Leu375CysfsX20 |
| | 1147delG | 1147delG | Not determined |
| | 119delC | 119delC | Not determined |
| | 1214delGC | 1214_1215delGC | Ser405AsnfsX30 |
| | 1263–1317del | 1263–1317del | Not determined |
| | 1284delA | 1284delA | GlyAspfsX15 |
| | 1326insT | 1326dupT | Val443CysfsX26 |
| | 1447-1466del20,insTG | 1447_1466delinsTG | Leu483_Met489delinsTrp |

| Category | Allele Name | cDNA nucleotide<br>substitution | Amino Acid substitution |
|---|---|---|---|
| | Substitutions | | |
| | A190T | 685G>A | Ala229Thr |
| | A190E | 686C>A | Ala229Glu |
| | A341T | 1138G>A | Ala380Thr |
| | A456P | 1483G > C | Ala495Pro |
| | C16S | 164G > C | Cys55Ser |
| | C342Y | 1142G>A | Cys381Tyr |
| | D380A | 1256A>C | Asp419Ala |
| | D399N | 1312G>A | Asp438Asn |
| | D409H | 1342G > C | Asp448His |
| | D409V | 1343A>T | Asp448Val |
| | E41K | 238G>A | Glu80Lys |
| | E233Stop | 814G>T | Glu272X |
| | E388Stop | 1279G>T | Glu427X |
| | F213I | 754T > A | Phe252lle |
| | F251L | 870C>A | Phe290Leu |
| | G195E | 701G>A | Gly234Glu |
| | G195W | 700G>T | Gly234Trp |
| | G202R | 721G > A | Gly241Arg |
| | G325R | 1090G > A | Gly364Arg |
| | G355D | 1181G>A | Gly394Asp |
| | G389E | 1283G>A | Gly428Glu |
| | G390R | 1285G>A | Gly429Arg |
| | H255Q | 882T>G | His294Gln |
| | H311R | 1049A>G | His350Arg |
| | I119T | 473T > C | lle158Thr |
| | I402F | 1321A>T | lle441Phe |
| | K74Stop | 337A>T | Lys113X |
| | K157Q | 586A>C | Lys196Gln |
| | K157N | 588G>T | Lys196Asn |
| | K198E | 709A>G | Lys237Glu |
| | K425E | 1390A>G | Lys464Glu |
| | L197F | 706C>T | Leu236Phe |
| | L240P | 836T>C | Leu279Pro |

| Category | Allele Name | cDNA nucleotide substitution | Amino Acid substitution |
|---|---|---|---|
| | L385P | 1271T>C | Leu424Pro |
| | L444P | 1448T>C | Leu483Pro |
| | L444R | 1448T>G | Leu483Arg |
| | N392I | 1292A>T | Asn431lle |
| | N462K | 1503C>G | Asn501Lys |
| | P178S | 649C > T | Pro217Ser |
| | P182L | 662C > T | Pro221Leu |
| | P266L | 914C>T | Pro305Leu |
| | P415R | 1361C>G | Pro454Arg |
| | Q73Stop | 334C>T | Gln112X |
| | Q169Stop | 622C>T | Gln208X |
| | Q350Stop | 1165C>T | Gln389X |
| | Q414Stop | 1357C>T | Gln453X |
| | Q414R | 1358A>G | Gln453Arg |
| | R47Stop | 256C>T | Arg86X |
| | R120W | 475C>T | Arg159Trp |
| | R120Q | 476G > A | Arg159Gln |
| | R131C | 508C > T | Arg170Cys |
| | R131L | 509G > T | Arg170Leu |
| | R163Stop | 604C>T | Arg202X |
| | R257Q | 887G > A | Arg296Gln |
| | R257Stop | 886C>T | Arg296X |
| | R285H | 971G > A | Arg324His |
| | R353G | 1174C>G | Arg392Gly |
| | R359Stop | 1192C>T | Arg398X |
| | R463C | 1504C > T | Arg502Cys |
| | R463Q | 1505G>A | Arg502Gln |
| | S107L | 437C > T | Ser146Leu |
| | S173Stop | 635C>G | Ser212X |
| | S237P | 826T>C | Ser276Pro |
| | S364R | 1207A>C | Ser403Arg |
| | T231R | 809C>G | Thr270Arg |
| | T491I | 1589C > T | Thr530lle |
| | V394L | 1297G > T | Val433Leu |

| Category | Allele Name | cDNA nucleotide substitution | Amino Acid substitution |
|---|---|---|---|
| | V398L | 1309G>C | Val437Leu |
| | V398F | 1309G>T | Val437Phe |
| | W179Stop | 653G>A | Trp218X |
| | W(-4)Stop | 108G>A | Trp36X |
| | W378Stop | 1250G>A | Trp417X |
| | Y135Stop | 522T>A | Tyr174X |
| | Y304C | 1028A>G | Tyr343Cys |
| | Y304Stop | 1029T>G | Tyr343X |
| | 841-842insTGA | 839_841dupTGA | Leu280_Ser281insMet |
| | Splice variants | - | |
| | IVS10+2t>a | 1505+2t>a | Not determined |
| | IVS10(+2) | 1505+2t>g | Not determined |
| | IVS2+1g>a | 115+1g>a | Not determined |
| | IVS2+1g>t | 115+1g>t | Not determined |
| | (-203)a>g + IVS4-2a>g | (-203a>g; 455-2a>g) | Not determined |
| | IVS5+1g>t | 588+1g>t | Not determined |
| Other GBA Mutations | 222-224delTAC | 222_224del TAC | Thr75del |
| | A90T | 385G>A | Ala129Thr |
| | A232G | 812C>G | Ala271Gly |
| | C342G | 1141T>G | Cys381Gly |
| | C342R | 1141T>C | Cys381Arg |
| | D127V | 497A>T | Asp166Val |
| | D140H | 535G > C | Asp179His |
| | D409G | 1343A>G | Asp448Gly |
| | F37V | 226T>G | Phe76Val |
| | F216Y | 764T>A | Phe255Tyr |
| | F397S | 1307T>C | Phe436Ser |
| | G46E | 254G > A | Gly85Glu |
| | G189V | 683G > T | Gly228Val |
| | G193W | 694G>T | Gly232Trp |
| | G377S | 1246G > A | Gly416Ser |
| | G377C | 1246G>T | Gly416Cys |
| | 1402T | 1322T>C | lle441Thr |

| Category | Allele Name | cDNA nucleotide substitution | Amino Acid substitution |
|---|---|---|---|
| | K79N | 354G>C | Lys118Asn |
| | K413Q | 1354A>C | Lys452Gln |
| | L66P | 314T>C | Leu105Pro |
| | L371V | 1228C>G | Leu410Val |
| | M123V | 484A > G | Met162Val |
| | N117D | 466A > G | Asn156Asp |
| | N188R | 680_681 delinsGG | Asn227Arg |
| | N188S | 680A > G | Asn227Ser |
| | N370S | 1226A > G | Asn409Ser |
| | N396T | 1304A>C | Asn435Thr |
| | P122S | 481C>T | Pro161Ser |
| | P159L | 593C > T | Pro198Leu |
| | P159T | 592C > A | Pro198Thr |
| | P266R | 914C > G | Pro305Arg |
| | P289L | 983C>T | Pro328Leu |
| | P401L | 1319C>T | Pro440Leu |
| | R48W | 259C > T | Arg87Trp |
| | R170C | 625C>T | Arg209Cys |
| | R170P | 626G>C | Arg209Pro |
| | R359Q | 1193G>A | Arg398GIn |
| | R395C | 1300C>T | Arg434Cys |
| | R433G | 1414A>G | Arg472Gly |
| | R496C | 1603C>T | Arg535Cys |
| | R496H | 1604G>A | Arg535His |
| | S271G | 928A>G | Ser310Gly |
| | S271N | 929G>A | Ser310Asn |
| | S364T | 1208G>C | Ser403Thr |
| | S364N | 1208G>A | Ser403Asn |
| | S366G | 1213A>G | Ser405Gly |
| | T43I | 245C>T | Thr82lle |
| | T134I | 518C>T | Thr173lle |
| | T323I | 1085C>T | Thr362lle |
| | V15L | 160G>T | Val54Leu |
| | V352L | 1171G>C | Val391Leu |

15-Dec-2020 Version number: 2

| Category | Allele Name | cDNA nucleotide substitution | Amino Acid substitution |
|---|---|---|---|
| | V375L | 1240G>T | Val414Leu |
| | V375G | 1241T>G | Val414Gly |
| | W184R | 667T>C | Trp223Arg |
| | W312C | 1053G>T | Trp351Cys |
| | W378G | 1249T>G | Trp417Gly |
| Sequence variants where history of RBD or co- | E326K | 1093G>A | Glu365Lys |
| occurrence of any mutation on the list are required | Т369М | 1223C>T | Thr408Met |

Note: If the patient has a GBA mutation that is not on this list, a consult will be required to determine the eligibility of the patient. Abbreviation: cDNA: complementary deoxyribonucleic acid; GBA:  $\beta$ -glucocerebrosidase gene; RBD: rapid eye movement sleep behavior disorder.

Appendix C MDS-UPDRS scoring algorithm







15-Dec-2020 Version number: 2



## Appendix D PD-CRS scoring algorithm



# Appendix E MoCA scoring algorithm



# Appendix F BDI-II scoring algorithm





15-Dec-2020 Version number: 2





Appendix G PDQ-39 scoring algorithm





#### Appendix H EQ-5D-5L scoring algorithm

Computing EQ-5D-5L crosswalk index values with SAS using the United Kingdom (UK) value set

The variables for the 5 dimensions of the EQ-5D-5L descriptive system should be named 'mobility', 'selfcare', 'activity', 'pain', and 'anxiety'. If they are given different names the syntax code below will not work properly. The 5 variables should contain the values for the different dimensions in the EQ-5D health profile (ie, 1, 2, 3, 4 or 5). The variable 'EQindex' contains the values of the EQ-5D-5L crosswalk index values on the basis of the UK set of weights.

You can copy and paste the syntax below directly into a SAS syntax window.

```
*SAS syntax code for the computation of index*
*values with the UK TTO value set*
*******************************
data Euroqol.UK tto;
set Euroqol.EQ5D states;
EQindex = .;
if (mobility=1 and selfcare=1 and activity=1 and pain=1 and anxiety=1) then EQindex = 1.000;
if (mobility=1 and selfcare=1 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.879;
if (mobility=1 and selfcare=1 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.848;
if (mobility=1 and selfcare=1 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.635;
if (mobility=1 and selfcare=1 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.414;
if (mobility=1 and selfcare=1 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.837;
if (mobility=1 and selfcare=1 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.768;
if (mobility=1 and selfcare=1 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.750;
if (mobility=1 and selfcare=1 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.537;
if (mobility=1 and selfcare=1 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.316;
if (mobility=1 and selfcare=1 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.796;
if (mobility=1 and selfcare=1 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.740;
if (mobility=1 and selfcare=1 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.725;
if (mobility=1 and selfcare=1 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.512;
if (mobility=1 and selfcare=1 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.291;
if (mobility=1 and selfcare=1 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.584;
if (mobility=1 and selfcare=1 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.527;
if (mobility=1 and selfcare=1 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.513;
if (mobility=1 and selfcare=1 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.352;
if (mobility=1 and selfcare=1 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.186;
if (mobility=1 and selfcare=1 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.264;
if (mobility=1 and selfcare=1 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.208;
if (mobility=1 and selfcare=1 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.193;
if (mobility=1 and selfcare=1 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.112;
if (mobility=1 and selfcare=1 and activity=1 and pain=5 and anxiety=5) then EQindex = 0.028;
if (mobility=1 and selfcare=1 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.906;
if (mobility=1 and selfcare=1 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.837;
```

if (mobility=1 and selfcare=1 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.819;

```
if (mobility=1 and selfcare=1 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.606;
if (mobility=1 and selfcare=1 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.385;
if (mobility=1 and selfcare=1 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.795;
if (mobility=1 and selfcare=1 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.736;
if (mobility=1 and selfcare=1 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.721;
if (mobility=1 and selfcare=1 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.508;
if (mobility=1 and selfcare=1 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.287;
if (mobility=1 and selfcare=1 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.767;
if (mobility=1 and selfcare=1 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.711;
if (mobility=1 and selfcare=1 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.696;
if (mobility=1 and selfcare=1 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.483;
if (mobility=1 and selfcare=1 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.262;
if (mobility=1 and selfcare=1 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.555;
if (mobility=1 and selfcare=1 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.498;
if (mobility=1 and selfcare=1 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.484;
if (mobility=1 and selfcare=1 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.323;
if (mobility=1 and selfcare=1 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.157;
if (mobility=1 and selfcare=1 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.235;
if (mobility=1 and selfcare=1 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.179;
if (mobility=1 and selfcare=1 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.164;
if (mobility=1 and selfcare=1 and activity=2 and pain=5 and anxiety=4) then EQindex = 0.083;
if (mobility=1 and selfcare=1 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.001;
if (mobility=1 and selfcare=1 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.883;
if (mobility=1 and selfcare=1 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.827;
if (mobility=1 and selfcare=1 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.812;
if (mobility=1 and selfcare=1 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.599;
if (mobility=1 and selfcare=1 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.378;
if (mobility=1 and selfcare=1 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.785;
if (mobility=1 and selfcare=1 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.728;
if (mobility=1 and selfcare=1 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.714;
if (mobility=1 and selfcare=1 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.501;
if (mobility=1 and selfcare=1 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.280;
if (mobility=1 and selfcare=1 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.760;
if (mobility=1 and selfcare=1 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.704;
if (mobility=1 and selfcare=1 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.689;
if (mobility=1 and selfcare=1 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.476;
if (mobility=1 and selfcare=1 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.255;
if (mobility=1 and selfcare=1 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.548;
if (mobility=1 and selfcare=1 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.491;
if (mobility=1 and selfcare=1 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.477;
if (mobility=1 and selfcare=1 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.316;
if (mobility=1 and selfcare=1 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.150;
if (mobility=1 and selfcare=1 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.228;
if (mobility=1 and selfcare=1 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.172;
if (mobility=1 and selfcare=1 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.157;
if (mobility=1 and selfcare=1 and activity=3 and pain=5 and anxiety=4) then EQindex = 0.076;
```

```
if (mobility=1 and selfcare=1 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.008;
if (mobility=1 and selfcare=1 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.776;
if (mobility=1 and selfcare=1 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.719;
if (mobility=1 and selfcare=1 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.705;
if (mobility=1 and selfcare=1 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.535;
if (mobility=1 and selfcare=1 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.359;
if (mobility=1 and selfcare=1 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.677;
if (mobility=1 and selfcare=1 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.621;
if (mobility=1 and selfcare=1 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.606;
if (mobility=1 and selfcare=1 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.437;
if (mobility=1 and selfcare=1 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.260;
if (mobility=1 and selfcare=1 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.653;
if (mobility=1 and selfcare=1 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.596;
if (mobility=1 and selfcare=1 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.582;
if (mobility=1 and selfcare=1 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.412;
if (mobility=1 and selfcare=1 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.236;
if (mobility=1 and selfcare=1 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.475;
if (mobility=1 and selfcare=1 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.419;
if (mobility=1 and selfcare=1 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.404;
if (mobility=1 and selfcare=1 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.270;
if (mobility=1 and selfcare=1 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.131;
if (mobility=1 and selfcare=1 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.209;
if (mobility=1 and selfcare=1 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.153;
if (mobility=1 and selfcare=1 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.138;
if (mobility=1 and selfcare=1 and activity=4 and pain=5 and anxiety=4) then EQindex = 0.057;
if (mobility=1 and selfcare=1 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.027;
if (mobility=1 and selfcare=1 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.556;
if (mobility=1 and selfcare=1 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.500;
if (mobility=1 and selfcare=1 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.485;
if (mobility=1 and selfcare=1 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.404;
if (mobility=1 and selfcare=1 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.320;
if (mobility=1 and selfcare=1 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.458;
if (mobility=1 and selfcare=1 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.401;
if (mobility=1 and selfcare=1 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.387;
if (mobility=1 and selfcare=1 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.306;
if (mobility=1 and selfcare=1 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.222;
if (mobility=1 and selfcare=1 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.433;
if (mobility=1 and selfcare=1 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.377;
if (mobility=1 and selfcare=1 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.362;
if (mobility=1 and selfcare=1 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.281;
if (mobility=1 and selfcare=1 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.197;
if (mobility=1 and selfcare=1 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.328;
if (mobility=1 and selfcare=1 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.272;
if (mobility=1 and selfcare=1 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.257;
if (mobility=1 and selfcare=1 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.176;
if (mobility=1 and selfcare=1 and activity=5 and pain=4 and anxiety=5) then EQindex = 0.092;
```

```
if (mobility=1 and selfcare=1 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.170;
if (mobility=1 and selfcare=1 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.114;
if (mobility=1 and selfcare=1 and activity=5 and pain=5 and anxiety=3) then EQindex = 0.099;
if (mobility=1 and selfcare=1 and activity=5 and pain=5 and anxiety=4) then EQindex = 0.018;
if (mobility=1 and selfcare=1 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.066;
if (mobility=1 and selfcare=2 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.846;
if (mobility=1 and selfcare=2 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.779;
if (mobility=1 and selfcare=2 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.761;
if (mobility=1 and selfcare=2 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.548;
if (mobility=1 and selfcare=2 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.327;
if (mobility=1 and selfcare=2 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.737;
if (mobility=1 and selfcare=2 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.678;
if (mobility=1 and selfcare=2 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.663;
if (mobility=1 and selfcare=2 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.450;
if (mobility=1 and selfcare=2 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.229;
if (mobility=1 and selfcare=2 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.709;
if (mobility=1 and selfcare=2 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.653;
if (mobility=1 and selfcare=2 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.638;
if (mobility=1 and selfcare=2 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.425;
if (mobility=1 and selfcare=2 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.204;
if (mobility=1 and selfcare=2 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.497;
if (mobility=1 and selfcare=2 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.441;
if (mobility=1 and selfcare=2 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.426;
if (mobility=1 and selfcare=2 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.266;
if (mobility=1 and selfcare=2 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.099;
if (mobility=1 and selfcare=2 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.177;
if (mobility=1 and selfcare=2 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.121;
if (mobility=1 and selfcare=2 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.106;
if (mobility=1 and selfcare=2 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.025;
if (mobility=1 and selfcare=2 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.059;
if (mobility=1 and selfcare=2 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.806;
if (mobility=1 and selfcare=2 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.748;
if (mobility=1 and selfcare=2 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.733;
if (mobility=1 and selfcare=2 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.520;
if (mobility=1 and selfcare=2 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.299;
if (mobility=1 and selfcare=2 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.706;
if (mobility=1 and selfcare=2 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.649;
if (mobility=1 and selfcare=2 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.634;
if (mobility=1 and selfcare=2 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.421;
if (mobility=1 and selfcare=2 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.200;
if (mobility=1 and selfcare=2 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.681;
if (mobility=1 and selfcare=2 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.624;
if (mobility=1 and selfcare=2 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.610;
if (mobility=1 and selfcare=2 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.397;
if (mobility=1 and selfcare=2 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.176;
if (mobility=1 and selfcare=2 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.468;
```

```
if (mobility=1 and selfcare=2 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.412;
if (mobility=1 and selfcare=2 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.397;
if (mobility=1 and selfcare=2 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.237;
if (mobility=1 and selfcare=2 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.071;
if (mobility=1 and selfcare=2 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.149;
if (mobility=1 and selfcare=2 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.092;
if (mobility=1 and selfcare=2 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.078;
if (mobility=1 and selfcare=2 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.003;
if (mobility=1 and selfcare=2 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.088;
if (mobility=1 and selfcare=2 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.796;
if (mobility=1 and selfcare=2 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.740;
if (mobility=1 and selfcare=2 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.725;
if (mobility=1 and selfcare=2 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.512;
if (mobility=1 and selfcare=2 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.291;
if (mobility=1 and selfcare=2 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.698;
if (mobility=1 and selfcare=2 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.642;
if (mobility=1 and selfcare=2 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.627;
if (mobility=1 and selfcare=2 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.414;
if (mobility=1 and selfcare=2 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.193;
if (mobility=1 and selfcare=2 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.673;
if (mobility=1 and selfcare=2 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.617;
if (mobility=1 and selfcare=2 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.602;
if (mobility=1 and selfcare=2 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.389;
if (mobility=1 and selfcare=2 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.168;
if (mobility=1 and selfcare=2 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.461;
if (mobility=1 and selfcare=2 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.405;
if (mobility=1 and selfcare=2 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.390;
if (mobility=1 and selfcare=2 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.230;
if (mobility=1 and selfcare=2 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.063;
if (mobility=1 and selfcare=2 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.141;
if (mobility=1 and selfcare=2 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.085;
if (mobility=1 and selfcare=2 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.070;
if (mobility=1 and selfcare=2 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.011;
if (mobility=1 and selfcare=2 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.095;
if (mobility=1 and selfcare=2 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.689;
if (mobility=1 and selfcare=2 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.633;
if (mobility=1 and selfcare=2 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.618;
if (mobility=1 and selfcare=2 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.448;
if (mobility=1 and selfcare=2 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.272;
if (mobility=1 and selfcare=2 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.591;
if (mobility=1 and selfcare=2 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.534;
if (mobility=1 and selfcare=2 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.520;
if (mobility=1 and selfcare=2 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.350;
if (mobility=1 and selfcare=2 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.174;
if (mobility=1 and selfcare=2 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.566;
if (mobility=1 and selfcare=2 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.510;
```

```
if (mobility=1 and selfcare=2 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.495;
if (mobility=1 and selfcare=2 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.325;
if (mobility=1 and selfcare=2 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.149;
if (mobility=1 and selfcare=2 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.389;
if (mobility=1 and selfcare=2 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.332;
if (mobility=1 and selfcare=2 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.318;
if (mobility=1 and selfcare=2 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.184;
if (mobility=1 and selfcare=2 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.044;
if (mobility=1 and selfcare=2 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.122;
if (mobility=1 and selfcare=2 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.066;
if (mobility=1 and selfcare=2 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.051;
if (mobility=1 and selfcare=2 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.030;
if (mobility=1 and selfcare=2 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.114;
if (mobility=1 and selfcare=2 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.469;
if (mobility=1 and selfcare=2 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.413;
if (mobility=1 and selfcare=2 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.398;
if (mobility=1 and selfcare=2 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.317;
if (mobility=1 and selfcare=2 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.233;
if (mobility=1 and selfcare=2 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.371;
if (mobility=1 and selfcare=2 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.315;
if (mobility=1 and selfcare=2 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.300;
if (mobility=1 and selfcare=2 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.219;
if (mobility=1 and selfcare=2 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.135;
if (mobility=1 and selfcare=2 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.346;
if (mobility=1 and selfcare=2 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.290;
if (mobility=1 and selfcare=2 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.275;
if (mobility=1 and selfcare=2 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.194;
if (mobility=1 and selfcare=2 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.110;
if (mobility=1 and selfcare=2 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.241;
if (mobility=1 and selfcare=2 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.185;
if (mobility=1 and selfcare=2 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.170;
if (mobility=1 and selfcare=2 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.089;
if (mobility=1 and selfcare=2 and activity=5 and pain=4 and anxiety=5) then EQindex = 0.005;
if (mobility=1 and selfcare=2 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.083;
if (mobility=1 and selfcare=2 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.027;
if (mobility=1 and selfcare=2 and activity=5 and pain=5 and anxiety=3) then EQindex = 0.012;
if (mobility=1 and selfcare=2 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.069;
if (mobility=1 and selfcare=2 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.153;
if (mobility=1 and selfcare=3 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.815;
if (mobility=1 and selfcare=3 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.759;
if (mobility=1 and selfcare=3 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.744;
if (mobility=1 and selfcare=3 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.531;
if (mobility=1 and selfcare=3 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.310;
if (mobility=1 and selfcare=3 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.717;
if (mobility=1 and selfcare=3 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.660;
if (mobility=1 and selfcare=3 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.646;
```

```
if (mobility=1 and selfcare=3 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.433;
if (mobility=1 and selfcare=3 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.212;
if (mobility=1 and selfcare=3 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.692;
if (mobility=1 and selfcare=3 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.636;
if (mobility=1 and selfcare=3 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.621;
if (mobility=1 and selfcare=3 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.408;
if (mobility=1 and selfcare=3 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.187;
if (mobility=1 and selfcare=3 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.480;
if (mobility=1 and selfcare=3 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.423;
if (mobility=1 and selfcare=3 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.409;
if (mobility=1 and selfcare=3 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.248;
if (mobility=1 and selfcare=3 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.082;
if (mobility=1 and selfcare=3 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.160;
if (mobility=1 and selfcare=3 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.104;
if (mobility=1 and selfcare=3 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.089;
if (mobility=1 and selfcare=3 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.008;
if (mobility=1 and selfcare=3 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.076;
if (mobility=1 and selfcare=3 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.786;
if (mobility=1 and selfcare=3 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.730;
if (mobility=1 and selfcare=3 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.715;
if (mobility=1 and selfcare=3 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.502;
if (mobility=1 and selfcare=3 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.281;
if (mobility=1 and selfcare=3 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.688;
if (mobility=1 and selfcare=3 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.631;
if (mobility=1 and selfcare=3 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.617;
if (mobility=1 and selfcare=3 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.404;
if (mobility=1 and selfcare=3 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.183;
if (mobility=1 and selfcare=3 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.663;
if (mobility=1 and selfcare=3 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.607;
if (mobility=1 and selfcare=3 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.592;
if (mobility=1 and selfcare=3 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.379;
if (mobility=1 and selfcare=3 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.158;
if (mobility=1 and selfcare=3 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.451;
if (mobility=1 and selfcare=3 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.394;
if (mobility=1 and selfcare=3 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.380;
if (mobility=1 and selfcare=3 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.219;
if (mobility=1 and selfcare=3 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.053;
if (mobility=1 and selfcare=3 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.131;
if (mobility=1 and selfcare=3 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.075;
if (mobility=1 and selfcare=3 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.060;
if (mobility=1 and selfcare=3 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.021;
if (mobility=1 and selfcare=3 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.105;
if (mobility=1 and selfcare=3 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.779;
if (mobility=1 and selfcare=3 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.723;
if (mobility=1 and selfcare=3 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.708;
if (mobility=1 and selfcare=3 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.495;
```

```
if (mobility=1 and selfcare=3 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.274;
if (mobility=1 and selfcare=3 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.681;
if (mobility=1 and selfcare=3 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.624;
if (mobility=1 and selfcare=3 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.610;
if (mobility=1 and selfcare=3 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.397;
if (mobility=1 and selfcare=3 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.176;
if (mobility=1 and selfcare=3 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.656;
if (mobility=1 and selfcare=3 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.600;
if (mobility=1 and selfcare=3 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.585;
if (mobility=1 and selfcare=3 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.372;
if (mobility=1 and selfcare=3 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.151;
if (mobility=1 and selfcare=3 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.444;
if (mobility=1 and selfcare=3 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.387;
if (mobility=1 and selfcare=3 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.373;
if (mobility=1 and selfcare=3 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.212;
if (mobility=1 and selfcare=3 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.046;
if (mobility=1 and selfcare=3 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.124;
if (mobility=1 and selfcare=3 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.068;
if (mobility=1 and selfcare=3 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.053;
if (mobility=1 and selfcare=3 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.028;
if (mobility=1 and selfcare=3 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.112;
if (mobility=1 and selfcare=3 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.672;
if (mobility=1 and selfcare=3 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.615;
if (mobility=1 and selfcare=3 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.601;
if (mobility=1 and selfcare=3 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.431;
if (mobility=1 and selfcare=3 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.255;
if (mobility=1 and selfcare=3 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.573;
if (mobility=1 and selfcare=3 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.517;
if (mobility=1 and selfcare=3 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.502;
if (mobility=1 and selfcare=3 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.333;
if (mobility=1 and selfcare=3 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.156;
if (mobility=1 and selfcare=3 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.549;
if (mobility=1 and selfcare=3 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.492;
if (mobility=1 and selfcare=3 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.478;
if (mobility=1 and selfcare=3 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.308;
if (mobility=1 and selfcare=3 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.132;
if (mobility=1 and selfcare=3 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.371;
if (mobility=1 and selfcare=3 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.315;
if (mobility=1 and selfcare=3 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.300;
if (mobility=1 and selfcare=3 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.166;
if (mobility=1 and selfcare=3 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.027;
if (mobility=1 and selfcare=3 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.105;
if (mobility=1 and selfcare=3 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.049;
if (mobility=1 and selfcare=3 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.034;
if (mobility=1 and selfcare=3 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.047;
if (mobility=1 and selfcare=3 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.131;
```

```
if (mobility=1 and selfcare=3 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.452;
if (mobility=1 and selfcare=3 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.396;
if (mobility=1 and selfcare=3 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.381;
if (mobility=1 and selfcare=3 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.300;
if (mobility=1 and selfcare=3 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.216;
if (mobility=1 and selfcare=3 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.354;
if (mobility=1 and selfcare=3 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.297;
if (mobility=1 and selfcare=3 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.283;
if (mobility=1 and selfcare=3 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.202;
if (mobility=1 and selfcare=3 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.118;
if (mobility=1 and selfcare=3 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.329;
if (mobility=1 and selfcare=3 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.273;
if (mobility=1 and selfcare=3 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.258;
if (mobility=1 and selfcare=3 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.177;
if (mobility=1 and selfcare=3 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.093;
if (mobility=1 and selfcare=3 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.224;
if (mobility=1 and selfcare=3 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.168;
if (mobility=1 and selfcare=3 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.153;
if (mobility=1 and selfcare=3 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.072;
if (mobility=1 and selfcare=3 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.012;
if (mobility=1 and selfcare=3 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.066;
if (mobility=1 and selfcare=3 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.010;
if (mobility=1 and selfcare=3 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.005;
if (mobility=1 and selfcare=3 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.086;
if (mobility=1 and selfcare=3 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.170;
if (mobility=1 and selfcare=4 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.723;
if (mobility=1 and selfcare=4 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.667;
if (mobility=1 and selfcare=4 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.652;
if (mobility=1 and selfcare=4 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.471;
if (mobility=1 and selfcare=4 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.283;
if (mobility=1 and selfcare=4 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.624;
if (mobility=1 and selfcare=4 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.568;
if (mobility=1 and selfcare=4 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.553;
if (mobility=1 and selfcare=4 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.373;
if (mobility=1 and selfcare=4 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.185;
if (mobility=1 and selfcare=4 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.600;
if (mobility=1 and selfcare=4 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.544;
if (mobility=1 and selfcare=4 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.529;
if (mobility=1 and selfcare=4 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.348;
if (mobility=1 and selfcare=4 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.160;
if (mobility=1 and selfcare=4 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.414;
if (mobility=1 and selfcare=4 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.357;
if (mobility=1 and selfcare=4 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.343;
if (mobility=1 and selfcare=4 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.202;
if (mobility=1 and selfcare=4 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.055;
if (mobility=1 and selfcare=4 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.133;
```

```
if (mobility=1 and selfcare=4 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.077;
if (mobility=1 and selfcare=4 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.062;
if (mobility=1 and selfcare=4 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.019;
if (mobility=1 and selfcare=4 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.103;
if (mobility=1 and selfcare=4 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.694;
if (mobility=1 and selfcare=4 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.638;
if (mobility=1 and selfcare=4 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.623;
if (mobility=1 and selfcare=4 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.442;
if (mobility=1 and selfcare=4 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.254;
if (mobility=1 and selfcare=4 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.596;
if (mobility=1 and selfcare=4 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.539;
if (mobility=1 and selfcare=4 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.525;
if (mobility=1 and selfcare=4 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.344;
if (mobility=1 and selfcare=4 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.156;
if (mobility=1 and selfcare=4 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.571;
if (mobility=1 and selfcare=4 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.515;
if (mobility=1 and selfcare=4 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.500;
if (mobility=1 and selfcare=4 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.319;
if (mobility=1 and selfcare=4 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.131;
if (mobility=1 and selfcare=4 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.385;
if (mobility=1 and selfcare=4 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.328;
if (mobility=1 and selfcare=4 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.314;
if (mobility=1 and selfcare=4 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.173;
if (mobility=1 and selfcare=4 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.026;
if (mobility=1 and selfcare=4 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.104;
if (mobility=1 and selfcare=4 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.048;
if (mobility=1 and selfcare=4 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.033;
if (mobility=1 and selfcare=4 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.048;
if (mobility=1 and selfcare=4 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.132;
if (mobility=1 and selfcare=4 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.687;
if (mobility=1 and selfcare=4 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.631;
if (mobility=1 and selfcare=4 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.616;
if (mobility=1 and selfcare=4 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.435;
if (mobility=1 and selfcare=4 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.247;
if (mobility=1 and selfcare=4 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.588;
if (mobility=1 and selfcare=4 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.532;
if (mobility=1 and selfcare=4 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.517;
if (mobility=1 and selfcare=4 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.337;
if (mobility=1 and selfcare=4 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.149;
if (mobility=1 and selfcare=4 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.564;
if (mobility=1 and selfcare=4 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.508;
if (mobility=1 and selfcare=4 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.493;
if (mobility=1 and selfcare=4 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.312;
if (mobility=1 and selfcare=4 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.124;
if (mobility=1 and selfcare=4 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.378;
if (mobility=1 and selfcare=4 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.321;
```

```
if (mobility=1 and selfcare=4 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.307;
if (mobility=1 and selfcare=4 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.166;
if (mobility=1 and selfcare=4 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.019;
if (mobility=1 and selfcare=4 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.097;
if (mobility=1 and selfcare=4 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.041;
if (mobility=1 and selfcare=4 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.026;
if (mobility=1 and selfcare=4 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.055;
if (mobility=1 and selfcare=4 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.139;
if (mobility=1 and selfcare=4 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.601;
if (mobility=1 and selfcare=4 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.545;
if (mobility=1 and selfcare=4 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.530;
if (mobility=1 and selfcare=4 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.382;
if (mobility=1 and selfcare=4 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.228;
if (mobility=1 and selfcare=4 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.502;
if (mobility=1 and selfcare=4 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.446;
if (mobility=1 and selfcare=4 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.431;
if (mobility=1 and selfcare=4 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.283;
if (mobility=1 and selfcare=4 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.130;
if (mobility=1 and selfcare=4 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.478;
if (mobility=1 and selfcare=4 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.422;
if (mobility=1 and selfcare=4 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.407;
if (mobility=1 and selfcare=4 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.259;
if (mobility=1 and selfcare=4 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.105;
if (mobility=1 and selfcare=4 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.318;
if (mobility=1 and selfcare=4 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.262;
if (mobility=1 and selfcare=4 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.247;
if (mobility=1 and selfcare=4 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.126;
if (mobility=1 and selfcare=4 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.000;
if (mobility=1 and selfcare=4 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.078;
if (mobility=1 and selfcare=4 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.022;
if (mobility=1 and selfcare=4 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.007;
if (mobility=1 and selfcare=4 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.074;
if (mobility=1 and selfcare=4 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.158;
if (mobility=1 and selfcare=4 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.425;
if (mobility=1 and selfcare=4 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.369;
if (mobility=1 and selfcare=4 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.354;
if (mobility=1 and selfcare=4 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.273;
if (mobility=1 and selfcare=4 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.189;
if (mobility=1 and selfcare=4 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.327;
if (mobility=1 and selfcare=4 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.270;
if (mobility=1 and selfcare=4 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.256;
if (mobility=1 and selfcare=4 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.175;
if (mobility=1 and selfcare=4 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.091;
if (mobility=1 and selfcare=4 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.302;
if (mobility=1 and selfcare=4 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.246;
if (mobility=1 and selfcare=4 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.231;
```

```
if (mobility=1 and selfcare=4 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.150;
if (mobility=1 and selfcare=4 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.066;
if (mobility=1 and selfcare=4 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.197;
if (mobility=1 and selfcare=4 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.141;
if (mobility=1 and selfcare=4 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.126;
if (mobility=1 and selfcare=4 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.045;
if (mobility=1 and selfcare=4 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.039;
if (mobility=1 and selfcare=4 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.039;
if (mobility=1 and selfcare=4 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.017;
if (mobility=1 and selfcare=4 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.032;
if (mobility=1 and selfcare=4 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.113;
if (mobility=1 and selfcare=4 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.197;
if (mobility=1 and selfcare=5 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.436;
if (mobility=1 and selfcare=5 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.380;
if (mobility=1 and selfcare=5 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.365;
if (mobility=1 and selfcare=5 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.284;
if (mobility=1 and selfcare=5 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.200;
if (mobility=1 and selfcare=5 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.338;
if (mobility=1 and selfcare=5 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.281;
if (mobility=1 and selfcare=5 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.267;
if (mobility=1 and selfcare=5 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.186;
if (mobility=1 and selfcare=5 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.102;
if (mobility=1 and selfcare=5 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.313;
if (mobility=1 and selfcare=5 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.257;
if (mobility=1 and selfcare=5 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.242;
if (mobility=1 and selfcare=5 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.161;
if (mobility=1 and selfcare=5 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.077;
if (mobility=1 and selfcare=5 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.208;
if (mobility=1 and selfcare=5 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.152;
if (mobility=1 and selfcare=5 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.137;
if (mobility=1 and selfcare=5 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.056;
if (mobility=1 and selfcare=5 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.028;
if (mobility=1 and selfcare=5 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.050;
if (mobility=1 and selfcare=5 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.006;
if (mobility=1 and selfcare=5 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.021;
if (mobility=1 and selfcare=5 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.102;
if (mobility=1 and selfcare=5 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.186;
if (mobility=1 and selfcare=5 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.407;
if (mobility=1 and selfcare=5 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.351;
if (mobility=1 and selfcare=5 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.336;
if (mobility=1 and selfcare=5 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.255;
if (mobility=1 and selfcare=5 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.171;
if (mobility=1 and selfcare=5 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.309;
if (mobility=1 and selfcare=5 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.252;
if (mobility=1 and selfcare=5 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.238;
if (mobility=1 and selfcare=5 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.157;
```
```
if (mobility=1 and selfcare=5 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.073;
if (mobility=1 and selfcare=5 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.284;
if (mobility=1 and selfcare=5 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.228;
if (mobility=1 and selfcare=5 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.213;
if (mobility=1 and selfcare=5 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.132;
if (mobility=1 and selfcare=5 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.048;
if (mobility=1 and selfcare=5 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.179;
if (mobility=1 and selfcare=5 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.123;
if (mobility=1 and selfcare=5 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.108;
if (mobility=1 and selfcare=5 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.027;
if (mobility=1 and selfcare=5 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.057;
if (mobility=1 and selfcare=5 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.021;
if (mobility=1 and selfcare=5 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.035;
if (mobility=1 and selfcare=5 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.050;
if (mobility=1 and selfcare=5 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.131;
if (mobility=1 and selfcare=5 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.215;
if (mobility=1 and selfcare=5 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.400;
if (mobility=1 and selfcare=5 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.344;
if (mobility=1 and selfcare=5 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.329;
if (mobility=1 and selfcare=5 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.248;
if (mobility=1 and selfcare=5 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.164;
if (mobility=1 and selfcare=5 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.302;
if (mobility=1 and selfcare=5 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.245;
if (mobility=1 and selfcare=5 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.231;
if (mobility=1 and selfcare=5 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.150;
if (mobility=1 and selfcare=5 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.066;
if (mobility=1 and selfcare=5 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.277;
if (mobility=1 and selfcare=5 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.221;
if (mobility=1 and selfcare=5 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.206;
if (mobility=1 and selfcare=5 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.125;
if (mobility=1 and selfcare=5 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.041;
if (mobility=1 and selfcare=5 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.172;
if (mobility=1 and selfcare=5 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.116;
if (mobility=1 and selfcare=5 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.101;
if (mobility=1 and selfcare=5 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.020;
if (mobility=1 and selfcare=5 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.064;
if (mobility=1 and selfcare=5 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.014;
if (mobility=1 and selfcare=5 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.042;
if (mobility=1 and selfcare=5 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.057;
if (mobility=1 and selfcare=5 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.138;
if (mobility=1 and selfcare=5 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.222;
if (mobility=1 and selfcare=5 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.381;
if (mobility=1 and selfcare=5 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.325;
if (mobility=1 and selfcare=5 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.310;
if (mobility=1 and selfcare=5 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.229;
if (mobility=1 and selfcare=5 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.145;
```

```
if (mobility=1 and selfcare=5 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.282;
if (mobility=1 and selfcare=5 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.226;
if (mobility=1 and selfcare=5 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.211;
if (mobility=1 and selfcare=5 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.130;
if (mobility=1 and selfcare=5 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.046;
if (mobility=1 and selfcare=5 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.258;
if (mobility=1 and selfcare=5 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.202;
if (mobility=1 and selfcare=5 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.187;
if (mobility=1 and selfcare=5 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.106;
if (mobility=1 and selfcare=5 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.022;
if (mobility=1 and selfcare=5 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.153;
if (mobility=1 and selfcare=5 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.097;
if (mobility=1 and selfcare=5 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.082;
if (mobility=1 and selfcare=5 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.001;
if (mobility=1 and selfcare=5 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.083;
if (mobility=1 and selfcare=5 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.005;
if (mobility=1 and selfcare=5 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.061;
if (mobility=1 and selfcare=5 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.076;
if (mobility=1 and selfcare=5 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.157;
if (mobility=1 and selfcare=5 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.241;
if (mobility=1 and selfcare=5 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.342;
if (mobility=1 and selfcare=5 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.286;
if (mobility=1 and selfcare=5 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.271;
if (mobility=1 and selfcare=5 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.190;
if (mobility=1 and selfcare=5 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.106;
if (mobility=1 and selfcare=5 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.244;
if (mobility=1 and selfcare=5 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.187;
if (mobility=1 and selfcare=5 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.173;
if (mobility=1 and selfcare=5 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.092;
if (mobility=1 and selfcare=5 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.008;
if (mobility=1 and selfcare=5 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.219;
if (mobility=1 and selfcare=5 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.163;
if (mobility=1 and selfcare=5 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.148;
if (mobility=1 and selfcare=5 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.067;
if (mobility=1 and selfcare=5 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.017;
if (mobility=1 and selfcare=5 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.114;
if (mobility=1 and selfcare=5 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.058;
if (mobility=1 and selfcare=5 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.043;
if (mobility=1 and selfcare=5 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.038;
if (mobility=1 and selfcare=5 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.122;
if (mobility=1 and selfcare=5 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.044;
if (mobility=1 and selfcare=5 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.100;
if (mobility=1 and selfcare=5 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.115;
if (mobility=1 and selfcare=5 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.196;
if (mobility=1 and selfcare=5 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.280;
if (mobility=2 and selfcare=1 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.877;
```

```
if (mobility=2 and selfcare=1 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.809;
if (mobility=2 and selfcare=1 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.791;
if (mobility=2 and selfcare=1 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.578;
if (mobility=2 and selfcare=1 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.357;
if (mobility=2 and selfcare=1 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.767;
if (mobility=2 and selfcare=1 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.708;
if (mobility=2 and selfcare=1 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.693;
if (mobility=2 and selfcare=1 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.480;
if (mobility=2 and selfcare=1 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.259;
if (mobility=2 and selfcare=1 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.739;
if (mobility=2 and selfcare=1 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.683;
if (mobility=2 and selfcare=1 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.668;
if (mobility=2 and selfcare=1 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.455;
if (mobility=2 and selfcare=1 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.234;
if (mobility=2 and selfcare=1 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.527;
if (mobility=2 and selfcare=1 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.470;
if (mobility=2 and selfcare=1 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.456;
if (mobility=2 and selfcare=1 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.296;
if (mobility=2 and selfcare=1 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.129;
if (mobility=2 and selfcare=1 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.207;
if (mobility=2 and selfcare=1 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.151;
if (mobility=2 and selfcare=1 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.136;
if (mobility=2 and selfcare=1 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.055;
if (mobility=2 and selfcare=1 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.029;
if (mobility=2 and selfcare=1 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.836;
if (mobility=2 and selfcare=1 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.778;
if (mobility=2 and selfcare=1 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.762;
if (mobility=2 and selfcare=1 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.549;
if (mobility=2 and selfcare=1 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.328;
if (mobility=2 and selfcare=1 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.735;
if (mobility=2 and selfcare=1 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.679;
if (mobility=2 and selfcare=1 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.664;
if (mobility=2 and selfcare=1 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.451;
if (mobility=2 and selfcare=1 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.230;
if (mobility=2 and selfcare=1 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.710;
if (mobility=2 and selfcare=1 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.654;
if (mobility=2 and selfcare=1 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.639;
if (mobility=2 and selfcare=1 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.426;
if (mobility=2 and selfcare=1 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.205;
if (mobility=2 and selfcare=1 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.498;
if (mobility=2 and selfcare=1 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.442;
if (mobility=2 and selfcare=1 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.427;
if (mobility=2 and selfcare=1 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.267;
if (mobility=2 and selfcare=1 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.100;
if (mobility=2 and selfcare=1 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.178;
if (mobility=2 and selfcare=1 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.122;
```

```
if (mobility=2 and selfcare=1 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.107;
if (mobility=2 and selfcare=1 and activity=2 and pain=5 and anxiety=4) then EQindex = 0.026;
if (mobility=2 and selfcare=1 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.058;
if (mobility=2 and selfcare=1 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.826;
if (mobility=2 and selfcare=1 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.770;
if (mobility=2 and selfcare=1 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.755;
if (mobility=2 and selfcare=1 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.542;
if (mobility=2 and selfcare=1 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.321;
if (mobility=2 and selfcare=1 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.728;
if (mobility=2 and selfcare=1 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.671;
if (mobility=2 and selfcare=1 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.657;
if (mobility=2 and selfcare=1 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.444;
if (mobility=2 and selfcare=1 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.223;
if (mobility=2 and selfcare=1 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.703;
if (mobility=2 and selfcare=1 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.647;
if (mobility=2 and selfcare=1 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.632;
if (mobility=2 and selfcare=1 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.419;
if (mobility=2 and selfcare=1 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.198;
if (mobility=2 and selfcare=1 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.491;
if (mobility=2 and selfcare=1 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.434;
if (mobility=2 and selfcare=1 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.420;
if (mobility=2 and selfcare=1 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.260;
if (mobility=2 and selfcare=1 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.093;
if (mobility=2 and selfcare=1 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.171;
if (mobility=2 and selfcare=1 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.115;
if (mobility=2 and selfcare=1 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.100;
if (mobility=2 and selfcare=1 and activity=3 and pain=5 and anxiety=4) then EQindex = 0.019;
if (mobility=2 and selfcare=1 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.065;
if (mobility=2 and selfcare=1 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.719;
if (mobility=2 and selfcare=1 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.663;
if (mobility=2 and selfcare=1 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.648;
if (mobility=2 and selfcare=1 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.478;
if (mobility=2 and selfcare=1 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.302;
if (mobility=2 and selfcare=1 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.620;
if (mobility=2 and selfcare=1 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.564;
if (mobility=2 and selfcare=1 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.549;
if (mobility=2 and selfcare=1 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.380;
if (mobility=2 and selfcare=1 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.204;
if (mobility=2 and selfcare=1 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.596;
if (mobility=2 and selfcare=1 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.540;
if (mobility=2 and selfcare=1 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.525;
if (mobility=2 and selfcare=1 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.355;
if (mobility=2 and selfcare=1 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.179;
if (mobility=2 and selfcare=1 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.419;
if (mobility=2 and selfcare=1 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.362;
if (mobility=2 and selfcare=1 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.348;
```

```
if (mobility=2 and selfcare=1 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.213;
if (mobility=2 and selfcare=1 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.074;
if (mobility=2 and selfcare=1 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.152;
if (mobility=2 and selfcare=1 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.096;
if (mobility=2 and selfcare=1 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.081;
if (mobility=2 and selfcare=1 and activity=4 and pain=5 and anxiety=4) then EQindex = 0.000;
if (mobility=2 and selfcare=1 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.084;
if (mobility=2 and selfcare=1 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.499;
if (mobility=2 and selfcare=1 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.443;
if (mobility=2 and selfcare=1 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.428;
if (mobility=2 and selfcare=1 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.347;
if (mobility=2 and selfcare=1 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.263;
if (mobility=2 and selfcare=1 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.401;
if (mobility=2 and selfcare=1 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.344;
if (mobility=2 and selfcare=1 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.330;
if (mobility=2 and selfcare=1 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.249;
if (mobility=2 and selfcare=1 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.165;
if (mobility=2 and selfcare=1 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.376;
if (mobility=2 and selfcare=1 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.320;
if (mobility=2 and selfcare=1 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.305;
if (mobility=2 and selfcare=1 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.224;
if (mobility=2 and selfcare=1 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.140;
if (mobility=2 and selfcare=1 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.271;
if (mobility=2 and selfcare=1 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.215;
if (mobility=2 and selfcare=1 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.200;
if (mobility=2 and selfcare=1 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.119;
if (mobility=2 and selfcare=1 and activity=5 and pain=4 and anxiety=5) then EQindex = 0.035;
if (mobility=2 and selfcare=1 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.113;
if (mobility=2 and selfcare=1 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.057;
if (mobility=2 and selfcare=1 and activity=5 and pain=5 and anxiety=3) then EQindex = 0.042;
if (mobility=2 and selfcare=1 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.039;
if (mobility=2 and selfcare=1 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.123;
if (mobility=2 and selfcare=2 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.778;
if (mobility=2 and selfcare=2 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.720;
if (mobility=2 and selfcare=2 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.705;
if (mobility=2 and selfcare=2 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.492;
if (mobility=2 and selfcare=2 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.271;
if (mobility=2 and selfcare=2 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.678;
if (mobility=2 and selfcare=2 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.621;
if (mobility=2 and selfcare=2 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.606;
if (mobility=2 and selfcare=2 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.393;
if (mobility=2 and selfcare=2 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.172;
if (mobility=2 and selfcare=2 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.653;
if (mobility=2 and selfcare=2 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.596;
if (mobility=2 and selfcare=2 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.582;
if (mobility=2 and selfcare=2 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.369;
```

```
if (mobility=2 and selfcare=2 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.148;
if (mobility=2 and selfcare=2 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.440;
if (mobility=2 and selfcare=2 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.384;
if (mobility=2 and selfcare=2 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.369;
if (mobility=2 and selfcare=2 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.209;
if (mobility=2 and selfcare=2 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.043;
if (mobility=2 and selfcare=2 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.121;
if (mobility=2 and selfcare=2 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.064;
if (mobility=2 and selfcare=2 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.050;
if (mobility=2 and selfcare=2 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.031;
if (mobility=2 and selfcare=2 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.115;
if (mobility=2 and selfcare=2 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.747;
if (mobility=2 and selfcare=2 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.691;
if (mobility=2 and selfcare=2 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.676;
if (mobility=2 and selfcare=2 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.463;
if (mobility=2 and selfcare=2 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.242;
if (mobility=2 and selfcare=2 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.648;
if (mobility=2 and selfcare=2 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.592;
if (mobility=2 and selfcare=2 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.577;
if (mobility=2 and selfcare=2 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.364;
if (mobility=2 and selfcare=2 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.143;
if (mobility=2 and selfcare=2 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.624;
if (mobility=2 and selfcare=2 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.567;
if (mobility=2 and selfcare=2 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.553;
if (mobility=2 and selfcare=2 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.340;
if (mobility=2 and selfcare=2 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.119;
if (mobility=2 and selfcare=2 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.411;
if (mobility=2 and selfcare=2 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.355;
if (mobility=2 and selfcare=2 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.340;
if (mobility=2 and selfcare=2 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.180;
if (mobility=2 and selfcare=2 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.014;
if (mobility=2 and selfcare=2 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.092;
if (mobility=2 and selfcare=2 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.035;
if (mobility=2 and selfcare=2 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.021;
if (mobility=2 and selfcare=2 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.060;
if (mobility=2 and selfcare=2 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.144;
if (mobility=2 and selfcare=2 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.740;
if (mobility=2 and selfcare=2 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.683;
if (mobility=2 and selfcare=2 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.669;
if (mobility=2 and selfcare=2 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.456;
if (mobility=2 and selfcare=2 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.235;
if (mobility=2 and selfcare=2 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.641;
if (mobility=2 and selfcare=2 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.585;
if (mobility=2 and selfcare=2 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.570;
if (mobility=2 and selfcare=2 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.357;
if (mobility=2 and selfcare=2 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.136;
```

```
if (mobility=2 and selfcare=2 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.617;
if (mobility=2 and selfcare=2 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.560;
if (mobility=2 and selfcare=2 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.546;
if (mobility=2 and selfcare=2 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.333;
if (mobility=2 and selfcare=2 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.112;
if (mobility=2 and selfcare=2 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.404;
if (mobility=2 and selfcare=2 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.348;
if (mobility=2 and selfcare=2 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.333;
if (mobility=2 and selfcare=2 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.173;
if (mobility=2 and selfcare=2 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.007;
if (mobility=2 and selfcare=2 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.085;
if (mobility=2 and selfcare=2 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.028;
if (mobility=2 and selfcare=2 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.014;
if (mobility=2 and selfcare=2 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.067;
if (mobility=2 and selfcare=2 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.151;
if (mobility=2 and selfcare=2 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.632;
if (mobility=2 and selfcare=2 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.576;
if (mobility=2 and selfcare=2 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.561;
if (mobility=2 and selfcare=2 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.392;
if (mobility=2 and selfcare=2 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.216;
if (mobility=2 and selfcare=2 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.534;
if (mobility=2 and selfcare=2 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.477;
if (mobility=2 and selfcare=2 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.463;
if (mobility=2 and selfcare=2 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.293;
if (mobility=2 and selfcare=2 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.117;
if (mobility=2 and selfcare=2 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.509;
if (mobility=2 and selfcare=2 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.453;
if (mobility=2 and selfcare=2 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.438;
if (mobility=2 and selfcare=2 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.269;
if (mobility=2 and selfcare=2 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.093;
if (mobility=2 and selfcare=2 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.332;
if (mobility=2 and selfcare=2 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.276;
if (mobility=2 and selfcare=2 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.261;
if (mobility=2 and selfcare=2 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.127;
if (mobility=2 and selfcare=2 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.013;
if (mobility=2 and selfcare=2 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.066;
if (mobility=2 and selfcare=2 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.009;
if (mobility=2 and selfcare=2 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.005;
if (mobility=2 and selfcare=2 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.086;
if (mobility=2 and selfcare=2 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.170;
if (mobility=2 and selfcare=2 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.413;
if (mobility=2 and selfcare=2 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.356;
if (mobility=2 and selfcare=2 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.342;
if (mobility=2 and selfcare=2 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.261;
if (mobility=2 and selfcare=2 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.177;
if (mobility=2 and selfcare=2 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.314;
```

```
if (mobility=2 and selfcare=2 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.258;
if (mobility=2 and selfcare=2 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.243;
if (mobility=2 and selfcare=2 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.162;
if (mobility=2 and selfcare=2 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.078;
if (mobility=2 and selfcare=2 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.290;
if (mobility=2 and selfcare=2 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.233;
if (mobility=2 and selfcare=2 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.219;
if (mobility=2 and selfcare=2 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.138;
if (mobility=2 and selfcare=2 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.054;
if (mobility=2 and selfcare=2 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.185;
if (mobility=2 and selfcare=2 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.128;
if (mobility=2 and selfcare=2 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.114;
if (mobility=2 and selfcare=2 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.033;
if (mobility=2 and selfcare=2 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.051;
if (mobility=2 and selfcare=2 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.027;
if (mobility=2 and selfcare=2 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.030;
if (mobility=2 and selfcare=2 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.044;
if (mobility=2 and selfcare=2 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.125;
if (mobility=2 and selfcare=2 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.209;
if (mobility=2 and selfcare=3 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.758;
if (mobility=2 and selfcare=3 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.702;
if (mobility=2 and selfcare=3 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.687;
if (mobility=2 and selfcare=3 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.474;
if (mobility=2 and selfcare=3 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.253;
if (mobility=2 and selfcare=3 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.660;
if (mobility=2 and selfcare=3 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.603;
if (mobility=2 and selfcare=3 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.589;
if (mobility=2 and selfcare=3 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.376;
if (mobility=2 and selfcare=3 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.155;
if (mobility=2 and selfcare=3 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.635;
if (mobility=2 and selfcare=3 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.579;
if (mobility=2 and selfcare=3 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.564;
if (mobility=2 and selfcare=3 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.351;
if (mobility=2 and selfcare=3 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.130;
if (mobility=2 and selfcare=3 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.423;
if (mobility=2 and selfcare=3 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.366;
if (mobility=2 and selfcare=3 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.352;
if (mobility=2 and selfcare=3 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.192;
if (mobility=2 and selfcare=3 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.025;
if (mobility=2 and selfcare=3 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.103;
if (mobility=2 and selfcare=3 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.047;
if (mobility=2 and selfcare=3 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.032;
if (mobility=2 and selfcare=3 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.049;
if (mobility=2 and selfcare=3 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.133;
if (mobility=2 and selfcare=3 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.729;
if (mobility=2 and selfcare=3 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.673;
```

```
if (mobility=2 and selfcare=3 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.658;
if (mobility=2 and selfcare=3 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.445;
if (mobility=2 and selfcare=3 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.224;
if (mobility=2 and selfcare=3 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.631;
if (mobility=2 and selfcare=3 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.575;
if (mobility=2 and selfcare=3 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.560;
if (mobility=2 and selfcare=3 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.347;
if (mobility=2 and selfcare=3 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.126;
if (mobility=2 and selfcare=3 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.606;
if (mobility=2 and selfcare=3 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.550;
if (mobility=2 and selfcare=3 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.535;
if (mobility=2 and selfcare=3 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.322;
if (mobility=2 and selfcare=3 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.101;
if (mobility=2 and selfcare=3 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.394;
if (mobility=2 and selfcare=3 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.338;
if (mobility=2 and selfcare=3 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.323;
if (mobility=2 and selfcare=3 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.163;
if (mobility=2 and selfcare=3 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.004;
if (mobility=2 and selfcare=3 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.074;
if (mobility=2 and selfcare=3 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.018;
if (mobility=2 and selfcare=3 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.003;
if (mobility=2 and selfcare=3 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.078;
if (mobility=2 and selfcare=3 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.162;
if (mobility=2 and selfcare=3 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.722;
if (mobility=2 and selfcare=3 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.666;
if (mobility=2 and selfcare=3 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.651;
if (mobility=2 and selfcare=3 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.438;
if (mobility=2 and selfcare=3 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.217;
if (mobility=2 and selfcare=3 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.624;
if (mobility=2 and selfcare=3 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.567;
if (mobility=2 and selfcare=3 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.553;
if (mobility=2 and selfcare=3 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.340;
if (mobility=2 and selfcare=3 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.119;
if (mobility=2 and selfcare=3 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.599;
if (mobility=2 and selfcare=3 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.543;
if (mobility=2 and selfcare=3 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.528;
if (mobility=2 and selfcare=3 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.315;
if (mobility=2 and selfcare=3 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.094;
if (mobility=2 and selfcare=3 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.387;
if (mobility=2 and selfcare=3 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.330;
if (mobility=2 and selfcare=3 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.316;
if (mobility=2 and selfcare=3 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.156;
if (mobility=2 and selfcare=3 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.011;
if (mobility=2 and selfcare=3 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.067;
if (mobility=2 and selfcare=3 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.011;
if (mobility=2 and selfcare=3 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.004;
```

```
if (mobility=2 and selfcare=3 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.085;
if (mobility=2 and selfcare=3 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.169;
if (mobility=2 and selfcare=3 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.615;
if (mobility=2 and selfcare=3 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.559;
if (mobility=2 and selfcare=3 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.544;
if (mobility=2 and selfcare=3 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.374;
if (mobility=2 and selfcare=3 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.198;
if (mobility=2 and selfcare=3 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.516;
if (mobility=2 and selfcare=3 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.460;
if (mobility=2 and selfcare=3 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.445;
if (mobility=2 and selfcare=3 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.276;
if (mobility=2 and selfcare=3 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.100;
if (mobility=2 and selfcare=3 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.492;
if (mobility=2 and selfcare=3 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.436;
if (mobility=2 and selfcare=3 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.421;
if (mobility=2 and selfcare=3 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.251;
if (mobility=2 and selfcare=3 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.075;
if (mobility=2 and selfcare=3 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.315;
if (mobility=2 and selfcare=3 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.258;
if (mobility=2 and selfcare=3 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.244;
if (mobility=2 and selfcare=3 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.109;
if (mobility=2 and selfcare=3 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.030;
if (mobility=2 and selfcare=3 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.048;
if (mobility=2 and selfcare=3 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.008;
if (mobility=2 and selfcare=3 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.023;
if (mobility=2 and selfcare=3 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.104;
if (mobility=2 and selfcare=3 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.188;
if (mobility=2 and selfcare=3 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.395;
if (mobility=2 and selfcare=3 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.339;
if (mobility=2 and selfcare=3 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.324;
if (mobility=2 and selfcare=3 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.243;
if (mobility=2 and selfcare=3 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.159;
if (mobility=2 and selfcare=3 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.297;
if (mobility=2 and selfcare=3 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.240;
if (mobility=2 and selfcare=3 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.226;
if (mobility=2 and selfcare=3 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.145;
if (mobility=2 and selfcare=3 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.061;
if (mobility=2 and selfcare=3 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.272;
if (mobility=2 and selfcare=3 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.216;
if (mobility=2 and selfcare=3 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.201;
if (mobility=2 and selfcare=3 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.120;
if (mobility=2 and selfcare=3 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.036;
if (mobility=2 and selfcare=3 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.167;
if (mobility=2 and selfcare=3 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.111;
if (mobility=2 and selfcare=3 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.096;
if (mobility=2 and selfcare=3 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.015;
```

```
if (mobility=2 and selfcare=3 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.069;
if (mobility=2 and selfcare=3 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.009;
if (mobility=2 and selfcare=3 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.047;
if (mobility=2 and selfcare=3 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.062;
if (mobility=2 and selfcare=3 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.143;
if (mobility=2 and selfcare=3 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.227;
if (mobility=2 and selfcare=4 and activity=1 and pain=1 and anxiety=1) then EOindex = 0.666;
if (mobility=2 and selfcare=4 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.610;
if (mobility=2 and selfcare=4 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.595;
if (mobility=2 and selfcare=4 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.414;
if (mobility=2 and selfcare=4 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.227;
if (mobility=2 and selfcare=4 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.568;
if (mobility=2 and selfcare=4 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.511;
if (mobility=2 and selfcare=4 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.497;
if (mobility=2 and selfcare=4 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.316;
if (mobility=2 and selfcare=4 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.128;
if (mobility=2 and selfcare=4 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.543;
if (mobility=2 and selfcare=4 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.487;
if (mobility=2 and selfcare=4 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.472;
if (mobility=2 and selfcare=4 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.291;
if (mobility=2 and selfcare=4 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.104;
if (mobility=2 and selfcare=4 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.357;
if (mobility=2 and selfcare=4 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.300;
if (mobility=2 and selfcare=4 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.286;
if (mobility=2 and selfcare=4 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.145;
if (mobility=2 and selfcare=4 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.002;
if (mobility=2 and selfcare=4 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.077;
if (mobility=2 and selfcare=4 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.020;
if (mobility=2 and selfcare=4 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.006;
if (mobility=2 and selfcare=4 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.076;
if (mobility=2 and selfcare=4 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.160;
if (mobility=2 and selfcare=4 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.637;
if (mobility=2 and selfcare=4 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.581;
if (mobility=2 and selfcare=4 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.566;
if (mobility=2 and selfcare=4 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.385;
if (mobility=2 and selfcare=4 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.198;
if (mobility=2 and selfcare=4 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.539;
if (mobility=2 and selfcare=4 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.482;
if (mobility=2 and selfcare=4 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.468;
if (mobility=2 and selfcare=4 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.287;
if (mobility=2 and selfcare=4 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.099;
if (mobility=2 and selfcare=4 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.514;
if (mobility=2 and selfcare=4 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.458;
if (mobility=2 and selfcare=4 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.443;
if (mobility=2 and selfcare=4 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.262;
if (mobility=2 and selfcare=4 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.075;
```

```
if (mobility=2 and selfcare=4 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.328;
if (mobility=2 and selfcare=4 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.272;
if (mobility=2 and selfcare=4 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.257;
if (mobility=2 and selfcare=4 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.116;
if (mobility=2 and selfcare=4 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.030;
if (mobility=2 and selfcare=4 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.048;
if (mobility=2 and selfcare=4 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.009;
if (mobility=2 and selfcare=4 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.023;
if (mobility=2 and selfcare=4 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.104;
if (mobility=2 and selfcare=4 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.188;
if (mobility=2 and selfcare=4 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.630;
if (mobility=2 and selfcare=4 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.574;
if (mobility=2 and selfcare=4 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.559;
if (mobility=2 and selfcare=4 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.378;
if (mobility=2 and selfcare=4 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.191;
if (mobility=2 and selfcare=4 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.532;
if (mobility=2 and selfcare=4 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.475;
if (mobility=2 and selfcare=4 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.461;
if (mobility=2 and selfcare=4 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.280;
if (mobility=2 and selfcare=4 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.092;
if (mobility=2 and selfcare=4 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.507;
if (mobility=2 and selfcare=4 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.451;
if (mobility=2 and selfcare=4 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.436;
if (mobility=2 and selfcare=4 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.255;
if (mobility=2 and selfcare=4 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.068;
if (mobility=2 and selfcare=4 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.321;
if (mobility=2 and selfcare=4 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.264;
if (mobility=2 and selfcare=4 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.250;
if (mobility=2 and selfcare=4 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.109;
if (mobility=2 and selfcare=4 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.038;
if (mobility=2 and selfcare=4 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.041;
if (mobility=2 and selfcare=4 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.016;
if (mobility=2 and selfcare=4 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.031;
if (mobility=2 and selfcare=4 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.112;
if (mobility=2 and selfcare=4 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.196;
if (mobility=2 and selfcare=4 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.544;
if (mobility=2 and selfcare=4 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.488;
if (mobility=2 and selfcare=4 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.473;
if (mobility=2 and selfcare=4 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.325;
if (mobility=2 and selfcare=4 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.172;
if (mobility=2 and selfcare=4 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.446;
if (mobility=2 and selfcare=4 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.389;
if (mobility=2 and selfcare=4 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.375;
if (mobility=2 and selfcare=4 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.227;
if (mobility=2 and selfcare=4 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.073;
if (mobility=2 and selfcare=4 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.421;
```

```
if (mobility=2 and selfcare=4 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.365;
if (mobility=2 and selfcare=4 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.350;
if (mobility=2 and selfcare=4 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.202;
if (mobility=2 and selfcare=4 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.049;
if (mobility=2 and selfcare=4 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.262;
if (mobility=2 and selfcare=4 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.205;
if (mobility=2 and selfcare=4 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.191;
if (mobility=2 and selfcare=4 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.069;
if (mobility=2 and selfcare=4 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.057;
if (mobility=2 and selfcare=4 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.022;
if (mobility=2 and selfcare=4 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.035;
if (mobility=2 and selfcare=4 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.050;
if (mobility=2 and selfcare=4 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.131;
if (mobility=2 and selfcare=4 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.215;
if (mobility=2 and selfcare=4 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.369;
if (mobility=2 and selfcare=4 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.312;
if (mobility=2 and selfcare=4 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.298;
if (mobility=2 and selfcare=4 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.217;
if (mobility=2 and selfcare=4 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.133;
if (mobility=2 and selfcare=4 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.270;
if (mobility=2 and selfcare=4 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.214;
if (mobility=2 and selfcare=4 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.199;
if (mobility=2 and selfcare=4 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.118;
if (mobility=2 and selfcare=4 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.034;
if (mobility=2 and selfcare=4 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.246;
if (mobility=2 and selfcare=4 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.189;
if (mobility=2 and selfcare=4 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.175;
if (mobility=2 and selfcare=4 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.094;
if (mobility=2 and selfcare=4 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.010;
if (mobility=2 and selfcare=4 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.140;
if (mobility=2 and selfcare=4 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.084;
if (mobility=2 and selfcare=4 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.069;
if (mobility=2 and selfcare=4 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.012;
if (mobility=2 and selfcare=4 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.096;
if (mobility=2 and selfcare=4 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.018;
if (mobility=2 and selfcare=4 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.074;
if (mobility=2 and selfcare=4 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.089;
if (mobility=2 and selfcare=4 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.170;
if (mobility=2 and selfcare=4 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.254;
if (mobility=2 and selfcare=5 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.379;
if (mobility=2 and selfcare=5 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.323;
if (mobility=2 and selfcare=5 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.308;
if (mobility=2 and selfcare=5 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.227;
if (mobility=2 and selfcare=5 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.143;
if (mobility=2 and selfcare=5 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.281;
if (mobility=2 and selfcare=5 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.224;
```

```
if (mobility=2 and selfcare=5 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.210;
if (mobility=2 and selfcare=5 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.129;
if (mobility=2 and selfcare=5 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.045;
if (mobility=2 and selfcare=5 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.256;
if (mobility=2 and selfcare=5 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.200;
if (mobility=2 and selfcare=5 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.185;
if (mobility=2 and selfcare=5 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.104;
if (mobility=2 and selfcare=5 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.020;
if (mobility=2 and selfcare=5 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.151;
if (mobility=2 and selfcare=5 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.095;
if (mobility=2 and selfcare=5 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.080;
if (mobility=2 and selfcare=5 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.001;
if (mobility=2 and selfcare=5 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.085;
if (mobility=2 and selfcare=5 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.007;
if (mobility=2 and selfcare=5 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.063;
if (mobility=2 and selfcare=5 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.078;
if (mobility=2 and selfcare=5 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.159;
if (mobility=2 and selfcare=5 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.243;
if (mobility=2 and selfcare=5 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.350;
if (mobility=2 and selfcare=5 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.294;
if (mobility=2 and selfcare=5 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.279;
if (mobility=2 and selfcare=5 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.198;
if (mobility=2 and selfcare=5 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.114;
if (mobility=2 and selfcare=5 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.252;
if (mobility=2 and selfcare=5 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.196;
if (mobility=2 and selfcare=5 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.181;
if (mobility=2 and selfcare=5 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.100;
if (mobility=2 and selfcare=5 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.016;
if (mobility=2 and selfcare=5 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.227;
if (mobility=2 and selfcare=5 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.171;
if (mobility=2 and selfcare=5 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.156;
if (mobility=2 and selfcare=5 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.075;
if (mobility=2 and selfcare=5 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.009;
if (mobility=2 and selfcare=5 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.122;
if (mobility=2 and selfcare=5 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.066;
if (mobility=2 and selfcare=5 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.051;
if (mobility=2 and selfcare=5 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.030;
if (mobility=2 and selfcare=5 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.114;
if (mobility=2 and selfcare=5 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.036;
if (mobility=2 and selfcare=5 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.092;
if (mobility=2 and selfcare=5 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.107;
if (mobility=2 and selfcare=5 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.188;
if (mobility=2 and selfcare=5 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.272;
if (mobility=2 and selfcare=5 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.343;
if (mobility=2 and selfcare=5 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.287;
if (mobility=2 and selfcare=5 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.272;
```

```
if (mobility=2 and selfcare=5 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.191;
if (mobility=2 and selfcare=5 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.107;
if (mobility=2 and selfcare=5 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.245;
if (mobility=2 and selfcare=5 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.188;
if (mobility=2 and selfcare=5 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.174;
if (mobility=2 and selfcare=5 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.093;
if (mobility=2 and selfcare=5 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.009;
if (mobility=2 and selfcare=5 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.220;
if (mobility=2 and selfcare=5 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.164;
if (mobility=2 and selfcare=5 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.149;
if (mobility=2 and selfcare=5 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.068;
if (mobility=2 and selfcare=5 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.016;
if (mobility=2 and selfcare=5 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.115;
if (mobility=2 and selfcare=5 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.059;
if (mobility=2 and selfcare=5 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.044;
if (mobility=2 and selfcare=5 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.037;
if (mobility=2 and selfcare=5 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.121;
if (mobility=2 and selfcare=5 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.043;
if (mobility=2 and selfcare=5 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.099;
if (mobility=2 and selfcare=5 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.114;
if (mobility=2 and selfcare=5 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.195;
if (mobility=2 and selfcare=5 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.279;
if (mobility=2 and selfcare=5 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.324;
if (mobility=2 and selfcare=5 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.268;
if (mobility=2 and selfcare=5 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.253;
if (mobility=2 and selfcare=5 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.172;
if (mobility=2 and selfcare=5 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.088;
if (mobility=2 and selfcare=5 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.226;
if (mobility=2 and selfcare=5 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.169;
if (mobility=2 and selfcare=5 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.155;
if (mobility=2 and selfcare=5 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.074;
if (mobility=2 and selfcare=5 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.010;
if (mobility=2 and selfcare=5 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.201;
if (mobility=2 and selfcare=5 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.145;
if (mobility=2 and selfcare=5 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.130;
if (mobility=2 and selfcare=5 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.049;
if (mobility=2 and selfcare=5 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.035;
if (mobility=2 and selfcare=5 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.096;
if (mobility=2 and selfcare=5 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.040;
if (mobility=2 and selfcare=5 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.025;
if (mobility=2 and selfcare=5 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.056;
if (mobility=2 and selfcare=5 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.140;
if (mobility=2 and selfcare=5 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.062;
if (mobility=2 and selfcare=5 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.118;
if (mobility=2 and selfcare=5 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.133;
if (mobility=2 and selfcare=5 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.214;
```

```
if (mobility=2 and selfcare=5 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.298;
if (mobility=2 and selfcare=5 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.285;
if (mobility=2 and selfcare=5 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.229;
if (mobility=2 and selfcare=5 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.214;
if (mobility=2 and selfcare=5 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.133;
if (mobility=2 and selfcare=5 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.049;
if (mobility=2 and selfcare=5 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.187;
if (mobility=2 and selfcare=5 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.130;
if (mobility=2 and selfcare=5 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.116;
if (mobility=2 and selfcare=5 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.035;
if (mobility=2 and selfcare=5 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.049;
if (mobility=2 and selfcare=5 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.162;
if (mobility=2 and selfcare=5 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.106;
if (mobility=2 and selfcare=5 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.091;
if (mobility=2 and selfcare=5 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.010;
if (mobility=2 and selfcare=5 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.074;
if (mobility=2 and selfcare=5 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.057;
if (mobility=2 and selfcare=5 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.001;
if (mobility=2 and selfcare=5 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.014;
if (mobility=2 and selfcare=5 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.095;
if (mobility=2 and selfcare=5 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.179;
if (mobility=2 and selfcare=5 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.101;
if (mobility=2 and selfcare=5 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.157;
if (mobility=2 and selfcare=5 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.172;
if (mobility=2 and selfcare=5 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.253;
if (mobility=2 and selfcare=5 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.337;
if (mobility=3 and selfcare=1 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.850;
if (mobility=3 and selfcare=1 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.794;
if (mobility=3 and selfcare=1 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.779;
if (mobility=3 and selfcare=1 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.566;
if (mobility=3 and selfcare=1 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.345;
if (mobility=3 and selfcare=1 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.752;
if (mobility=3 and selfcare=1 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.695;
if (mobility=3 and selfcare=1 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.681;
if (mobility=3 and selfcare=1 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.468;
if (mobility=3 and selfcare=1 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.247;
if (mobility=3 and selfcare=1 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.727;
if (mobility=3 and selfcare=1 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.671;
if (mobility=3 and selfcare=1 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.656;
if (mobility=3 and selfcare=1 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.443;
if (mobility=3 and selfcare=1 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.222;
if (mobility=3 and selfcare=1 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.515;
if (mobility=3 and selfcare=1 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.458;
if (mobility=3 and selfcare=1 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.444;
if (mobility=3 and selfcare=1 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.283;
if (mobility=3 and selfcare=1 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.117;
```

```
if (mobility=3 and selfcare=1 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.195;
if (mobility=3 and selfcare=1 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.139;
if (mobility=3 and selfcare=1 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.124;
if (mobility=3 and selfcare=1 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.043;
if (mobility=3 and selfcare=1 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.041;
if (mobility=3 and selfcare=1 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.821;
if (mobility=3 and selfcare=1 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.765;
if (mobility=3 and selfcare=1 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.750;
if (mobility=3 and selfcare=1 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.537;
if (mobility=3 and selfcare=1 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.316;
if (mobility=3 and selfcare=1 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.723;
if (mobility=3 and selfcare=1 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.666;
if (mobility=3 and selfcare=1 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.652;
if (mobility=3 and selfcare=1 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.439;
if (mobility=3 and selfcare=1 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.218;
if (mobility=3 and selfcare=1 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.698;
if (mobility=3 and selfcare=1 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.642;
if (mobility=3 and selfcare=1 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.627;
if (mobility=3 and selfcare=1 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.414;
if (mobility=3 and selfcare=1 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.193;
if (mobility=3 and selfcare=1 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.486;
if (mobility=3 and selfcare=1 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.429;
if (mobility=3 and selfcare=1 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.415;
if (mobility=3 and selfcare=1 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.254;
if (mobility=3 and selfcare=1 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.088;
if (mobility=3 and selfcare=1 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.166;
if (mobility=3 and selfcare=1 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.110;
if (mobility=3 and selfcare=1 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.095;
if (mobility=3 and selfcare=1 and activity=2 and pain=5 and anxiety=4) then EQindex = 0.014;
if (mobility=3 and selfcare=1 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.070;
if (mobility=3 and selfcare=1 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.814;
if (mobility=3 and selfcare=1 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.758;
if (mobility=3 and selfcare=1 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.743;
if (mobility=3 and selfcare=1 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.530;
if (mobility=3 and selfcare=1 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.309;
if (mobility=3 and selfcare=1 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.716;
if (mobility=3 and selfcare=1 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.659;
if (mobility=3 and selfcare=1 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.645;
if (mobility=3 and selfcare=1 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.432;
if (mobility=3 and selfcare=1 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.211;
if (mobility=3 and selfcare=1 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.691;
if (mobility=3 and selfcare=1 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.635;
if (mobility=3 and selfcare=1 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.620;
if (mobility=3 and selfcare=1 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.407;
if (mobility=3 and selfcare=1 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.186;
if (mobility=3 and selfcare=1 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.479;
```

```
if (mobility=3 and selfcare=1 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.422;
if (mobility=3 and selfcare=1 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.408;
if (mobility=3 and selfcare=1 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.247;
if (mobility=3 and selfcare=1 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.081;
if (mobility=3 and selfcare=1 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.159;
if (mobility=3 and selfcare=1 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.103;
if (mobility=3 and selfcare=1 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.088;
if (mobility=3 and selfcare=1 and activity=3 and pain=5 and anxiety=4) then EQindex = 0.007;
if (mobility=3 and selfcare=1 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.077;
if (mobility=3 and selfcare=1 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.707;
if (mobility=3 and selfcare=1 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.650;
if (mobility=3 and selfcare=1 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.636;
if (mobility=3 and selfcare=1 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.466;
if (mobility=3 and selfcare=1 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.290;
if (mobility=3 and selfcare=1 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.608;
if (mobility=3 and selfcare=1 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.552;
if (mobility=3 and selfcare=1 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.537;
if (mobility=3 and selfcare=1 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.368;
if (mobility=3 and selfcare=1 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.191;
if (mobility=3 and selfcare=1 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.584;
if (mobility=3 and selfcare=1 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.527;
if (mobility=3 and selfcare=1 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.513;
if (mobility=3 and selfcare=1 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.343;
if (mobility=3 and selfcare=1 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.167;
if (mobility=3 and selfcare=1 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.406;
if (mobility=3 and selfcare=1 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.350;
if (mobility=3 and selfcare=1 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.335;
if (mobility=3 and selfcare=1 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.201;
if (mobility=3 and selfcare=1 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.062;
if (mobility=3 and selfcare=1 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.140;
if (mobility=3 and selfcare=1 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.084;
if (mobility=3 and selfcare=1 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.069;
if (mobility=3 and selfcare=1 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.012;
if (mobility=3 and selfcare=1 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.096;
if (mobility=3 and selfcare=1 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.487;
if (mobility=3 and selfcare=1 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.431;
if (mobility=3 and selfcare=1 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.416;
if (mobility=3 and selfcare=1 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.335;
if (mobility=3 and selfcare=1 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.251;
if (mobility=3 and selfcare=1 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.389;
if (mobility=3 and selfcare=1 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.332;
if (mobility=3 and selfcare=1 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.318;
if (mobility=3 and selfcare=1 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.237;
if (mobility=3 and selfcare=1 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.153;
if (mobility=3 and selfcare=1 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.364;
if (mobility=3 and selfcare=1 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.308;
```

```
if (mobility=3 and selfcare=1 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.293;
if (mobility=3 and selfcare=1 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.212;
if (mobility=3 and selfcare=1 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.128;
if (mobility=3 and selfcare=1 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.259;
if (mobility=3 and selfcare=1 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.203;
if (mobility=3 and selfcare=1 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.188;
if (mobility=3 and selfcare=1 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.107;
if (mobility=3 and selfcare=1 and activity=5 and pain=4 and anxiety=5) then EQindex = 0.023;
if (mobility=3 and selfcare=1 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.101;
if (mobility=3 and selfcare=1 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.045;
if (mobility=3 and selfcare=1 and activity=5 and pain=5 and anxiety=3) then EQindex = 0.030;
if (mobility=3 and selfcare=1 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.051;
if (mobility=3 and selfcare=1 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.135;
if (mobility=3 and selfcare=2 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.763;
if (mobility=3 and selfcare=2 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.707;
if (mobility=3 and selfcare=2 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.692;
if (mobility=3 and selfcare=2 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.479;
if (mobility=3 and selfcare=2 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.258;
if (mobility=3 and selfcare=2 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.665;
if (mobility=3 and selfcare=2 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.609;
if (mobility=3 and selfcare=2 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.594;
if (mobility=3 and selfcare=2 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.381;
if (mobility=3 and selfcare=2 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.160;
if (mobility=3 and selfcare=2 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.640;
if (mobility=3 and selfcare=2 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.584;
if (mobility=3 and selfcare=2 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.569;
if (mobility=3 and selfcare=2 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.356;
if (mobility=3 and selfcare=2 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.135;
if (mobility=3 and selfcare=2 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.428;
if (mobility=3 and selfcare=2 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.372;
if (mobility=3 and selfcare=2 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.357;
if (mobility=3 and selfcare=2 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.197;
if (mobility=3 and selfcare=2 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.030;
if (mobility=3 and selfcare=2 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.108;
if (mobility=3 and selfcare=2 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.052;
if (mobility=3 and selfcare=2 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.037;
if (mobility=3 and selfcare=2 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.044;
if (mobility=3 and selfcare=2 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.128;
if (mobility=3 and selfcare=2 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.735;
if (mobility=3 and selfcare=2 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.678;
if (mobility=3 and selfcare=2 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.664;
if (mobility=3 and selfcare=2 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.451;
if (mobility=3 and selfcare=2 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.230;
if (mobility=3 and selfcare=2 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.636;
if (mobility=3 and selfcare=2 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.580;
if (mobility=3 and selfcare=2 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.565;
```

```
if (mobility=3 and selfcare=2 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.352;
if (mobility=3 and selfcare=2 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.131;
if (mobility=3 and selfcare=2 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.612;
if (mobility=3 and selfcare=2 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.555;
if (mobility=3 and selfcare=2 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.541;
if (mobility=3 and selfcare=2 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.328;
if (mobility=3 and selfcare=2 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.107;
if (mobility=3 and selfcare=2 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.399;
if (mobility=3 and selfcare=2 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.343;
if (mobility=3 and selfcare=2 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.328;
if (mobility=3 and selfcare=2 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.168;
if (mobility=3 and selfcare=2 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.002;
if (mobility=3 and selfcare=2 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.080;
if (mobility=3 and selfcare=2 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.023;
if (mobility=3 and selfcare=2 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.009;
if (mobility=3 and selfcare=2 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.072;
if (mobility=3 and selfcare=2 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.157;
if (mobility=3 and selfcare=2 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.727;
if (mobility=3 and selfcare=2 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.671;
if (mobility=3 and selfcare=2 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.656;
if (mobility=3 and selfcare=2 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.443;
if (mobility=3 and selfcare=2 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.222;
if (mobility=3 and selfcare=2 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.629;
if (mobility=3 and selfcare=2 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.573;
if (mobility=3 and selfcare=2 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.558;
if (mobility=3 and selfcare=2 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.345;
if (mobility=3 and selfcare=2 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.124;
if (mobility=3 and selfcare=2 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.604;
if (mobility=3 and selfcare=2 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.548;
if (mobility=3 and selfcare=2 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.533;
if (mobility=3 and selfcare=2 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.320;
if (mobility=3 and selfcare=2 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.099;
if (mobility=3 and selfcare=2 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.392;
if (mobility=3 and selfcare=2 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.336;
if (mobility=3 and selfcare=2 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.321;
if (mobility=3 and selfcare=2 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.161;
if (mobility=3 and selfcare=2 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.006;
if (mobility=3 and selfcare=2 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.072;
if (mobility=3 and selfcare=2 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.016;
if (mobility=3 and selfcare=2 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.001;
if (mobility=3 and selfcare=2 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.080;
if (mobility=3 and selfcare=2 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.164;
if (mobility=3 and selfcare=2 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.620;
if (mobility=3 and selfcare=2 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.564;
if (mobility=3 and selfcare=2 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.549;
if (mobility=3 and selfcare=2 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.379;
```

```
if (mobility=3 and selfcare=2 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.203;
if (mobility=3 and selfcare=2 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.522;
if (mobility=3 and selfcare=2 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.465;
if (mobility=3 and selfcare=2 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.451;
if (mobility=3 and selfcare=2 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.281;
if (mobility=3 and selfcare=2 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.105;
if (mobility=3 and selfcare=2 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.497;
if (mobility=3 and selfcare=2 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.441;
if (mobility=3 and selfcare=2 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.426;
if (mobility=3 and selfcare=2 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.256;
if (mobility=3 and selfcare=2 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.080;
if (mobility=3 and selfcare=2 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.320;
if (mobility=3 and selfcare=2 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.263;
if (mobility=3 and selfcare=2 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.249;
if (mobility=3 and selfcare=2 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.115;
if (mobility=3 and selfcare=2 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.025;
if (mobility=3 and selfcare=2 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.053;
if (mobility=3 and selfcare=2 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.003;
if (mobility=3 and selfcare=2 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.018;
if (mobility=3 and selfcare=2 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.099;
if (mobility=3 and selfcare=2 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.183;
if (mobility=3 and selfcare=2 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.400;
if (mobility=3 and selfcare=2 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.344;
if (mobility=3 and selfcare=2 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.329;
if (mobility=3 and selfcare=2 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.248;
if (mobility=3 and selfcare=2 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.164;
if (mobility=3 and selfcare=2 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.302;
if (mobility=3 and selfcare=2 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.246;
if (mobility=3 and selfcare=2 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.231;
if (mobility=3 and selfcare=2 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.150;
if (mobility=3 and selfcare=2 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.066;
if (mobility=3 and selfcare=2 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.277;
if (mobility=3 and selfcare=2 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.221;
if (mobility=3 and selfcare=2 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.206;
if (mobility=3 and selfcare=2 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.125;
if (mobility=3 and selfcare=2 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.041;
if (mobility=3 and selfcare=2 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.172;
if (mobility=3 and selfcare=2 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.116;
if (mobility=3 and selfcare=2 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.101;
if (mobility=3 and selfcare=2 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.020;
if (mobility=3 and selfcare=2 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.064;
if (mobility=3 and selfcare=2 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.014;
if (mobility=3 and selfcare=2 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.042;
if (mobility=3 and selfcare=2 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.057;
if (mobility=3 and selfcare=2 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.138;
if (mobility=3 and selfcare=2 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.222;
```

```
if (mobility=3 and selfcare=3 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.746;
if (mobility=3 and selfcare=3 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.690;
if (mobility=3 and selfcare=3 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.675;
if (mobility=3 and selfcare=3 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.462;
if (mobility=3 and selfcare=3 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.241;
if (mobility=3 and selfcare=3 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.648;
if (mobility=3 and selfcare=3 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.591;
if (mobility=3 and selfcare=3 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.577;
if (mobility=3 and selfcare=3 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.364;
if (mobility=3 and selfcare=3 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.143;
if (mobility=3 and selfcare=3 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.623;
if (mobility=3 and selfcare=3 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.567;
if (mobility=3 and selfcare=3 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.552;
if (mobility=3 and selfcare=3 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.339;
if (mobility=3 and selfcare=3 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.118;
if (mobility=3 and selfcare=3 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.411;
if (mobility=3 and selfcare=3 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.354;
if (mobility=3 and selfcare=3 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.340;
if (mobility=3 and selfcare=3 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.179;
if (mobility=3 and selfcare=3 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.013;
if (mobility=3 and selfcare=3 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.091;
if (mobility=3 and selfcare=3 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.035;
if (mobility=3 and selfcare=3 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.020;
if (mobility=3 and selfcare=3 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.061;
if (mobility=3 and selfcare=3 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.145;
if (mobility=3 and selfcare=3 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.717;
if (mobility=3 and selfcare=3 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.661;
if (mobility=3 and selfcare=3 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.646;
if (mobility=3 and selfcare=3 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.433;
if (mobility=3 and selfcare=3 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.212;
if (mobility=3 and selfcare=3 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.619;
if (mobility=3 and selfcare=3 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.562;
if (mobility=3 and selfcare=3 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.548;
if (mobility=3 and selfcare=3 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.335;
if (mobility=3 and selfcare=3 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.114;
if (mobility=3 and selfcare=3 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.594;
if (mobility=3 and selfcare=3 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.538;
if (mobility=3 and selfcare=3 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.523;
if (mobility=3 and selfcare=3 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.310;
if (mobility=3 and selfcare=3 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.089;
if (mobility=3 and selfcare=3 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.382;
if (mobility=3 and selfcare=3 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.325;
if (mobility=3 and selfcare=3 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.311;
if (mobility=3 and selfcare=3 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.150;
if (mobility=3 and selfcare=3 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.016;
if (mobility=3 and selfcare=3 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.062;
```

```
if (mobility=3 and selfcare=3 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.006;
if (mobility=3 and selfcare=3 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.009;
if (mobility=3 and selfcare=3 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.090;
if (mobility=3 and selfcare=3 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.174;
if (mobility=3 and selfcare=3 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.710;
if (mobility=3 and selfcare=3 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.654;
if (mobility=3 and selfcare=3 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.639;
if (mobility=3 and selfcare=3 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.426;
if (mobility=3 and selfcare=3 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.205;
if (mobility=3 and selfcare=3 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.612;
if (mobility=3 and selfcare=3 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.555;
if (mobility=3 and selfcare=3 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.541;
if (mobility=3 and selfcare=3 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.328;
if (mobility=3 and selfcare=3 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.107;
if (mobility=3 and selfcare=3 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.587;
if (mobility=3 and selfcare=3 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.531;
if (mobility=3 and selfcare=3 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.516;
if (mobility=3 and selfcare=3 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.303;
if (mobility=3 and selfcare=3 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.082;
if (mobility=3 and selfcare=3 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.375;
if (mobility=3 and selfcare=3 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.318;
if (mobility=3 and selfcare=3 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.304;
if (mobility=3 and selfcare=3 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.143;
if (mobility=3 and selfcare=3 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.023;
if (mobility=3 and selfcare=3 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.055;
if (mobility=3 and selfcare=3 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.001;
if (mobility=3 and selfcare=3 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.016;
if (mobility=3 and selfcare=3 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.097;
if (mobility=3 and selfcare=3 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.181;
if (mobility=3 and selfcare=3 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.603;
if (mobility=3 and selfcare=3 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.546;
if (mobility=3 and selfcare=3 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.532;
if (mobility=3 and selfcare=3 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.362;
if (mobility=3 and selfcare=3 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.186;
if (mobility=3 and selfcare=3 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.504;
if (mobility=3 and selfcare=3 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.448;
if (mobility=3 and selfcare=3 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.433;
if (mobility=3 and selfcare=3 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.264;
if (mobility=3 and selfcare=3 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.087;
if (mobility=3 and selfcare=3 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.480;
if (mobility=3 and selfcare=3 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.423;
if (mobility=3 and selfcare=3 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.409;
if (mobility=3 and selfcare=3 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.239;
if (mobility=3 and selfcare=3 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.063;
if (mobility=3 and selfcare=3 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.302;
if (mobility=3 and selfcare=3 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.246;
```

```
if (mobility=3 and selfcare=3 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.231;
if (mobility=3 and selfcare=3 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.097;
if (mobility=3 and selfcare=3 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.042;
if (mobility=3 and selfcare=3 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.036;
if (mobility=3 and selfcare=3 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.020;
if (mobility=3 and selfcare=3 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.035;
if (mobility=3 and selfcare=3 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.116;
if (mobility=3 and selfcare=3 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.200;
if (mobility=3 and selfcare=3 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.383;
if (mobility=3 and selfcare=3 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.327;
if (mobility=3 and selfcare=3 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.312;
if (mobility=3 and selfcare=3 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.231;
if (mobility=3 and selfcare=3 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.147;
if (mobility=3 and selfcare=3 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.285;
if (mobility=3 and selfcare=3 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.228;
if (mobility=3 and selfcare=3 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.214;
if (mobility=3 and selfcare=3 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.133;
if (mobility=3 and selfcare=3 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.049;
if (mobility=3 and selfcare=3 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.260;
if (mobility=3 and selfcare=3 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.204;
if (mobility=3 and selfcare=3 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.189;
if (mobility=3 and selfcare=3 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.108;
if (mobility=3 and selfcare=3 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.024;
if (mobility=3 and selfcare=3 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.155;
if (mobility=3 and selfcare=3 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.099;
if (mobility=3 and selfcare=3 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.084;
if (mobility=3 and selfcare=3 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.003;
if (mobility=3 and selfcare=3 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.081;
if (mobility=3 and selfcare=3 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.003;
if (mobility=3 and selfcare=3 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.059;
if (mobility=3 and selfcare=3 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.074;
if (mobility=3 and selfcare=3 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.155;
if (mobility=3 and selfcare=3 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.239;
if (mobility=3 and selfcare=4 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.654;
if (mobility=3 and selfcare=4 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.598;
if (mobility=3 and selfcare=4 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.583;
if (mobility=3 and selfcare=4 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.402;
if (mobility=3 and selfcare=4 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.214;
if (mobility=3 and selfcare=4 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.555;
if (mobility=3 and selfcare=4 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.499;
if (mobility=3 and selfcare=4 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.484;
if (mobility=3 and selfcare=4 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.304;
if (mobility=3 and selfcare=4 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.116;
if (mobility=3 and selfcare=4 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.531;
if (mobility=3 and selfcare=4 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.475;
if (mobility=3 and selfcare=4 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.460;
```

```
if (mobility=3 and selfcare=4 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.279;
if (mobility=3 and selfcare=4 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.091;
if (mobility=3 and selfcare=4 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.345;
if (mobility=3 and selfcare=4 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.288;
if (mobility=3 and selfcare=4 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.274;
if (mobility=3 and selfcare=4 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.133;
if (mobility=3 and selfcare=4 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.014;
if (mobility=3 and selfcare=4 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.064;
if (mobility=3 and selfcare=4 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.008;
if (mobility=3 and selfcare=4 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.007;
if (mobility=3 and selfcare=4 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.088;
if (mobility=3 and selfcare=4 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.172;
if (mobility=3 and selfcare=4 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.625;
if (mobility=3 and selfcare=4 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.569;
if (mobility=3 and selfcare=4 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.554;
if (mobility=3 and selfcare=4 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.373;
if (mobility=3 and selfcare=4 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.185;
if (mobility=3 and selfcare=4 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.527;
if (mobility=3 and selfcare=4 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.470;
if (mobility=3 and selfcare=4 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.456;
if (mobility=3 and selfcare=4 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.275;
if (mobility=3 and selfcare=4 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.087;
if (mobility=3 and selfcare=4 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.502;
if (mobility=3 and selfcare=4 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.446;
if (mobility=3 and selfcare=4 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.431;
if (mobility=3 and selfcare=4 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.250;
if (mobility=3 and selfcare=4 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.062;
if (mobility=3 and selfcare=4 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.316;
if (mobility=3 and selfcare=4 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.259;
if (mobility=3 and selfcare=4 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.245;
if (mobility=3 and selfcare=4 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.104;
if (mobility=3 and selfcare=4 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.043;
if (mobility=3 and selfcare=4 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.035;
if (mobility=3 and selfcare=4 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.021;
if (mobility=3 and selfcare=4 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.036;
if (mobility=3 and selfcare=4 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.117;
if (mobility=3 and selfcare=4 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.201;
if (mobility=3 and selfcare=4 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.618;
if (mobility=3 and selfcare=4 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.562;
if (mobility=3 and selfcare=4 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.547;
if (mobility=3 and selfcare=4 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.366;
if (mobility=3 and selfcare=4 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.178;
if (mobility=3 and selfcare=4 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.519;
if (mobility=3 and selfcare=4 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.463;
if (mobility=3 and selfcare=4 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.448;
if (mobility=3 and selfcare=4 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.268;
```

```
if (mobility=3 and selfcare=4 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.080;
if (mobility=3 and selfcare=4 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.495;
if (mobility=3 and selfcare=4 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.439;
if (mobility=3 and selfcare=4 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.424;
if (mobility=3 and selfcare=4 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.243;
if (mobility=3 and selfcare=4 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.055;
if (mobility=3 and selfcare=4 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.309;
if (mobility=3 and selfcare=4 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.252;
if (mobility=3 and selfcare=4 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.238;
if (mobility=3 and selfcare=4 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.097;
if (mobility=3 and selfcare=4 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.050;
if (mobility=3 and selfcare=4 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.028;
if (mobility=3 and selfcare=4 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.028;
if (mobility=3 and selfcare=4 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.043;
if (mobility=3 and selfcare=4 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.124;
if (mobility=3 and selfcare=4 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.208;
if (mobility=3 and selfcare=4 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.532;
if (mobility=3 and selfcare=4 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.476;
if (mobility=3 and selfcare=4 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.461;
if (mobility=3 and selfcare=4 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.313;
if (mobility=3 and selfcare=4 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.159;
if (mobility=3 and selfcare=4 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.433;
if (mobility=3 and selfcare=4 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.377;
if (mobility=3 and selfcare=4 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.362;
if (mobility=3 and selfcare=4 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.214;
if (mobility=3 and selfcare=4 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.061;
if (mobility=3 and selfcare=4 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.409;
if (mobility=3 and selfcare=4 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.353;
if (mobility=3 and selfcare=4 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.338;
if (mobility=3 and selfcare=4 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.190;
if (mobility=3 and selfcare=4 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.036;
if (mobility=3 and selfcare=4 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.249;
if (mobility=3 and selfcare=4 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.193;
if (mobility=3 and selfcare=4 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.178;
if (mobility=3 and selfcare=4 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.057;
if (mobility=3 and selfcare=4 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.069;
if (mobility=3 and selfcare=4 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.009;
if (mobility=3 and selfcare=4 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.047;
if (mobility=3 and selfcare=4 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.062;
if (mobility=3 and selfcare=4 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.143;
if (mobility=3 and selfcare=4 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.227;
if (mobility=3 and selfcare=4 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.356;
if (mobility=3 and selfcare=4 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.300;
if (mobility=3 and selfcare=4 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.285;
if (mobility=3 and selfcare=4 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.204;
if (mobility=3 and selfcare=4 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.120;
```

```
if (mobility=3 and selfcare=4 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.258;
if (mobility=3 and selfcare=4 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.201;
if (mobility=3 and selfcare=4 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.187;
if (mobility=3 and selfcare=4 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.106;
if (mobility=3 and selfcare=4 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.022;
if (mobility=3 and selfcare=4 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.233;
if (mobility=3 and selfcare=4 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.177;
if (mobility=3 and selfcare=4 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.162;
if (mobility=3 and selfcare=4 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.081;
if (mobility=3 and selfcare=4 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.003;
if (mobility=3 and selfcare=4 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.128;
if (mobility=3 and selfcare=4 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.072;
if (mobility=3 and selfcare=4 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.057;
if (mobility=3 and selfcare=4 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.024;
if (mobility=3 and selfcare=4 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.108;
if (mobility=3 and selfcare=4 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.030;
if (mobility=3 and selfcare=4 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.086;
if (mobility=3 and selfcare=4 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.101;
if (mobility=3 and selfcare=4 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.182;
if (mobility=3 and selfcare=4 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.266;
if (mobility=3 and selfcare=5 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.367;
if (mobility=3 and selfcare=5 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.311;
if (mobility=3 and selfcare=5 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.296;
if (mobility=3 and selfcare=5 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.215;
if (mobility=3 and selfcare=5 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.131;
if (mobility=3 and selfcare=5 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.269;
if (mobility=3 and selfcare=5 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.212;
if (mobility=3 and selfcare=5 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.198;
if (mobility=3 and selfcare=5 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.117;
if (mobility=3 and selfcare=5 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.033;
if (mobility=3 and selfcare=5 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.244;
if (mobility=3 and selfcare=5 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.188;
if (mobility=3 and selfcare=5 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.173;
if (mobility=3 and selfcare=5 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.092;
if (mobility=3 and selfcare=5 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.008;
if (mobility=3 and selfcare=5 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.139;
if (mobility=3 and selfcare=5 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.083;
if (mobility=3 and selfcare=5 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.068;
if (mobility=3 and selfcare=5 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.013;
if (mobility=3 and selfcare=5 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.097;
if (mobility=3 and selfcare=5 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.019;
if (mobility=3 and selfcare=5 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.075;
if (mobility=3 and selfcare=5 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.090;
if (mobility=3 and selfcare=5 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.171;
if (mobility=3 and selfcare=5 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.255;
if (mobility=3 and selfcare=5 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.338;
```

```
if (mobility=3 and selfcare=5 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.282;
if (mobility=3 and selfcare=5 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.267;
if (mobility=3 and selfcare=5 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.186;
if (mobility=3 and selfcare=5 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.102;
if (mobility=3 and selfcare=5 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.240;
if (mobility=3 and selfcare=5 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.183;
if (mobility=3 and selfcare=5 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.169;
if (mobility=3 and selfcare=5 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.088;
if (mobility=3 and selfcare=5 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.004;
if (mobility=3 and selfcare=5 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.215;
if (mobility=3 and selfcare=5 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.159;
if (mobility=3 and selfcare=5 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.144;
if (mobility=3 and selfcare=5 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.063;
if (mobility=3 and selfcare=5 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.021;
if (mobility=3 and selfcare=5 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.110;
if (mobility=3 and selfcare=5 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.054;
if (mobility=3 and selfcare=5 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.039;
if (mobility=3 and selfcare=5 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.042;
if (mobility=3 and selfcare=5 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.126;
if (mobility=3 and selfcare=5 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.048;
if (mobility=3 and selfcare=5 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.104;
if (mobility=3 and selfcare=5 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.119;
if (mobility=3 and selfcare=5 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.200;
if (mobility=3 and selfcare=5 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.284;
if (mobility=3 and selfcare=5 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.331;
if (mobility=3 and selfcare=5 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.275;
if (mobility=3 and selfcare=5 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.260;
if (mobility=3 and selfcare=5 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.179;
if (mobility=3 and selfcare=5 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.095;
if (mobility=3 and selfcare=5 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.233;
if (mobility=3 and selfcare=5 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.176;
if (mobility=3 and selfcare=5 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.162;
if (mobility=3 and selfcare=5 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.081;
if (mobility=3 and selfcare=5 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.004;
if (mobility=3 and selfcare=5 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.208;
if (mobility=3 and selfcare=5 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.152;
if (mobility=3 and selfcare=5 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.137;
if (mobility=3 and selfcare=5 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.056;
if (mobility=3 and selfcare=5 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.028;
if (mobility=3 and selfcare=5 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.103;
if (mobility=3 and selfcare=5 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.047;
if (mobility=3 and selfcare=5 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.032;
if (mobility=3 and selfcare=5 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.049;
if (mobility=3 and selfcare=5 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.133;
if (mobility=3 and selfcare=5 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.055;
if (mobility=3 and selfcare=5 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.111;
```

```
if (mobility=3 and selfcare=5 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.126;
if (mobility=3 and selfcare=5 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.207;
if (mobility=3 and selfcare=5 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.291;
if (mobility=3 and selfcare=5 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.312;
if (mobility=3 and selfcare=5 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.256;
if (mobility=3 and selfcare=5 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.241;
if (mobility=3 and selfcare=5 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.160;
if (mobility=3 and selfcare=5 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.076;
if (mobility=3 and selfcare=5 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.213;
if (mobility=3 and selfcare=5 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.157;
if (mobility=3 and selfcare=5 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.142;
if (mobility=3 and selfcare=5 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.061;
if (mobility=3 and selfcare=5 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.023;
if (mobility=3 and selfcare=5 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.189;
if (mobility=3 and selfcare=5 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.133;
if (mobility=3 and selfcare=5 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.118;
if (mobility=3 and selfcare=5 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.037;
if (mobility=3 and selfcare=5 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.047;
if (mobility=3 and selfcare=5 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.084;
if (mobility=3 and selfcare=5 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.028;
if (mobility=3 and selfcare=5 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.013;
if (mobility=3 and selfcare=5 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.068;
if (mobility=3 and selfcare=5 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.152;
if (mobility=3 and selfcare=5 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.074;
if (mobility=3 and selfcare=5 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.130;
if (mobility=3 and selfcare=5 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.145;
if (mobility=3 and selfcare=5 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.226;
if (mobility=3 and selfcare=5 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.310;
if (mobility=3 and selfcare=5 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.273;
if (mobility=3 and selfcare=5 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.217;
if (mobility=3 and selfcare=5 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.202;
if (mobility=3 and selfcare=5 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.121;
if (mobility=3 and selfcare=5 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.037;
if (mobility=3 and selfcare=5 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.175;
if (mobility=3 and selfcare=5 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.118;
if (mobility=3 and selfcare=5 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.104;
if (mobility=3 and selfcare=5 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.023;
if (mobility=3 and selfcare=5 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.062;
if (mobility=3 and selfcare=5 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.150;
if (mobility=3 and selfcare=5 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.094;
if (mobility=3 and selfcare=5 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.079;
if (mobility=3 and selfcare=5 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.002;
if (mobility=3 and selfcare=5 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.086;
if (mobility=3 and selfcare=5 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.045;
if (mobility=3 and selfcare=5 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.011;
if (mobility=3 and selfcare=5 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.026;
```

```
if (mobility=3 and selfcare=5 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.107;
if (mobility=3 and selfcare=5 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.191;
if (mobility=3 and selfcare=5 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.113;
if (mobility=3 and selfcare=5 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.169;
if (mobility=3 and selfcare=5 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.184;
if (mobility=3 and selfcare=5 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.265;
if (mobility=3 and selfcare=5 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.349;
if (mobility=4 and selfcare=1 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.813;
if (mobility=4 and selfcare=1 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.757;
if (mobility=4 and selfcare=1 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.742;
if (mobility=4 and selfcare=1 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.539;
if (mobility=4 and selfcare=1 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.327;
if (mobility=4 and selfcare=1 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.714;
if (mobility=4 and selfcare=1 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.658;
if (mobility=4 and selfcare=1 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.643;
if (mobility=4 and selfcare=1 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.440;
if (mobility=4 and selfcare=1 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.229;
if (mobility=4 and selfcare=1 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.690;
if (mobility=4 and selfcare=1 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.634;
if (mobility=4 and selfcare=1 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.619;
if (mobility=4 and selfcare=1 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.416;
if (mobility=4 and selfcare=1 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.204;
if (mobility=4 and selfcare=1 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.485;
if (mobility=4 and selfcare=1 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.429;
if (mobility=4 and selfcare=1 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.414;
if (mobility=4 and selfcare=1 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.260;
if (mobility=4 and selfcare=1 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.099;
if (mobility=4 and selfcare=1 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.177;
if (mobility=4 and selfcare=1 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.121;
if (mobility=4 and selfcare=1 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.106;
if (mobility=4 and selfcare=1 and activity=1 and pain=5 and anxiety=4) then EQindex = 0.025;
if (mobility=4 and selfcare=1 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.059;
if (mobility=4 and selfcare=1 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.784;
if (mobility=4 and selfcare=1 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.728;
if (mobility=4 and selfcare=1 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.713;
if (mobility=4 and selfcare=1 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.510;
if (mobility=4 and selfcare=1 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.299;
if (mobility=4 and selfcare=1 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.686;
if (mobility=4 and selfcare=1 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.629;
if (mobility=4 and selfcare=1 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.615;
if (mobility=4 and selfcare=1 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.411;
if (mobility=4 and selfcare=1 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.200;
if (mobility=4 and selfcare=1 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.661;
if (mobility=4 and selfcare=1 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.605;
if (mobility=4 and selfcare=1 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.590;
if (mobility=4 and selfcare=1 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.387;
```

```
if (mobility=4 and selfcare=1 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.176;
if (mobility=4 and selfcare=1 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.456;
if (mobility=4 and selfcare=1 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.400;
if (mobility=4 and selfcare=1 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.385;
if (mobility=4 and selfcare=1 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.231;
if (mobility=4 and selfcare=1 and activity=2 and pain=4 and anxiety=5) then EQindex = 0.070;
if (mobility=4 and selfcare=1 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.149;
if (mobility=4 and selfcare=1 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.092;
if (mobility=4 and selfcare=1 and activity=2 and pain=5 and anxiety=3) then EQindex = 0.078;
if (mobility=4 and selfcare=1 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.004;
if (mobility=4 and selfcare=1 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.088;
if (mobility=4 and selfcare=1 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.777;
if (mobility=4 and selfcare=1 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.721;
if (mobility=4 and selfcare=1 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.706;
if (mobility=4 and selfcare=1 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.503;
if (mobility=4 and selfcare=1 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.291;
if (mobility=4 and selfcare=1 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.678;
if (mobility=4 and selfcare=1 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.622;
if (mobility=4 and selfcare=1 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.607;
if (mobility=4 and selfcare=1 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.404;
if (mobility=4 and selfcare=1 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.193;
if (mobility=4 and selfcare=1 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.654;
if (mobility=4 and selfcare=1 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.598;
if (mobility=4 and selfcare=1 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.583;
if (mobility=4 and selfcare=1 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.380;
if (mobility=4 and selfcare=1 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.168;
if (mobility=4 and selfcare=1 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.449;
if (mobility=4 and selfcare=1 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.393;
if (mobility=4 and selfcare=1 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.378;
if (mobility=4 and selfcare=1 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.224;
if (mobility=4 and selfcare=1 and activity=3 and pain=4 and anxiety=5) then EQindex = 0.063;
if (mobility=4 and selfcare=1 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.141;
if (mobility=4 and selfcare=1 and activity=3 and pain=5 and anxiety=2) then EQindex = 0.085;
if (mobility=4 and selfcare=1 and activity=3 and pain=5 and anxiety=3) then EQindex = 0.070;
if (mobility=4 and selfcare=1 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.011;
if (mobility=4 and selfcare=1 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.095;
if (mobility=4 and selfcare=1 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.676;
if (mobility=4 and selfcare=1 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.620;
if (mobility=4 and selfcare=1 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.605;
if (mobility=4 and selfcare=1 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.442;
if (mobility=4 and selfcare=1 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.272;
if (mobility=4 and selfcare=1 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.577;
if (mobility=4 and selfcare=1 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.521;
if (mobility=4 and selfcare=1 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.506;
if (mobility=4 and selfcare=1 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.343;
if (mobility=4 and selfcare=1 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.174;
```

```
if (mobility=4 and selfcare=1 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.553;
if (mobility=4 and selfcare=1 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.497;
if (mobility=4 and selfcare=1 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.482;
if (mobility=4 and selfcare=1 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.319;
if (mobility=4 and selfcare=1 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.149;
if (mobility=4 and selfcare=1 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.381;
if (mobility=4 and selfcare=1 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.325;
if (mobility=4 and selfcare=1 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.310;
if (mobility=4 and selfcare=1 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.180;
if (mobility=4 and selfcare=1 and activity=4 and pain=4 and anxiety=5) then EQindex = 0.044;
if (mobility=4 and selfcare=1 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.122;
if (mobility=4 and selfcare=1 and activity=4 and pain=5 and anxiety=2) then EQindex = 0.066;
if (mobility=4 and selfcare=1 and activity=4 and pain=5 and anxiety=3) then EQindex = 0.051;
if (mobility=4 and selfcare=1 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.030;
if (mobility=4 and selfcare=1 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.114;
if (mobility=4 and selfcare=1 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.469;
if (mobility=4 and selfcare=1 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.413;
if (mobility=4 and selfcare=1 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.398;
if (mobility=4 and selfcare=1 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.317;
if (mobility=4 and selfcare=1 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.233;
if (mobility=4 and selfcare=1 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.371;
if (mobility=4 and selfcare=1 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.315;
if (mobility=4 and selfcare=1 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.300;
if (mobility=4 and selfcare=1 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.219;
if (mobility=4 and selfcare=1 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.135;
if (mobility=4 and selfcare=1 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.346;
if (mobility=4 and selfcare=1 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.290;
if (mobility=4 and selfcare=1 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.275;
if (mobility=4 and selfcare=1 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.194;
if (mobility=4 and selfcare=1 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.110;
if (mobility=4 and selfcare=1 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.241;
if (mobility=4 and selfcare=1 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.185;
if (mobility=4 and selfcare=1 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.170;
if (mobility=4 and selfcare=1 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.089;
if (mobility=4 and selfcare=1 and activity=5 and pain=4 and anxiety=5) then EQindex = 0.005;
if (mobility=4 and selfcare=1 and activity=5 and pain=5 and anxiety=1) then EQindex = 0.083;
if (mobility=4 and selfcare=1 and activity=5 and pain=5 and anxiety=2) then EQindex = 0.027;
if (mobility=4 and selfcare=1 and activity=5 and pain=5 and anxiety=3) then EQindex = 0.012;
if (mobility=4 and selfcare=1 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.069;
if (mobility=4 and selfcare=1 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.153;
if (mobility=4 and selfcare=2 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.726;
if (mobility=4 and selfcare=2 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.670;
if (mobility=4 and selfcare=2 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.655;
if (mobility=4 and selfcare=2 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.452;
if (mobility=4 and selfcare=2 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.241;
if (mobility=4 and selfcare=2 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.628;
```

```
if (mobility=4 and selfcare=2 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.572;
if (mobility=4 and selfcare=2 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.557;
if (mobility=4 and selfcare=2 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.353;
if (mobility=4 and selfcare=2 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.142;
if (mobility=4 and selfcare=2 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.603;
if (mobility=4 and selfcare=2 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.547;
if (mobility=4 and selfcare=2 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.532;
if (mobility=4 and selfcare=2 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.329;
if (mobility=4 and selfcare=2 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.118;
if (mobility=4 and selfcare=2 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.399;
if (mobility=4 and selfcare=2 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.342;
if (mobility=4 and selfcare=2 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.328;
if (mobility=4 and selfcare=2 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.173;
if (mobility=4 and selfcare=2 and activity=1 and pain=4 and anxiety=5) then EQindex = 0.013;
if (mobility=4 and selfcare=2 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.091;
if (mobility=4 and selfcare=2 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.034;
if (mobility=4 and selfcare=2 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.020;
if (mobility=4 and selfcare=2 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.061;
if (mobility=4 and selfcare=2 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.145;
if (mobility=4 and selfcare=2 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.698;
if (mobility=4 and selfcare=2 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.641;
if (mobility=4 and selfcare=2 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.627;
if (mobility=4 and selfcare=2 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.423;
if (mobility=4 and selfcare=2 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.212;
if (mobility=4 and selfcare=2 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.599;
if (mobility=4 and selfcare=2 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.543;
if (mobility=4 and selfcare=2 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.528;
if (mobility=4 and selfcare=2 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.325;
if (mobility=4 and selfcare=2 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.113;
if (mobility=4 and selfcare=2 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.575;
if (mobility=4 and selfcare=2 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.518;
if (mobility=4 and selfcare=2 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.504;
if (mobility=4 and selfcare=2 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.300;
if (mobility=4 and selfcare=2 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.089;
if (mobility=4 and selfcare=2 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.370;
if (mobility=4 and selfcare=2 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.313;
if (mobility=4 and selfcare=2 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.299;
if (mobility=4 and selfcare=2 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.144;
if (mobility=4 and selfcare=2 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.016;
if (mobility=4 and selfcare=2 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.062;
if (mobility=4 and selfcare=2 and activity=2 and pain=5 and anxiety=2) then EQindex = 0.006;
if (mobility=4 and selfcare=2 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.009;
if (mobility=4 and selfcare=2 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.090;
if (mobility=4 and selfcare=2 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.174;
if (mobility=4 and selfcare=2 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.690;
if (mobility=4 and selfcare=2 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.634;
```

```
if (mobility=4 and selfcare=2 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.619;
if (mobility=4 and selfcare=2 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.416;
if (mobility=4 and selfcare=2 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.205;
if (mobility=4 and selfcare=2 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.592;
if (mobility=4 and selfcare=2 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.536;
if (mobility=4 and selfcare=2 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.521;
if (mobility=4 and selfcare=2 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.317;
if (mobility=4 and selfcare=2 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.106;
if (mobility=4 and selfcare=2 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.567;
if (mobility=4 and selfcare=2 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.511;
if (mobility=4 and selfcare=2 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.496;
if (mobility=4 and selfcare=2 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.293;
if (mobility=4 and selfcare=2 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.082;
if (mobility=4 and selfcare=2 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.363;
if (mobility=4 and selfcare=2 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.306;
if (mobility=4 and selfcare=2 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.292;
if (mobility=4 and selfcare=2 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.137;
if (mobility=4 and selfcare=2 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.023;
if (mobility=4 and selfcare=2 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.055;
if (mobility=4 and selfcare=2 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.002;
if (mobility=4 and selfcare=2 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.016;
if (mobility=4 and selfcare=2 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.097;
if (mobility=4 and selfcare=2 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.181;
if (mobility=4 and selfcare=2 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.589;
if (mobility=4 and selfcare=2 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.533;
if (mobility=4 and selfcare=2 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.518;
if (mobility=4 and selfcare=2 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.355;
if (mobility=4 and selfcare=2 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.186;
if (mobility=4 and selfcare=2 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.491;
if (mobility=4 and selfcare=2 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.434;
if (mobility=4 and selfcare=2 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.420;
if (mobility=4 and selfcare=2 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.257;
if (mobility=4 and selfcare=2 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.087;
if (mobility=4 and selfcare=2 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.466;
if (mobility=4 and selfcare=2 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.410;
if (mobility=4 and selfcare=2 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.395;
if (mobility=4 and selfcare=2 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.232;
if (mobility=4 and selfcare=2 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.063;
if (mobility=4 and selfcare=2 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.294;
if (mobility=4 and selfcare=2 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.238;
if (mobility=4 and selfcare=2 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.223;
if (mobility=4 and selfcare=2 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.093;
if (mobility=4 and selfcare=2 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.042;
if (mobility=4 and selfcare=2 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.036;
if (mobility=4 and selfcare=2 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.021;
if (mobility=4 and selfcare=2 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.035;
```

```
if (mobility=4 and selfcare=2 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.116;
if (mobility=4 and selfcare=2 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.200;
if (mobility=4 and selfcare=2 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.383;
if (mobility=4 and selfcare=2 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.326;
if (mobility=4 and selfcare=2 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.312;
if (mobility=4 and selfcare=2 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.231;
if (mobility=4 and selfcare=2 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.147;
if (mobility=4 and selfcare=2 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.284;
if (mobility=4 and selfcare=2 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.228;
if (mobility=4 and selfcare=2 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.213;
if (mobility=4 and selfcare=2 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.132;
if (mobility=4 and selfcare=2 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.048;
if (mobility=4 and selfcare=2 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.260;
if (mobility=4 and selfcare=2 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.203;
if (mobility=4 and selfcare=2 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.189;
if (mobility=4 and selfcare=2 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.108;
if (mobility=4 and selfcare=2 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.024;
if (mobility=4 and selfcare=2 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.155;
if (mobility=4 and selfcare=2 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.098;
if (mobility=4 and selfcare=2 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.084;
if (mobility=4 and selfcare=2 and activity=5 and pain=4 and anxiety=4) then EQindex = 0.003;
if (mobility=4 and selfcare=2 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.081;
if (mobility=4 and selfcare=2 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.003;
if (mobility=4 and selfcare=2 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.060;
if (mobility=4 and selfcare=2 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.074;
if (mobility=4 and selfcare=2 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.155;
if (mobility=4 and selfcare=2 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.239;
if (mobility=4 and selfcare=3 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.709;
if (mobility=4 and selfcare=3 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.653;
if (mobility=4 and selfcare=3 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.638;
if (mobility=4 and selfcare=3 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.435;
if (mobility=4 and selfcare=3 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.223;
if (mobility=4 and selfcare=3 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.610;
if (mobility=4 and selfcare=3 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.554;
if (mobility=4 and selfcare=3 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.539;
if (mobility=4 and selfcare=3 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.336;
if (mobility=4 and selfcare=3 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.125;
if (mobility=4 and selfcare=3 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.586;
if (mobility=4 and selfcare=3 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.530;
if (mobility=4 and selfcare=3 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.515;
if (mobility=4 and selfcare=3 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.312;
if (mobility=4 and selfcare=3 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.100;
if (mobility=4 and selfcare=3 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.381;
if (mobility=4 and selfcare=3 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.325;
if (mobility=4 and selfcare=3 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.310;
if (mobility=4 and selfcare=3 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.156;
```

```
if (mobility=4 and selfcare=3 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.005;
if (mobility=4 and selfcare=3 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.073;
if (mobility=4 and selfcare=3 and activity=1 and pain=5 and anxiety=2) then EQindex = 0.017;
if (mobility=4 and selfcare=3 and activity=1 and pain=5 and anxiety=3) then EQindex = 0.002;
if (mobility=4 and selfcare=3 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.079;
if (mobility=4 and selfcare=3 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.163;
if (mobility=4 and selfcare=3 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.680;
if (mobility=4 and selfcare=3 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.624;
if (mobility=4 and selfcare=3 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.609;
if (mobility=4 and selfcare=3 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.406;
if (mobility=4 and selfcare=3 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.195;
if (mobility=4 and selfcare=3 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.582;
if (mobility=4 and selfcare=3 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.525;
if (mobility=4 and selfcare=3 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.511;
if (mobility=4 and selfcare=3 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.307;
if (mobility=4 and selfcare=3 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.096;
if (mobility=4 and selfcare=3 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.557;
if (mobility=4 and selfcare=3 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.501;
if (mobility=4 and selfcare=3 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.486;
if (mobility=4 and selfcare=3 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.283;
if (mobility=4 and selfcare=3 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.072;
if (mobility=4 and selfcare=3 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.352;
if (mobility=4 and selfcare=3 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.296;
if (mobility=4 and selfcare=3 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.281;
if (mobility=4 and selfcare=3 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.127;
if (mobility=4 and selfcare=3 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.034;
if (mobility=4 and selfcare=3 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.045;
if (mobility=4 and selfcare=3 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.012;
if (mobility=4 and selfcare=3 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.027;
if (mobility=4 and selfcare=3 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.108;
if (mobility=4 and selfcare=3 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.192;
if (mobility=4 and selfcare=3 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.673;
if (mobility=4 and selfcare=3 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.617;
if (mobility=4 and selfcare=3 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.602;
if (mobility=4 and selfcare=3 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.399;
if (mobility=4 and selfcare=3 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.187;
if (mobility=4 and selfcare=3 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.574;
if (mobility=4 and selfcare=3 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.518;
if (mobility=4 and selfcare=3 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.503;
if (mobility=4 and selfcare=3 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.300;
if (mobility=4 and selfcare=3 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.089;
if (mobility=4 and selfcare=3 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.550;
if (mobility=4 and selfcare=3 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.494;
if (mobility=4 and selfcare=3 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.479;
if (mobility=4 and selfcare=3 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.276;
if (mobility=4 and selfcare=3 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.064;
```
```
if (mobility=4 and selfcare=3 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.345;
if (mobility=4 and selfcare=3 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.289;
if (mobility=4 and selfcare=3 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.274;
if (mobility=4 and selfcare=3 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.120;
if (mobility=4 and selfcare=3 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.041;
if (mobility=4 and selfcare=3 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.037;
if (mobility=4 and selfcare=3 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.019;
if (mobility=4 and selfcare=3 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.034;
if (mobility=4 and selfcare=3 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.115;
if (mobility=4 and selfcare=3 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.199;
if (mobility=4 and selfcare=3 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.572;
if (mobility=4 and selfcare=3 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.516;
if (mobility=4 and selfcare=3 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.501;
if (mobility=4 and selfcare=3 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.338;
if (mobility=4 and selfcare=3 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.168;
if (mobility=4 and selfcare=3 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.473;
if (mobility=4 and selfcare=3 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.417;
if (mobility=4 and selfcare=3 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.402;
if (mobility=4 and selfcare=3 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.239;
if (mobility=4 and selfcare=3 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.070;
if (mobility=4 and selfcare=3 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.449;
if (mobility=4 and selfcare=3 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.393;
if (mobility=4 and selfcare=3 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.378;
if (mobility=4 and selfcare=3 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.215;
if (mobility=4 and selfcare=3 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.045;
if (mobility=4 and selfcare=3 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.277;
if (mobility=4 and selfcare=3 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.221;
if (mobility=4 and selfcare=3 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.206;
if (mobility=4 and selfcare=3 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.076;
if (mobility=4 and selfcare=3 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.060;
if (mobility=4 and selfcare=3 and activity=4 and pain=5 and anxiety=1) then EQindex = 0.018;
if (mobility=4 and selfcare=3 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.038;
if (mobility=4 and selfcare=3 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.053;
if (mobility=4 and selfcare=3 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.134;
if (mobility=4 and selfcare=3 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.218;
if (mobility=4 and selfcare=3 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.365;
if (mobility=4 and selfcare=3 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.309;
if (mobility=4 and selfcare=3 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.294;
if (mobility=4 and selfcare=3 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.213;
if (mobility=4 and selfcare=3 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.129;
if (mobility=4 and selfcare=3 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.267;
if (mobility=4 and selfcare=3 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.211;
if (mobility=4 and selfcare=3 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.196;
if (mobility=4 and selfcare=3 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.115;
if (mobility=4 and selfcare=3 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.031;
if (mobility=4 and selfcare=3 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.242;
```

```
if (mobility=4 and selfcare=3 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.186;
if (mobility=4 and selfcare=3 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.171;
if (mobility=4 and selfcare=3 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.090;
if (mobility=4 and selfcare=3 and activity=5 and pain=3 and anxiety=5) then EQindex = 0.006;
if (mobility=4 and selfcare=3 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.137;
if (mobility=4 and selfcare=3 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.081;
if (mobility=4 and selfcare=3 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.066;
if (mobility=4 and selfcare=3 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.015;
if (mobility=4 and selfcare=3 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.099;
if (mobility=4 and selfcare=3 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.021;
if (mobility=4 and selfcare=3 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.077;
if (mobility=4 and selfcare=3 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.092;
if (mobility=4 and selfcare=3 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.173;
if (mobility=4 and selfcare=3 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.257;
if (mobility=4 and selfcare=4 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.622;
if (mobility=4 and selfcare=4 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.565;
if (mobility=4 and selfcare=4 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.551;
if (mobility=4 and selfcare=4 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.377;
if (mobility=4 and selfcare=4 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.197;
if (mobility=4 and selfcare=4 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.523;
if (mobility=4 and selfcare=4 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.467;
if (mobility=4 and selfcare=4 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.452;
if (mobility=4 and selfcare=4 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.278;
if (mobility=4 and selfcare=4 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.098;
if (mobility=4 and selfcare=4 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.499;
if (mobility=4 and selfcare=4 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.442;
if (mobility=4 and selfcare=4 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.428;
if (mobility=4 and selfcare=4 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.254;
if (mobility=4 and selfcare=4 and activity=1 and pain=3 and anxiety=5) then EQindex = 0.074;
if (mobility=4 and selfcare=4 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.318;
if (mobility=4 and selfcare=4 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.262;
if (mobility=4 and selfcare=4 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.247;
if (mobility=4 and selfcare=4 and activity=1 and pain=4 and anxiety=4) then EQindex = 0.110;
if (mobility=4 and selfcare=4 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.032;
if (mobility=4 and selfcare=4 and activity=1 and pain=5 and anxiety=1) then EQindex = 0.047;
if (mobility=4 and selfcare=4 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.010;
if (mobility=4 and selfcare=4 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.024;
if (mobility=4 and selfcare=4 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.105;
if (mobility=4 and selfcare=4 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.189;
if (mobility=4 and selfcare=4 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.593;
if (mobility=4 and selfcare=4 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.536;
if (mobility=4 and selfcare=4 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.522;
if (mobility=4 and selfcare=4 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.348;
if (mobility=4 and selfcare=4 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.168;
if (mobility=4 and selfcare=4 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.494;
if (mobility=4 and selfcare=4 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.438;
```

```
if (mobility=4 and selfcare=4 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.423;
if (mobility=4 and selfcare=4 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.249;
if (mobility=4 and selfcare=4 and activity=2 and pain=2 and anxiety=5) then EQindex = 0.069;
if (mobility=4 and selfcare=4 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.470;
if (mobility=4 and selfcare=4 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.413;
if (mobility=4 and selfcare=4 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.399;
if (mobility=4 and selfcare=4 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.225;
if (mobility=4 and selfcare=4 and activity=2 and pain=3 and anxiety=5) then EQindex = 0.045;
if (mobility=4 and selfcare=4 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.289;
if (mobility=4 and selfcare=4 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.233;
if (mobility=4 and selfcare=4 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.218;
if (mobility=4 and selfcare=4 and activity=2 and pain=4 and anxiety=4) then EQindex = 0.082;
if (mobility=4 and selfcare=4 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.060;
if (mobility=4 and selfcare=4 and activity=2 and pain=5 and anxiety=1) then EQindex = 0.018;
if (mobility=4 and selfcare=4 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.039;
if (mobility=4 and selfcare=4 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.053;
if (mobility=4 and selfcare=4 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.134;
if (mobility=4 and selfcare=4 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.218;
if (mobility=4 and selfcare=4 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.586;
if (mobility=4 and selfcare=4 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.529;
if (mobility=4 and selfcare=4 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.515;
if (mobility=4 and selfcare=4 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.341;
if (mobility=4 and selfcare=4 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.161;
if (mobility=4 and selfcare=4 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.487;
if (mobility=4 and selfcare=4 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.431;
if (mobility=4 and selfcare=4 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.416;
if (mobility=4 and selfcare=4 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.242;
if (mobility=4 and selfcare=4 and activity=3 and pain=2 and anxiety=5) then EQindex = 0.062;
if (mobility=4 and selfcare=4 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.463;
if (mobility=4 and selfcare=4 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.406;
if (mobility=4 and selfcare=4 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.392;
if (mobility=4 and selfcare=4 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.218;
if (mobility=4 and selfcare=4 and activity=3 and pain=3 and anxiety=5) then EQindex = 0.038;
if (mobility=4 and selfcare=4 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.282;
if (mobility=4 and selfcare=4 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.226;
if (mobility=4 and selfcare=4 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.211;
if (mobility=4 and selfcare=4 and activity=3 and pain=4 and anxiety=4) then EQindex = 0.074;
if (mobility=4 and selfcare=4 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.068;
if (mobility=4 and selfcare=4 and activity=3 and pain=5 and anxiety=1) then EQindex = 0.011;
if (mobility=4 and selfcare=4 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.046;
if (mobility=4 and selfcare=4 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.060;
if (mobility=4 and selfcare=4 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.141;
if (mobility=4 and selfcare=4 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.225;
if (mobility=4 and selfcare=4 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.504;
if (mobility=4 and selfcare=4 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.448;
if (mobility=4 and selfcare=4 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.433;
```

```
if (mobility=4 and selfcare=4 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.290;
if (mobility=4 and selfcare=4 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.142;
if (mobility=4 and selfcare=4 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.406;
if (mobility=4 and selfcare=4 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.350;
if (mobility=4 and selfcare=4 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.335;
if (mobility=4 and selfcare=4 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.192;
if (mobility=4 and selfcare=4 and activity=4 and pain=2 and anxiety=5) then EQindex = 0.043;
if (mobility=4 and selfcare=4 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.381;
if (mobility=4 and selfcare=4 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.325;
if (mobility=4 and selfcare=4 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.310;
if (mobility=4 and selfcare=4 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.167;
if (mobility=4 and selfcare=4 and activity=4 and pain=3 and anxiety=5) then EQindex = 0.019;
if (mobility=4 and selfcare=4 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.226;
if (mobility=4 and selfcare=4 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.169;
if (mobility=4 and selfcare=4 and activity=4 and pain=4 and anxiety=3) then EQindex = 0.155;
if (mobility=4 and selfcare=4 and activity=4 and pain=4 and anxiety=4) then EQindex = 0.036;
if (mobility=4 and selfcare=4 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.087;
if (mobility=4 and selfcare=4 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.009;
if (mobility=4 and selfcare=4 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.065;
if (mobility=4 and selfcare=4 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.080;
if (mobility=4 and selfcare=4 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.160;
if (mobility=4 and selfcare=4 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.245;
if (mobility=4 and selfcare=4 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.339;
if (mobility=4 and selfcare=4 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.282;
if (mobility=4 and selfcare=4 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.268;
if (mobility=4 and selfcare=4 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.187;
if (mobility=4 and selfcare=4 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.103;
if (mobility=4 and selfcare=4 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.240;
if (mobility=4 and selfcare=4 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.184;
if (mobility=4 and selfcare=4 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.169;
if (mobility=4 and selfcare=4 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.088;
if (mobility=4 and selfcare=4 and activity=5 and pain=2 and anxiety=5) then EQindex = 0.004;
if (mobility=4 and selfcare=4 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.216;
if (mobility=4 and selfcare=4 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.159;
if (mobility=4 and selfcare=4 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.145;
if (mobility=4 and selfcare=4 and activity=5 and pain=3 and anxiety=4) then EQindex = 0.064;
if (mobility=4 and selfcare=4 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.020;
if (mobility=4 and selfcare=4 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.111;
if (mobility=4 and selfcare=4 and activity=5 and pain=4 and anxiety=2) then EQindex = 0.054;
if (mobility=4 and selfcare=4 and activity=5 and pain=4 and anxiety=3) then EQindex = 0.040;
if (mobility=4 and selfcare=4 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.041;
if (mobility=4 and selfcare=4 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.126;
if (mobility=4 and selfcare=4 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.047;
if (mobility=4 and selfcare=4 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.104;
if (mobility=4 and selfcare=4 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.118;
if (mobility=4 and selfcare=4 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.199;
```

```
if (mobility=4 and selfcare=4 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.283;
if (mobility=4 and selfcare=5 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.349;
if (mobility=4 and selfcare=5 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.293;
if (mobility=4 and selfcare=5 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.278;
if (mobility=4 and selfcare=5 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.197;
if (mobility=4 and selfcare=5 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.113;
if (mobility=4 and selfcare=5 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.251;
if (mobility=4 and selfcare=5 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.195;
if (mobility=4 and selfcare=5 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.180;
if (mobility=4 and selfcare=5 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.099;
if (mobility=4 and selfcare=5 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.015;
if (mobility=4 and selfcare=5 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.226;
if (mobility=4 and selfcare=5 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.170;
if (mobility=4 and selfcare=5 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.155;
if (mobility=4 and selfcare=5 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.074;
if (mobility=4 and selfcare=5 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.010;
if (mobility=4 and selfcare=5 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.121;
if (mobility=4 and selfcare=5 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.065;
if (mobility=4 and selfcare=5 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.050;
if (mobility=4 and selfcare=5 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.031;
if (mobility=4 and selfcare=5 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.115;
if (mobility=4 and selfcare=5 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.037;
if (mobility=4 and selfcare=5 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.093;
if (mobility=4 and selfcare=5 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.108;
if (mobility=4 and selfcare=5 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.189;
if (mobility=4 and selfcare=5 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.273;
if (mobility=4 and selfcare=5 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.321;
if (mobility=4 and selfcare=5 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.264;
if (mobility=4 and selfcare=5 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.250;
if (mobility=4 and selfcare=5 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.169;
if (mobility=4 and selfcare=5 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.085;
if (mobility=4 and selfcare=5 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.222;
if (mobility=4 and selfcare=5 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.166;
if (mobility=4 and selfcare=5 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.151;
if (mobility=4 and selfcare=5 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.070;
if (mobility=4 and selfcare=5 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.014;
if (mobility=4 and selfcare=5 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.198;
if (mobility=4 and selfcare=5 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.141;
if (mobility=4 and selfcare=5 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.127;
if (mobility=4 and selfcare=5 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.046;
if (mobility=4 and selfcare=5 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.039;
if (mobility=4 and selfcare=5 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.092;
if (mobility=4 and selfcare=5 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.036;
if (mobility=4 and selfcare=5 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.021;
if (mobility=4 and selfcare=5 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.060;
if (mobility=4 and selfcare=5 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.144;
```

```
if (mobility=4 and selfcare=5 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.066;
if (mobility=4 and selfcare=5 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.122;
if (mobility=4 and selfcare=5 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.137;
if (mobility=4 and selfcare=5 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.218;
if (mobility=4 and selfcare=5 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.302;
if (mobility=4 and selfcare=5 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.313;
if (mobility=4 and selfcare=5 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.257;
if (mobility=4 and selfcare=5 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.242;
if (mobility=4 and selfcare=5 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.161;
if (mobility=4 and selfcare=5 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.077;
if (mobility=4 and selfcare=5 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.215;
if (mobility=4 and selfcare=5 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.159;
if (mobility=4 and selfcare=5 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.144;
if (mobility=4 and selfcare=5 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.063;
if (mobility=4 and selfcare=5 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.021;
if (mobility=4 and selfcare=5 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.190;
if (mobility=4 and selfcare=5 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.134;
if (mobility=4 and selfcare=5 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.119;
if (mobility=4 and selfcare=5 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.038;
if (mobility=4 and selfcare=5 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.046;
if (mobility=4 and selfcare=5 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.085;
if (mobility=4 and selfcare=5 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.029;
if (mobility=4 and selfcare=5 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.014;
if (mobility=4 and selfcare=5 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.067;
if (mobility=4 and selfcare=5 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.151;
if (mobility=4 and selfcare=5 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.073;
if (mobility=4 and selfcare=5 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.129;
if (mobility=4 and selfcare=5 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.144;
if (mobility=4 and selfcare=5 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.225;
if (mobility=4 and selfcare=5 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.309;
if (mobility=4 and selfcare=5 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.294;
if (mobility=4 and selfcare=5 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.238;
if (mobility=4 and selfcare=5 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.223;
if (mobility=4 and selfcare=5 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.142;
if (mobility=4 and selfcare=5 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.058;
if (mobility=4 and selfcare=5 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.196;
if (mobility=4 and selfcare=5 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.139;
if (mobility=4 and selfcare=5 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.125;
if (mobility=4 and selfcare=5 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.044;
if (mobility=4 and selfcare=5 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.040;
if (mobility=4 and selfcare=5 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.171;
if (mobility=4 and selfcare=5 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.115;
if (mobility=4 and selfcare=5 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.100;
if (mobility=4 and selfcare=5 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.019;
if (mobility=4 and selfcare=5 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.065;
if (mobility=4 and selfcare=5 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.066;
```

```
if (mobility=4 and selfcare=5 and activity=4 and pain=4 and anxiety=2) then EQindex = 0.010;
if (mobility=4 and selfcare=5 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.005;
if (mobility=4 and selfcare=5 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.086;
if (mobility=4 and selfcare=5 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.170;
if (mobility=4 and selfcare=5 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.092;
if (mobility=4 and selfcare=5 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.148;
if (mobility=4 and selfcare=5 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.163;
if (mobility=4 and selfcare=5 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.244;
if (mobility=4 and selfcare=5 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.328;
if (mobility=4 and selfcare=5 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.255;
if (mobility=4 and selfcare=5 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.199;
if (mobility=4 and selfcare=5 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.184;
if (mobility=4 and selfcare=5 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.103;
if (mobility=4 and selfcare=5 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.019;
if (mobility=4 and selfcare=5 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.157;
if (mobility=4 and selfcare=5 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.101;
if (mobility=4 and selfcare=5 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.086;
if (mobility=4 and selfcare=5 and activity=5 and pain=2 and anxiety=4) then EQindex = 0.005;
if (mobility=4 and selfcare=5 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.079;
if (mobility=4 and selfcare=5 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.132;
if (mobility=4 and selfcare=5 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.076;
if (mobility=4 and selfcare=5 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.061;
if (mobility=4 and selfcare=5 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.020;
if (mobility=4 and selfcare=5 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.104;
if (mobility=4 and selfcare=5 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.027;
if (mobility=4 and selfcare=5 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.029;
if (mobility=4 and selfcare=5 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.044;
if (mobility=4 and selfcare=5 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.125;
if (mobility=4 and selfcare=5 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.209;
if (mobility=4 and selfcare=5 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.131;
if (mobility=4 and selfcare=5 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.187;
if (mobility=4 and selfcare=5 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.202;
if (mobility=4 and selfcare=5 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.283;
if (mobility=4 and selfcare=5 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.367;
if (mobility=5 and selfcare=1 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.336;
if (mobility=5 and selfcare=1 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.280;
if (mobility=5 and selfcare=1 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.265;
if (mobility=5 and selfcare=1 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.184;
if (mobility=5 and selfcare=1 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.100;
if (mobility=5 and selfcare=1 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.238;
if (mobility=5 and selfcare=1 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.181;
if (mobility=5 and selfcare=1 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.167;
if (mobility=5 and selfcare=1 and activity=1 and pain=2 and anxiety=4) then EQindex = 0.086;
if (mobility=5 and selfcare=1 and activity=1 and pain=2 and anxiety=5) then EQindex = 0.002;
if (mobility=5 and selfcare=1 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.213;
if (mobility=5 and selfcare=1 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.157;
```

```
if (mobility=5 and selfcare=1 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.142;
if (mobility=5 and selfcare=1 and activity=1 and pain=3 and anxiety=4) then EQindex = 0.061;
if (mobility=5 and selfcare=1 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.023;
if (mobility=5 and selfcare=1 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.108;
if (mobility=5 and selfcare=1 and activity=1 and pain=4 and anxiety=2) then EQindex = 0.052;
if (mobility=5 and selfcare=1 and activity=1 and pain=4 and anxiety=3) then EQindex = 0.037;
if (mobility=5 and selfcare=1 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.044;
if (mobility=5 and selfcare=1 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.128;
if (mobility=5 and selfcare=1 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.050;
if (mobility=5 and selfcare=1 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.106;
if (mobility=5 and selfcare=1 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.121;
if (mobility=5 and selfcare=1 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.202;
if (mobility=5 and selfcare=1 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.286;
if (mobility=5 and selfcare=1 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.307;
if (mobility=5 and selfcare=1 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.251;
if (mobility=5 and selfcare=1 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.236;
if (mobility=5 and selfcare=1 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.155;
if (mobility=5 and selfcare=1 and activity=2 and pain=1 and anxiety=5) then EQindex = 0.071;
if (mobility=5 and selfcare=1 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.209;
if (mobility=5 and selfcare=1 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.152;
if (mobility=5 and selfcare=1 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.138;
if (mobility=5 and selfcare=1 and activity=2 and pain=2 and anxiety=4) then EQindex = 0.057;
if (mobility=5 and selfcare=1 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.027;
if (mobility=5 and selfcare=1 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.184;
if (mobility=5 and selfcare=1 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.128;
if (mobility=5 and selfcare=1 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.113;
if (mobility=5 and selfcare=1 and activity=2 and pain=3 and anxiety=4) then EQindex = 0.032;
if (mobility=5 and selfcare=1 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.052;
if (mobility=5 and selfcare=1 and activity=2 and pain=4 and anxiety=1) then EQindex = 0.079;
if (mobility=5 and selfcare=1 and activity=2 and pain=4 and anxiety=2) then EQindex = 0.023;
if (mobility=5 and selfcare=1 and activity=2 and pain=4 and anxiety=3) then EQindex = 0.008;
if (mobility=5 and selfcare=1 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.073;
if (mobility=5 and selfcare=1 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.157;
if (mobility=5 and selfcare=1 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.079;
if (mobility=5 and selfcare=1 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.135;
if (mobility=5 and selfcare=1 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.150;
if (mobility=5 and selfcare=1 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.231;
if (mobility=5 and selfcare=1 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.315;
if (mobility=5 and selfcare=1 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.300;
if (mobility=5 and selfcare=1 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.244;
if (mobility=5 and selfcare=1 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.229;
if (mobility=5 and selfcare=1 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.148;
if (mobility=5 and selfcare=1 and activity=3 and pain=1 and anxiety=5) then EQindex = 0.064;
if (mobility=5 and selfcare=1 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.202;
if (mobility=5 and selfcare=1 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.145;
if (mobility=5 and selfcare=1 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.131;
```

```
if (mobility=5 and selfcare=1 and activity=3 and pain=2 and anxiety=4) then EQindex = 0.050;
if (mobility=5 and selfcare=1 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.035;
if (mobility=5 and selfcare=1 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.177;
if (mobility=5 and selfcare=1 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.121;
if (mobility=5 and selfcare=1 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.106;
if (mobility=5 and selfcare=1 and activity=3 and pain=3 and anxiety=4) then EQindex = 0.025;
if (mobility=5 and selfcare=1 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.059;
if (mobility=5 and selfcare=1 and activity=3 and pain=4 and anxiety=1) then EQindex = 0.072;
if (mobility=5 and selfcare=1 and activity=3 and pain=4 and anxiety=2) then EQindex = 0.016;
if (mobility=5 and selfcare=1 and activity=3 and pain=4 and anxiety=3) then EQindex = 0.001;
if (mobility=5 and selfcare=1 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.080;
if (mobility=5 and selfcare=1 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.164;
if (mobility=5 and selfcare=1 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.086;
if (mobility=5 and selfcare=1 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.142;
if (mobility=5 and selfcare=1 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.157;
if (mobility=5 and selfcare=1 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.238;
if (mobility=5 and selfcare=1 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.322;
if (mobility=5 and selfcare=1 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.281;
if (mobility=5 and selfcare=1 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.225;
if (mobility=5 and selfcare=1 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.210;
if (mobility=5 and selfcare=1 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.129;
if (mobility=5 and selfcare=1 and activity=4 and pain=1 and anxiety=5) then EQindex = 0.045;
if (mobility=5 and selfcare=1 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.182;
if (mobility=5 and selfcare=1 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.126;
if (mobility=5 and selfcare=1 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.111;
if (mobility=5 and selfcare=1 and activity=4 and pain=2 and anxiety=4) then EQindex = 0.030;
if (mobility=5 and selfcare=1 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.054;
if (mobility=5 and selfcare=1 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.158;
if (mobility=5 and selfcare=1 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.102;
if (mobility=5 and selfcare=1 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.087;
if (mobility=5 and selfcare=1 and activity=4 and pain=3 and anxiety=4) then EQindex = 0.006;
if (mobility=5 and selfcare=1 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.078;
if (mobility=5 and selfcare=1 and activity=4 and pain=4 and anxiety=1) then EQindex = 0.053;
if (mobility=5 and selfcare=1 and activity=4 and pain=4 and anxiety=2) then EQindex = -0.003;
if (mobility=5 and selfcare=1 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.018;
if (mobility=5 and selfcare=1 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.099;
if (mobility=5 and selfcare=1 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.183;
if (mobility=5 and selfcare=1 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.105;
if (mobility=5 and selfcare=1 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.161;
if (mobility=5 and selfcare=1 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.176;
if (mobility=5 and selfcare=1 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.257;
if (mobility=5 and selfcare=1 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.341;
if (mobility=5 and selfcare=1 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.242;
if (mobility=5 and selfcare=1 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.186;
if (mobility=5 and selfcare=1 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.171;
if (mobility=5 and selfcare=1 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.090;
```

```
if (mobility=5 and selfcare=1 and activity=5 and pain=1 and anxiety=5) then EQindex = 0.006;
if (mobility=5 and selfcare=1 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.144;
if (mobility=5 and selfcare=1 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.087;
if (mobility=5 and selfcare=1 and activity=5 and pain=2 and anxiety=3) then EQindex = 0.073;
if (mobility=5 and selfcare=1 and activity=5 and pain=2 and anxiety=4) then EQindex = -0.009;
if (mobility=5 and selfcare=1 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.093;
if (mobility=5 and selfcare=1 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.119;
if (mobility=5 and selfcare=1 and activity=5 and pain=3 and anxiety=2) then EQindex = 0.063;
if (mobility=5 and selfcare=1 and activity=5 and pain=3 and anxiety=3) then EQindex = 0.048;
if (mobility=5 and selfcare=1 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.033;
if (mobility=5 and selfcare=1 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.117;
if (mobility=5 and selfcare=1 and activity=5 and pain=4 and anxiety=1) then EQindex = 0.014;
if (mobility=5 and selfcare=1 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.042;
if (mobility=5 and selfcare=1 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.057;
if (mobility=5 and selfcare=1 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.138;
if (mobility=5 and selfcare=1 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.222;
if (mobility=5 and selfcare=1 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.144;
if (mobility=5 and selfcare=1 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.200;
if (mobility=5 and selfcare=1 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.215;
if (mobility=5 and selfcare=1 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.296;
if (mobility=5 and selfcare=1 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.380;
if (mobility=5 and selfcare=2 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.249;
if (mobility=5 and selfcare=2 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.193;
if (mobility=5 and selfcare=2 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.178;
if (mobility=5 and selfcare=2 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.097;
if (mobility=5 and selfcare=2 and activity=1 and pain=1 and anxiety=5) then EQindex = 0.013;
if (mobility=5 and selfcare=2 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.151;
if (mobility=5 and selfcare=2 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.095;
if (mobility=5 and selfcare=2 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.080;
if (mobility=5 and selfcare=2 and activity=1 and pain=2 and anxiety=4) then EQindex = -0.001;
if (mobility=5 and selfcare=2 and activity=1 and pain=2 and anxiety=5) then EQindex = -0.085;
if (mobility=5 and selfcare=2 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.126;
if (mobility=5 and selfcare=2 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.070;
if (mobility=5 and selfcare=2 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.055;
if (mobility=5 and selfcare=2 and activity=1 and pain=3 and anxiety=4) then EQindex = -0.026;
if (mobility=5 and selfcare=2 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.110;
if (mobility=5 and selfcare=2 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.021;
if (mobility=5 and selfcare=2 and activity=1 and pain=4 and anxiety=2) then EQindex = -0.035;
if (mobility=5 and selfcare=2 and activity=1 and pain=4 and anxiety=3) then EQindex = -0.050;
if (mobility=5 and selfcare=2 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.131;
if (mobility=5 and selfcare=2 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.215;
if (mobility=5 and selfcare=2 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.137;
if (mobility=5 and selfcare=2 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.193;
if (mobility=5 and selfcare=2 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.208;
if (mobility=5 and selfcare=2 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.289;
if (mobility=5 and selfcare=2 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.373;
```

```
if (mobility=5 and selfcare=2 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.221;
if (mobility=5 and selfcare=2 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.164;
if (mobility=5 and selfcare=2 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.150;
if (mobility=5 and selfcare=2 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.069;
if (mobility=5 and selfcare=2 and activity=2 and pain=1 and anxiety=5) then EQindex = -0.016;
if (mobility=5 and selfcare=2 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.122;
if (mobility=5 and selfcare=2 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.066;
if (mobility=5 and selfcare=2 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.051;
if (mobility=5 and selfcare=2 and activity=2 and pain=2 and anxiety=4) then EQindex = -0.030;
if (mobility=5 and selfcare=2 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.114;
if (mobility=5 and selfcare=2 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.098;
if (mobility=5 and selfcare=2 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.041;
if (mobility=5 and selfcare=2 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.027;
if (mobility=5 and selfcare=2 and activity=2 and pain=3 and anxiety=4) then EQindex = -0.054;
if (mobility=5 and selfcare=2 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.139;
if (mobility=5 and selfcare=2 and activity=2 and pain=4 and anxiety=1) then EQindex = -0.008;
if (mobility=5 and selfcare=2 and activity=2 and pain=4 and anxiety=2) then EQindex = -0.064;
if (mobility=5 and selfcare=2 and activity=2 and pain=4 and anxiety=3) then EQindex = -0.079;
if (mobility=5 and selfcare=2 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.160;
if (mobility=5 and selfcare=2 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.244;
if (mobility=5 and selfcare=2 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.166;
if (mobility=5 and selfcare=2 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.222;
if (mobility=5 and selfcare=2 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.237;
if (mobility=5 and selfcare=2 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.317;
if (mobility=5 and selfcare=2 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.402;
if (mobility=5 and selfcare=2 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.213;
if (mobility=5 and selfcare=2 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.157;
if (mobility=5 and selfcare=2 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.142;
if (mobility=5 and selfcare=2 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.061;
if (mobility=5 and selfcare=2 and activity=3 and pain=1 and anxiety=5) then EQindex = -0.023;
if (mobility=5 and selfcare=2 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.115;
if (mobility=5 and selfcare=2 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.059;
if (mobility=5 and selfcare=2 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.044;
if (mobility=5 and selfcare=2 and activity=3 and pain=2 and anxiety=4) then EQindex = -0.037;
if (mobility=5 and selfcare=2 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.121;
if (mobility=5 and selfcare=2 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.090;
if (mobility=5 and selfcare=2 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.034;
if (mobility=5 and selfcare=2 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.019;
if (mobility=5 and selfcare=2 and activity=3 and pain=3 and anxiety=4) then EQindex = -0.062;
if (mobility=5 and selfcare=2 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.146;
if (mobility=5 and selfcare=2 and activity=3 and pain=4 and anxiety=1) then EQindex = -0.015;
if (mobility=5 and selfcare=2 and activity=3 and pain=4 and anxiety=2) then EQindex = -0.071;
if (mobility=5 and selfcare=2 and activity=3 and pain=4 and anxiety=3) then EQindex = -0.086;
if (mobility=5 and selfcare=2 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.167;
if (mobility=5 and selfcare=2 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.251;
if (mobility=5 and selfcare=2 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.173;
```

```
if (mobility=5 and selfcare=2 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.229;
if (mobility=5 and selfcare=2 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.244;
if (mobility=5 and selfcare=2 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.325;
if (mobility=5 and selfcare=2 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.409;
if (mobility=5 and selfcare=2 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.194;
if (mobility=5 and selfcare=2 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.138;
if (mobility=5 and selfcare=2 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.123;
if (mobility=5 and selfcare=2 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.042;
if (mobility=5 and selfcare=2 and activity=4 and pain=1 and anxiety=5) then EQindex = -0.042;
if (mobility=5 and selfcare=2 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.096;
if (mobility=5 and selfcare=2 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.040;
if (mobility=5 and selfcare=2 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.025;
if (mobility=5 and selfcare=2 and activity=4 and pain=2 and anxiety=4) then EQindex = -0.056;
if (mobility=5 and selfcare=2 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.140;
if (mobility=5 and selfcare=2 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.071;
if (mobility=5 and selfcare=2 and activity=4 and pain=3 and anxiety=2) then EQindex = 0.015;
if (mobility=5 and selfcare=2 and activity=4 and pain=3 and anxiety=3) then EQindex = 0.000;
if (mobility=5 and selfcare=2 and activity=4 and pain=3 and anxiety=4) then EQindex = -0.081;
if (mobility=5 and selfcare=2 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.165;
if (mobility=5 and selfcare=2 and activity=4 and pain=4 and anxiety=1) then EQindex = -0.034;
if (mobility=5 and selfcare=2 and activity=4 and pain=4 and anxiety=2) then EQindex = -0.090;
if (mobility=5 and selfcare=2 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.105;
if (mobility=5 and selfcare=2 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.186;
if (mobility=5 and selfcare=2 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.270;
if (mobility=5 and selfcare=2 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.192;
if (mobility=5 and selfcare=2 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.248;
if (mobility=5 and selfcare=2 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.263;
if (mobility=5 and selfcare=2 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.344;
if (mobility=5 and selfcare=2 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.428;
if (mobility=5 and selfcare=2 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.155;
if (mobility=5 and selfcare=2 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.099;
if (mobility=5 and selfcare=2 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.084;
if (mobility=5 and selfcare=2 and activity=5 and pain=1 and anxiety=4) then EQindex = 0.003;
if (mobility=5 and selfcare=2 and activity=5 and pain=1 and anxiety=5) then EQindex = -0.081;
if (mobility=5 and selfcare=2 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.057;
if (mobility=5 and selfcare=2 and activity=5 and pain=2 and anxiety=2) then EQindex = 0.001;
if (mobility=5 and selfcare=2 and activity=5 and pain=2 and anxiety=3) then EQindex = -0.014;
if (mobility=5 and selfcare=2 and activity=5 and pain=2 and anxiety=4) then EQindex = -0.095;
if (mobility=5 and selfcare=2 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.179;
if (mobility=5 and selfcare=2 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.032;
if (mobility=5 and selfcare=2 and activity=5 and pain=3 and anxiety=2) then EQindex = -0.024;
if (mobility=5 and selfcare=2 and activity=5 and pain=3 and anxiety=3) then EQindex = -0.039;
if (mobility=5 and selfcare=2 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.120;
if (mobility=5 and selfcare=2 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.204;
if (mobility=5 and selfcare=2 and activity=5 and pain=4 and anxiety=1) then EQindex = -0.073;
if (mobility=5 and selfcare=2 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.129;
```

```
if (mobility=5 and selfcare=2 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.144;
if (mobility=5 and selfcare=2 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.225;
if (mobility=5 and selfcare=2 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.309;
if (mobility=5 and selfcare=2 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.231;
if (mobility=5 and selfcare=2 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.287;
if (mobility=5 and selfcare=2 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.302;
if (mobility=5 and selfcare=2 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.383;
if (mobility=5 and selfcare=2 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.467;
if (mobility=5 and selfcare=3 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.232;
if (mobility=5 and selfcare=3 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.176;
if (mobility=5 and selfcare=3 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.161;
if (mobility=5 and selfcare=3 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.080;
if (mobility=5 and selfcare=3 and activity=1 and pain=1 and anxiety=5) then EQindex = -0.004;
if (mobility=5 and selfcare=3 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.134;
if (mobility=5 and selfcare=3 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.077;
if (mobility=5 and selfcare=3 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.063;
if (mobility=5 and selfcare=3 and activity=1 and pain=2 and anxiety=4) then EQindex = -0.019;
if (mobility=5 and selfcare=3 and activity=1 and pain=2 and anxiety=5) then EQindex = -0.103;
if (mobility=5 and selfcare=3 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.109;
if (mobility=5 and selfcare=3 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.053;
if (mobility=5 and selfcare=3 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.038;
if (mobility=5 and selfcare=3 and activity=1 and pain=3 and anxiety=4) then EQindex = -0.043;
if (mobility=5 and selfcare=3 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.127;
if (mobility=5 and selfcare=3 and activity=1 and pain=4 and anxiety=1) then EQindex = 0.004;
if (mobility=5 and selfcare=3 and activity=1 and pain=4 and anxiety=2) then EQindex = -0.052;
if (mobility=5 and selfcare=3 and activity=1 and pain=4 and anxiety=3) then EQindex = -0.067;
if (mobility=5 and selfcare=3 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.148;
if (mobility=5 and selfcare=3 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.232;
if (mobility=5 and selfcare=3 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.154;
if (mobility=5 and selfcare=3 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.210;
if (mobility=5 and selfcare=3 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.225;
if (mobility=5 and selfcare=3 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.306;
if (mobility=5 and selfcare=3 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.390;
if (mobility=5 and selfcare=3 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.203;
if (mobility=5 and selfcare=3 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.147;
if (mobility=5 and selfcare=3 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.132;
if (mobility=5 and selfcare=3 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.051;
if (mobility=5 and selfcare=3 and activity=2 and pain=1 and anxiety=5) then EQindex = -0.033;
if (mobility=5 and selfcare=3 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.105;
if (mobility=5 and selfcare=3 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.048;
if (mobility=5 and selfcare=3 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.034;
if (mobility=5 and selfcare=3 and activity=2 and pain=2 and anxiety=4) then EQindex = -0.047;
if (mobility=5 and selfcare=3 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.131;
if (mobility=5 and selfcare=3 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.080;
if (mobility=5 and selfcare=3 and activity=2 and pain=3 and anxiety=2) then EQindex = 0.024;
if (mobility=5 and selfcare=3 and activity=2 and pain=3 and anxiety=3) then EQindex = 0.009;
```

```
if (mobility=5 and selfcare=3 and activity=2 and pain=3 and anxiety=4) then EQindex = -0.072;
if (mobility=5 and selfcare=3 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.156;
if (mobility=5 and selfcare=3 and activity=2 and pain=4 and anxiety=1) then EQindex = -0.025;
if (mobility=5 and selfcare=3 and activity=2 and pain=4 and anxiety=2) then EQindex = -0.081;
if (mobility=5 and selfcare=3 and activity=2 and pain=4 and anxiety=3) then EQindex = -0.096;
if (mobility=5 and selfcare=3 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.177;
if (mobility=5 and selfcare=3 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.261;
if (mobility=5 and selfcare=3 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.183;
if (mobility=5 and selfcare=3 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.239;
if (mobility=5 and selfcare=3 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.254;
if (mobility=5 and selfcare=3 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.335;
if (mobility=5 and selfcare=3 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.419;
if (mobility=5 and selfcare=3 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.196;
if (mobility=5 and selfcare=3 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.140;
if (mobility=5 and selfcare=3 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.125;
if (mobility=5 and selfcare=3 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.044;
if (mobility=5 and selfcare=3 and activity=3 and pain=1 and anxiety=5) then EQindex = -0.040;
if (mobility=5 and selfcare=3 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.098;
if (mobility=5 and selfcare=3 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.041;
if (mobility=5 and selfcare=3 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.027;
if (mobility=5 and selfcare=3 and activity=3 and pain=2 and anxiety=4) then EQindex = -0.055;
if (mobility=5 and selfcare=3 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.139;
if (mobility=5 and selfcare=3 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.073;
if (mobility=5 and selfcare=3 and activity=3 and pain=3 and anxiety=2) then EQindex = 0.017;
if (mobility=5 and selfcare=3 and activity=3 and pain=3 and anxiety=3) then EQindex = 0.002;
if (mobility=5 and selfcare=3 and activity=3 and pain=3 and anxiety=4) then EQindex = -0.079;
if (mobility=5 and selfcare=3 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.163;
if (mobility=5 and selfcare=3 and activity=3 and pain=4 and anxiety=1) then EQindex = -0.032;
if (mobility=5 and selfcare=3 and activity=3 and pain=4 and anxiety=2) then EQindex = -0.088;
if (mobility=5 and selfcare=3 and activity=3 and pain=4 and anxiety=3) then EQindex = -0.103;
if (mobility=5 and selfcare=3 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.184;
if (mobility=5 and selfcare=3 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.268;
if (mobility=5 and selfcare=3 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.190;
if (mobility=5 and selfcare=3 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.246;
if (mobility=5 and selfcare=3 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.261;
if (mobility=5 and selfcare=3 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.342;
if (mobility=5 and selfcare=3 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.426;
if (mobility=5 and selfcare=3 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.177;
if (mobility=5 and selfcare=3 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.121;
if (mobility=5 and selfcare=3 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.106;
if (mobility=5 and selfcare=3 and activity=4 and pain=1 and anxiety=4) then EQindex = 0.025;
if (mobility=5 and selfcare=3 and activity=4 and pain=1 and anxiety=5) then EQindex = -0.059;
if (mobility=5 and selfcare=3 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.078;
if (mobility=5 and selfcare=3 and activity=4 and pain=2 and anxiety=2) then EQindex = 0.022;
if (mobility=5 and selfcare=3 and activity=4 and pain=2 and anxiety=3) then EQindex = 0.007;
if (mobility=5 and selfcare=3 and activity=4 and pain=2 and anxiety=4) then EQindex = -0.074;
```

```
if (mobility=5 and selfcare=3 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.158;
if (mobility=5 and selfcare=3 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.054;
if (mobility=5 and selfcare=3 and activity=4 and pain=3 and anxiety=2) then EQindex = -0.002;
if (mobility=5 and selfcare=3 and activity=4 and pain=3 and anxiety=3) then EQindex = -0.017;
if (mobility=5 and selfcare=3 and activity=4 and pain=3 and anxiety=4) then EQindex = -0.098;
if (mobility=5 and selfcare=3 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.182;
if (mobility=5 and selfcare=3 and activity=4 and pain=4 and anxiety=1) then EQindex = -0.051;
if (mobility=5 and selfcare=3 and activity=4 and pain=4 and anxiety=2) then EQindex = -0.107;
if (mobility=5 and selfcare=3 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.122;
if (mobility=5 and selfcare=3 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.203;
if (mobility=5 and selfcare=3 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.287;
if (mobility=5 and selfcare=3 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.209;
if (mobility=5 and selfcare=3 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.265;
if (mobility=5 and selfcare=3 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.280;
if (mobility=5 and selfcare=3 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.361;
if (mobility=5 and selfcare=3 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.445;
if (mobility=5 and selfcare=3 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.138;
if (mobility=5 and selfcare=3 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.082;
if (mobility=5 and selfcare=3 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.067;
if (mobility=5 and selfcare=3 and activity=5 and pain=1 and anxiety=4) then EQindex = -0.014;
if (mobility=5 and selfcare=3 and activity=5 and pain=1 and anxiety=5) then EQindex = -0.098;
if (mobility=5 and selfcare=3 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.040;
if (mobility=5 and selfcare=3 and activity=5 and pain=2 and anxiety=2) then EQindex = -0.017;
if (mobility=5 and selfcare=3 and activity=5 and pain=2 and anxiety=3) then EQindex = -0.032;
if (mobility=5 and selfcare=3 and activity=5 and pain=2 and anxiety=4) then EQindex = -0.113;
if (mobility=5 and selfcare=3 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.197;
if (mobility=5 and selfcare=3 and activity=5 and pain=3 and anxiety=1) then EQindex = 0.015;
if (mobility=5 and selfcare=3 and activity=5 and pain=3 and anxiety=2) then EQindex = -0.041;
if (mobility=5 and selfcare=3 and activity=5 and pain=3 and anxiety=3) then EQindex = -0.056;
if (mobility=5 and selfcare=3 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.137;
if (mobility=5 and selfcare=3 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.221;
if (mobility=5 and selfcare=3 and activity=5 and pain=4 and anxiety=1) then EQindex = -0.090;
if (mobility=5 and selfcare=3 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.146;
if (mobility=5 and selfcare=3 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.161;
if (mobility=5 and selfcare=3 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.242;
if (mobility=5 and selfcare=3 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.326;
if (mobility=5 and selfcare=3 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.248;
if (mobility=5 and selfcare=3 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.304;
if (mobility=5 and selfcare=3 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.319;
if (mobility=5 and selfcare=3 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.400;
if (mobility=5 and selfcare=3 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.484;
if (mobility=5 and selfcare=4 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.205;
if (mobility=5 and selfcare=4 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.149;
if (mobility=5 and selfcare=4 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.134;
if (mobility=5 and selfcare=4 and activity=1 and pain=1 and anxiety=4) then EQindex = 0.053;
if (mobility=5 and selfcare=4 and activity=1 and pain=1 and anxiety=5) then EQindex = -0.031;
```

```
if (mobility=5 and selfcare=4 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.107;
if (mobility=5 and selfcare=4 and activity=1 and pain=2 and anxiety=2) then EQindex = 0.050;
if (mobility=5 and selfcare=4 and activity=1 and pain=2 and anxiety=3) then EQindex = 0.036;
if (mobility=5 and selfcare=4 and activity=1 and pain=2 and anxiety=4) then EQindex = -0.045;
if (mobility=5 and selfcare=4 and activity=1 and pain=2 and anxiety=5) then EQindex = -0.129;
if (mobility=5 and selfcare=4 and activity=1 and pain=3 and anxiety=1) then EQindex = 0.082;
if (mobility=5 and selfcare=4 and activity=1 and pain=3 and anxiety=2) then EQindex = 0.026;
if (mobility=5 and selfcare=4 and activity=1 and pain=3 and anxiety=3) then EQindex = 0.011;
if (mobility=5 and selfcare=4 and activity=1 and pain=3 and anxiety=4) then EQindex = -0.070;
if (mobility=5 and selfcare=4 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.154;
if (mobility=5 and selfcare=4 and activity=1 and pain=4 and anxiety=1) then EQindex = -0.023;
if (mobility=5 and selfcare=4 and activity=1 and pain=4 and anxiety=2) then EQindex = -0.079;
if (mobility=5 and selfcare=4 and activity=1 and pain=4 and anxiety=3) then EQindex = -0.094;
if (mobility=5 and selfcare=4 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.175;
if (mobility=5 and selfcare=4 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.259;
if (mobility=5 and selfcare=4 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.181;
if (mobility=5 and selfcare=4 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.237;
if (mobility=5 and selfcare=4 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.252;
if (mobility=5 and selfcare=4 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.333;
if (mobility=5 and selfcare=4 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.417;
if (mobility=5 and selfcare=4 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.176;
if (mobility=5 and selfcare=4 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.120;
if (mobility=5 and selfcare=4 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.105;
if (mobility=5 and selfcare=4 and activity=2 and pain=1 and anxiety=4) then EQindex = 0.024;
if (mobility=5 and selfcare=4 and activity=2 and pain=1 and anxiety=5) then EQindex = -0.060;
if (mobility=5 and selfcare=4 and activity=2 and pain=2 and anxiety=1) then EQindex = 0.078;
if (mobility=5 and selfcare=4 and activity=2 and pain=2 and anxiety=2) then EQindex = 0.022;
if (mobility=5 and selfcare=4 and activity=2 and pain=2 and anxiety=3) then EQindex = 0.007;
if (mobility=5 and selfcare=4 and activity=2 and pain=2 and anxiety=4) then EQindex = -0.074;
if (mobility=5 and selfcare=4 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.158;
if (mobility=5 and selfcare=4 and activity=2 and pain=3 and anxiety=1) then EQindex = 0.053;
if (mobility=5 and selfcare=4 and activity=2 and pain=3 and anxiety=2) then EQindex = -0.003;
if (mobility=5 and selfcare=4 and activity=2 and pain=3 and anxiety=3) then EQindex = -0.018;
if (mobility=5 and selfcare=4 and activity=2 and pain=3 and anxiety=4) then EQindex = -0.099;
if (mobility=5 and selfcare=4 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.183;
if (mobility=5 and selfcare=4 and activity=2 and pain=4 and anxiety=1) then EQindex = -0.052;
if (mobility=5 and selfcare=4 and activity=2 and pain=4 and anxiety=2) then EQindex = -0.108;
if (mobility=5 and selfcare=4 and activity=2 and pain=4 and anxiety=3) then EQindex = -0.123;
if (mobility=5 and selfcare=4 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.204;
if (mobility=5 and selfcare=4 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.288;
if (mobility=5 and selfcare=4 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.210;
if (mobility=5 and selfcare=4 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.266;
if (mobility=5 and selfcare=4 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.281;
if (mobility=5 and selfcare=4 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.362;
if (mobility=5 and selfcare=4 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.446;
if (mobility=5 and selfcare=4 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.169;
```

```
if (mobility=5 and selfcare=4 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.113;
if (mobility=5 and selfcare=4 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.098;
if (mobility=5 and selfcare=4 and activity=3 and pain=1 and anxiety=4) then EQindex = 0.017;
if (mobility=5 and selfcare=4 and activity=3 and pain=1 and anxiety=5) then EQindex = -0.067;
if (mobility=5 and selfcare=4 and activity=3 and pain=2 and anxiety=1) then EQindex = 0.071;
if (mobility=5 and selfcare=4 and activity=3 and pain=2 and anxiety=2) then EQindex = 0.014;
if (mobility=5 and selfcare=4 and activity=3 and pain=2 and anxiety=3) then EQindex = 0.000;
if (mobility=5 and selfcare=4 and activity=3 and pain=2 and anxiety=4) then EQindex = -0.081;
if (mobility=5 and selfcare=4 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.165;
if (mobility=5 and selfcare=4 and activity=3 and pain=3 and anxiety=1) then EQindex = 0.046;
if (mobility=5 and selfcare=4 and activity=3 and pain=3 and anxiety=2) then EQindex = -0.010;
if (mobility=5 and selfcare=4 and activity=3 and pain=3 and anxiety=3) then EQindex = -0.025;
if (mobility=5 and selfcare=4 and activity=3 and pain=3 and anxiety=4) then EQindex = -0.106;
if (mobility=5 and selfcare=4 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.190;
if (mobility=5 and selfcare=4 and activity=3 and pain=4 and anxiety=1) then EQindex = -0.059;
if (mobility=5 and selfcare=4 and activity=3 and pain=4 and anxiety=2) then EQindex = -0.115;
if (mobility=5 and selfcare=4 and activity=3 and pain=4 and anxiety=3) then EQindex = -0.130;
if (mobility=5 and selfcare=4 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.211;
if (mobility=5 and selfcare=4 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.295;
if (mobility=5 and selfcare=4 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.217;
if (mobility=5 and selfcare=4 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.273;
if (mobility=5 and selfcare=4 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.288;
if (mobility=5 and selfcare=4 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.369;
if (mobility=5 and selfcare=4 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.453;
if (mobility=5 and selfcare=4 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.150;
if (mobility=5 and selfcare=4 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.094;
if (mobility=5 and selfcare=4 and activity=4 and pain=1 and anxiety=3) then EQindex = 0.079;
if (mobility=5 and selfcare=4 and activity=4 and pain=1 and anxiety=4) then EQindex = -0.002;
if (mobility=5 and selfcare=4 and activity=4 and pain=1 and anxiety=5) then EQindex = -0.086;
if (mobility=5 and selfcare=4 and activity=4 and pain=2 and anxiety=1) then EQindex = 0.052;
if (mobility=5 and selfcare=4 and activity=4 and pain=2 and anxiety=2) then EQindex = -0.005;
if (mobility=5 and selfcare=4 and activity=4 and pain=2 and anxiety=3) then EQindex = -0.019;
if (mobility=5 and selfcare=4 and activity=4 and pain=2 and anxiety=4) then EQindex = -0.100;
if (mobility=5 and selfcare=4 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.184;
if (mobility=5 and selfcare=4 and activity=4 and pain=3 and anxiety=1) then EQindex = 0.027;
if (mobility=5 and selfcare=4 and activity=4 and pain=3 and anxiety=2) then EQindex = -0.029;
if (mobility=5 and selfcare=4 and activity=4 and pain=3 and anxiety=3) then EQindex = -0.044;
if (mobility=5 and selfcare=4 and activity=4 and pain=3 and anxiety=4) then EQindex = -0.125;
if (mobility=5 and selfcare=4 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.209;
if (mobility=5 and selfcare=4 and activity=4 and pain=4 and anxiety=1) then EQindex = -0.078;
if (mobility=5 and selfcare=4 and activity=4 and pain=4 and anxiety=2) then EQindex = -0.134;
if (mobility=5 and selfcare=4 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.149;
if (mobility=5 and selfcare=4 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.230;
if (mobility=5 and selfcare=4 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.314;
if (mobility=5 and selfcare=4 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.236;
if (mobility=5 and selfcare=4 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.292;
```

```
if (mobility=5 and selfcare=4 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.307;
if (mobility=5 and selfcare=4 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.388;
if (mobility=5 and selfcare=4 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.472;
if (mobility=5 and selfcare=4 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.111;
if (mobility=5 and selfcare=4 and activity=5 and pain=1 and anxiety=2) then EQindex = 0.055;
if (mobility=5 and selfcare=4 and activity=5 and pain=1 and anxiety=3) then EQindex = 0.040;
if (mobility=5 and selfcare=4 and activity=5 and pain=1 and anxiety=4) then EQindex = -0.041;
if (mobility=5 and selfcare=4 and activity=5 and pain=1 and anxiety=5) then EQindex = -0.125;
if (mobility=5 and selfcare=4 and activity=5 and pain=2 and anxiety=1) then EQindex = 0.013;
if (mobility=5 and selfcare=4 and activity=5 and pain=2 and anxiety=2) then EQindex = -0.044;
if (mobility=5 and selfcare=4 and activity=5 and pain=2 and anxiety=3) then EQindex = -0.058;
if (mobility=5 and selfcare=4 and activity=5 and pain=2 and anxiety=4) then EQindex = -0.139;
if (mobility=5 and selfcare=4 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.223;
if (mobility=5 and selfcare=4 and activity=5 and pain=3 and anxiety=1) then EQindex = -0.012;
if (mobility=5 and selfcare=4 and activity=5 and pain=3 and anxiety=2) then EQindex = -0.068;
if (mobility=5 and selfcare=4 and activity=5 and pain=3 and anxiety=3) then EQindex = -0.083;
if (mobility=5 and selfcare=4 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.164;
if (mobility=5 and selfcare=4 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.248;
if (mobility=5 and selfcare=4 and activity=5 and pain=4 and anxiety=1) then EQindex = -0.117;
if (mobility=5 and selfcare=4 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.173;
if (mobility=5 and selfcare=4 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.188;
if (mobility=5 and selfcare=4 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.269;
if (mobility=5 and selfcare=4 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.353;
if (mobility=5 and selfcare=4 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.275;
if (mobility=5 and selfcare=4 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.331;
if (mobility=5 and selfcare=4 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.346;
if (mobility=5 and selfcare=4 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.427;
if (mobility=5 and selfcare=4 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.511;
if (mobility=5 and selfcare=5 and activity=1 and pain=1 and anxiety=1) then EQindex = 0.122;
if (mobility=5 and selfcare=5 and activity=1 and pain=1 and anxiety=2) then EQindex = 0.066;
if (mobility=5 and selfcare=5 and activity=1 and pain=1 and anxiety=3) then EQindex = 0.051;
if (mobility=5 and selfcare=5 and activity=1 and pain=1 and anxiety=4) then EQindex = -0.030;
if (mobility=5 and selfcare=5 and activity=1 and pain=1 and anxiety=5) then EQindex = -0.114;
if (mobility=5 and selfcare=5 and activity=1 and pain=2 and anxiety=1) then EQindex = 0.024;
if (mobility=5 and selfcare=5 and activity=1 and pain=2 and anxiety=2) then EQindex = -0.033;
if (mobility=5 and selfcare=5 and activity=1 and pain=2 and anxiety=3) then EQindex = -0.048;
if (mobility=5 and selfcare=5 and activity=1 and pain=2 and anxiety=4) then EQindex = -0.129;
if (mobility=5 and selfcare=5 and activity=1 and pain=2 and anxiety=5) then EQindex = -0.213;
if (mobility=5 and selfcare=5 and activity=1 and pain=3 and anxiety=1) then EQindex = -0.001;
if (mobility=5 and selfcare=5 and activity=1 and pain=3 and anxiety=2) then EQindex = -0.057;
if (mobility=5 and selfcare=5 and activity=1 and pain=3 and anxiety=3) then EQindex = -0.072;
if (mobility=5 and selfcare=5 and activity=1 and pain=3 and anxiety=4) then EQindex = -0.153;
if (mobility=5 and selfcare=5 and activity=1 and pain=3 and anxiety=5) then EQindex = -0.237;
if (mobility=5 and selfcare=5 and activity=1 and pain=4 and anxiety=1) then EQindex = -0.106;
if (mobility=5 and selfcare=5 and activity=1 and pain=4 and anxiety=2) then EQindex = -0.162;
if (mobility=5 and selfcare=5 and activity=1 and pain=4 and anxiety=3) then EQindex = -0.177;
```

```
if (mobility=5 and selfcare=5 and activity=1 and pain=4 and anxiety=4) then EQindex = -0.258;
if (mobility=5 and selfcare=5 and activity=1 and pain=4 and anxiety=5) then EQindex = -0.342;
if (mobility=5 and selfcare=5 and activity=1 and pain=5 and anxiety=1) then EQindex = -0.264;
if (mobility=5 and selfcare=5 and activity=1 and pain=5 and anxiety=2) then EQindex = -0.320;
if (mobility=5 and selfcare=5 and activity=1 and pain=5 and anxiety=3) then EQindex = -0.335;
if (mobility=5 and selfcare=5 and activity=1 and pain=5 and anxiety=4) then EQindex = -0.416;
if (mobility=5 and selfcare=5 and activity=1 and pain=5 and anxiety=5) then EQindex = -0.500;
if (mobility=5 and selfcare=5 and activity=2 and pain=1 and anxiety=1) then EQindex = 0.093;
if (mobility=5 and selfcare=5 and activity=2 and pain=1 and anxiety=2) then EQindex = 0.037;
if (mobility=5 and selfcare=5 and activity=2 and pain=1 and anxiety=3) then EQindex = 0.022;
if (mobility=5 and selfcare=5 and activity=2 and pain=1 and anxiety=4) then EQindex = -0.059;
if (mobility=5 and selfcare=5 and activity=2 and pain=1 and anxiety=5) then EQindex = -0.143;
if (mobility=5 and selfcare=5 and activity=2 and pain=2 and anxiety=1) then EQindex = -0.005;
if (mobility=5 and selfcare=5 and activity=2 and pain=2 and anxiety=2) then EQindex = -0.062;
if (mobility=5 and selfcare=5 and activity=2 and pain=2 and anxiety=3) then EQindex = -0.076;
if (mobility=5 and selfcare=5 and activity=2 and pain=2 and anxiety=4) then EQindex = -0.157;
if (mobility=5 and selfcare=5 and activity=2 and pain=2 and anxiety=5) then EQindex = -0.241;
if (mobility=5 and selfcare=5 and activity=2 and pain=3 and anxiety=1) then EQindex = -0.030;
if (mobility=5 and selfcare=5 and activity=2 and pain=3 and anxiety=2) then EQindex = -0.086;
if (mobility=5 and selfcare=5 and activity=2 and pain=3 and anxiety=3) then EQindex = -0.101;
if (mobility=5 and selfcare=5 and activity=2 and pain=3 and anxiety=4) then EQindex = -0.182;
if (mobility=5 and selfcare=5 and activity=2 and pain=3 and anxiety=5) then EQindex = -0.266;
if (mobility=5 and selfcare=5 and activity=2 and pain=4 and anxiety=1) then EQindex = -0.135;
if (mobility=5 and selfcare=5 and activity=2 and pain=4 and anxiety=2) then EQindex = -0.191;
if (mobility=5 and selfcare=5 and activity=2 and pain=4 and anxiety=3) then EQindex = -0.206;
if (mobility=5 and selfcare=5 and activity=2 and pain=4 and anxiety=4) then EQindex = -0.287;
if (mobility=5 and selfcare=5 and activity=2 and pain=4 and anxiety=5) then EQindex = -0.371;
if (mobility=5 and selfcare=5 and activity=2 and pain=5 and anxiety=1) then EQindex = -0.293;
if (mobility=5 and selfcare=5 and activity=2 and pain=5 and anxiety=2) then EQindex = -0.349;
if (mobility=5 and selfcare=5 and activity=2 and pain=5 and anxiety=3) then EQindex = -0.364;
if (mobility=5 and selfcare=5 and activity=2 and pain=5 and anxiety=4) then EQindex = -0.445;
if (mobility=5 and selfcare=5 and activity=2 and pain=5 and anxiety=5) then EQindex = -0.529;
if (mobility=5 and selfcare=5 and activity=3 and pain=1 and anxiety=1) then EQindex = 0.086;
if (mobility=5 and selfcare=5 and activity=3 and pain=1 and anxiety=2) then EQindex = 0.030;
if (mobility=5 and selfcare=5 and activity=3 and pain=1 and anxiety=3) then EQindex = 0.015;
if (mobility=5 and selfcare=5 and activity=3 and pain=1 and anxiety=4) then EQindex = -0.066;
if (mobility=5 and selfcare=5 and activity=3 and pain=1 and anxiety=5) then EQindex = -0.150;
if (mobility=5 and selfcare=5 and activity=3 and pain=2 and anxiety=1) then EQindex = -0.013;
if (mobility=5 and selfcare=5 and activity=3 and pain=2 and anxiety=2) then EQindex = -0.069;
if (mobility=5 and selfcare=5 and activity=3 and pain=2 and anxiety=3) then EQindex = -0.084;
if (mobility=5 and selfcare=5 and activity=3 and pain=2 and anxiety=4) then EQindex = -0.165;
if (mobility=5 and selfcare=5 and activity=3 and pain=2 and anxiety=5) then EQindex = -0.249;
if (mobility=5 and selfcare=5 and activity=3 and pain=3 and anxiety=1) then EQindex = -0.037;
if (mobility=5 and selfcare=5 and activity=3 and pain=3 and anxiety=2) then EQindex = -0.093;
if (mobility=5 and selfcare=5 and activity=3 and pain=3 and anxiety=3) then EQindex = -0.108;
if (mobility=5 and selfcare=5 and activity=3 and pain=3 and anxiety=4) then EQindex = -0.189;
```

```
if (mobility=5 and selfcare=5 and activity=3 and pain=3 and anxiety=5) then EQindex = -0.273;
if (mobility=5 and selfcare=5 and activity=3 and pain=4 and anxiety=1) then EQindex = -0.142;
if (mobility=5 and selfcare=5 and activity=3 and pain=4 and anxiety=2) then EQindex = -0.198;
if (mobility=5 and selfcare=5 and activity=3 and pain=4 and anxiety=3) then EQindex = -0.213;
if (mobility=5 and selfcare=5 and activity=3 and pain=4 and anxiety=4) then EQindex = -0.294;
if (mobility=5 and selfcare=5 and activity=3 and pain=4 and anxiety=5) then EQindex = -0.378;
if (mobility=5 and selfcare=5 and activity=3 and pain=5 and anxiety=1) then EQindex = -0.300;
if (mobility=5 and selfcare=5 and activity=3 and pain=5 and anxiety=2) then EQindex = -0.356;
if (mobility=5 and selfcare=5 and activity=3 and pain=5 and anxiety=3) then EQindex = -0.371;
if (mobility=5 and selfcare=5 and activity=3 and pain=5 and anxiety=4) then EQindex = -0.452;
if (mobility=5 and selfcare=5 and activity=3 and pain=5 and anxiety=5) then EQindex = -0.536;
if (mobility=5 and selfcare=5 and activity=4 and pain=1 and anxiety=1) then EQindex = 0.067;
if (mobility=5 and selfcare=5 and activity=4 and pain=1 and anxiety=2) then EQindex = 0.011;
if (mobility=5 and selfcare=5 and activity=4 and pain=1 and anxiety=3) then EQindex = -0.004;
if (mobility=5 and selfcare=5 and activity=4 and pain=1 and anxiety=4) then EQindex = -0.085;
if (mobility=5 and selfcare=5 and activity=4 and pain=1 and anxiety=5) then EQindex = -0.169;
if (mobility=5 and selfcare=5 and activity=4 and pain=2 and anxiety=1) then EQindex = -0.032;
if (mobility=5 and selfcare=5 and activity=4 and pain=2 and anxiety=2) then EQindex = -0.088;
if (mobility=5 and selfcare=5 and activity=4 and pain=2 and anxiety=3) then EQindex = -0.103;
if (mobility=5 and selfcare=5 and activity=4 and pain=2 and anxiety=4) then EQindex = -0.184;
if (mobility=5 and selfcare=5 and activity=4 and pain=2 and anxiety=5) then EQindex = -0.268;
if (mobility=5 and selfcare=5 and activity=4 and pain=3 and anxiety=1) then EQindex = -0.056;
if (mobility=5 and selfcare=5 and activity=4 and pain=3 and anxiety=2) then EQindex = -0.112;
if (mobility=5 and selfcare=5 and activity=4 and pain=3 and anxiety=3) then EQindex = -0.127;
if (mobility=5 and selfcare=5 and activity=4 and pain=3 and anxiety=4) then EQindex = -0.208;
if (mobility=5 and selfcare=5 and activity=4 and pain=3 and anxiety=5) then EQindex = -0.292;
if (mobility=5 and selfcare=5 and activity=4 and pain=4 and anxiety=1) then EQindex = -0.161;
if (mobility=5 and selfcare=5 and activity=4 and pain=4 and anxiety=2) then EQindex = -0.217;
if (mobility=5 and selfcare=5 and activity=4 and pain=4 and anxiety=3) then EQindex = -0.232;
if (mobility=5 and selfcare=5 and activity=4 and pain=4 and anxiety=4) then EQindex = -0.313;
if (mobility=5 and selfcare=5 and activity=4 and pain=4 and anxiety=5) then EQindex = -0.397;
if (mobility=5 and selfcare=5 and activity=4 and pain=5 and anxiety=1) then EQindex = -0.319;
if (mobility=5 and selfcare=5 and activity=4 and pain=5 and anxiety=2) then EQindex = -0.375;
if (mobility=5 and selfcare=5 and activity=4 and pain=5 and anxiety=3) then EQindex = -0.390;
if (mobility=5 and selfcare=5 and activity=4 and pain=5 and anxiety=4) then EQindex = -0.471;
if (mobility=5 and selfcare=5 and activity=4 and pain=5 and anxiety=5) then EQindex = -0.555;
if (mobility=5 and selfcare=5 and activity=5 and pain=1 and anxiety=1) then EQindex = 0.028;
if (mobility=5 and selfcare=5 and activity=5 and pain=1 and anxiety=2) then EQindex = -0.028;
if (mobility=5 and selfcare=5 and activity=5 and pain=1 and anxiety=3) then EQindex = -0.043;
if (mobility=5 and selfcare=5 and activity=5 and pain=1 and anxiety=4) then EQindex = -0.124;
if (mobility=5 and selfcare=5 and activity=5 and pain=1 and anxiety=5) then EQindex = -0.208;
if (mobility=5 and selfcare=5 and activity=5 and pain=2 and anxiety=1) then EQindex = -0.071;
if (mobility=5 and selfcare=5 and activity=5 and pain=2 and anxiety=2) then EQindex = -0.127;
if (mobility=5 and selfcare=5 and activity=5 and pain=2 and anxiety=3) then EQindex = -0.142;
if (mobility=5 and selfcare=5 and activity=5 and pain=2 and anxiety=4) then EQindex = -0.223;
if (mobility=5 and selfcare=5 and activity=5 and pain=2 and anxiety=5) then EQindex = -0.307;
```

```
if (mobility=5 and selfcare=5 and activity=5 and pain=3 and anxiety=1) then EQindex = -0.095;
if (mobility=5 and selfcare=5 and activity=5 and pain=3 and anxiety=2) then EQindex = -0.151;
if (mobility=5 and selfcare=5 and activity=5 and pain=3 and anxiety=3) then EQindex = -0.166;
if (mobility=5 and selfcare=5 and activity=5 and pain=3 and anxiety=4) then EQindex = -0.247;
if (mobility=5 and selfcare=5 and activity=5 and pain=3 and anxiety=5) then EQindex = -0.331;
if (mobility=5 and selfcare=5 and activity=5 and pain=4 and anxiety=1) then EQindex = -0.200;
if (mobility=5 and selfcare=5 and activity=5 and pain=4 and anxiety=2) then EQindex = -0.256;
if (mobility=5 and selfcare=5 and activity=5 and pain=4 and anxiety=3) then EQindex = -0.271;
if (mobility=5 and selfcare=5 and activity=5 and pain=4 and anxiety=4) then EQindex = -0.352;
if (mobility=5 and selfcare=5 and activity=5 and pain=4 and anxiety=5) then EQindex = -0.436;
if (mobility=5 and selfcare=5 and activity=5 and pain=5 and anxiety=1) then EQindex = -0.358;
if (mobility=5 and selfcare=5 and activity=5 and pain=5 and anxiety=2) then EQindex = -0.414;
if (mobility=5 and selfcare=5 and activity=5 and pain=5 and anxiety=3) then EQindex = -0.429;
if (mobility=5 and selfcare=5 and activity=5 and pain=5 and anxiety=4) then EQindex = -0.510;
if (mobility=5 and selfcare=5 and activity=5 and pain=5 and anxiety=5) then EQindex = -0.594;
if (mobility = .) or (selfcare = .) or (activity = .) or (pain = .) or (anxiety = .) then EQindex = .;
```

output; run;

# Appendix I Falls Efficacy Scale scoring algorithm



Appendix J Health Related Productivity Questionnaire - scoring algorithm











# Appendix K Analysis procedure for internal data review and interim analysis

### 1. PURPOSE:

This document describes the processes that will be put in place to manage the planning, scope, implementation, reporting and dissemination of the internal blinded data review and Interim analysis by Internal Review Committee (IRC) for ACT14820 study from the time of the first internal data review to database lock for the complete study to protect the integrity of the study.

#### 2. BACKGROUND

### Study design:

ACT14820 is a two-part, multicenter, multiple-country, randomized, double-blinded, placebo-controlled study in early-stage PD patients carrying a GBA mutation.

The study will be divided into 2 consecutive parts.

**Part 1** will be a randomized, double-blinded, placebo-controlled dose escalation study, utilizing a sequential cohort design. Part 1 will allow selection of the dose of GZ/SAR402671 for Part 2. There will be 3 sequential cohorts that will be placebo-controlled:

- Cohort 1: 4 patients on GZ/SAR402671 4 mg and 1 patient on placebo
- Cohort 2: 4 patients on GZ/SAR402671 8 mg and 1 patient on placebo
- Cohort 3: 4 patients on GZ/SAR402671 15 mg and 1 patient on placebo

All patients must complete the first 4 week course of therapy with subsequent data review, demonstrating safety/tolerability before dose escalation to the next higher level can occur. Patients will not escalate to a higher dose during Part 1. No additional dose escalation of GZ/SAR402671 will occur above the highest proposed dose of 15 mg.

In Japan, each cohort will have a 3:1 ratio, and the total sample size will be approximately 12 Japanese patients (including 9 on GZ/SAR402671 and 3 on placebo):

- Japanese Cohort 1: 3 Japanese patients on GZ/SAR402671 4 mg and 1 Japanese patient on placebo
- Japanese Cohort 2: 3 Japanese patients on GZ/SAR402671 8 mg and 1 Japanese patient on placebo
- Japanese Cohort 3: 3 Japanese patients on GZ/SAR402671 15 mg and 1 Japanese patient on placebo

**Part 2** will be a randomized, double-blinded, placebo controlled, 2-arm study. Part 2 will start after the appropriate dose for Part 2 is selected, following the review of data from Part 1 in non-Japanese patients.

### Data reviews and interim analyses:

Different data review and interim analyses will be performed during the conduct of the study:

- #1 Internal blinded safety data review: an internal review committee (IRC) will perform blinded safety data review after the completion of 4 weeks of dosing in all patients from non-Japanese Cohort 1 prior to dosing of the subsequent cohort; the same process will be repeated after the completion of 4 weeks of dosing in all non-Japanese patients in Cohort 2. Review of blinded safety data from Japanese patients in Cohort 1 and Cohort 2 will follow the same process and will be performed separately. Specifically, the internal review committee will review the AE/SAE data and other available individual patient safety data from all the patients in each cohort in a blinded fashion. No additional dose escalations will occur above the highest proposed dose of 15mg. No dose escalation may occur until the last patient in a given cohort has completed 4 weeks of administration of IMP and data have been reviewed by the IRC
- #2 Internal unblinded data review at the end of Part 1 non-Japan: an internal review committee (IRC) will review in an un-blinded fashion the aggregate safety, pharmacodynamics (CSF GL1) and pharmacokinetic data from Part 1 in non-Japanese patients before Part 2 can occur. This committee will also select the dose for Part 2. The analysis and review for non-Japanese patients will be performed when all non-Japanese patients in Part 1 have completed 4 weeks of dosing and will not wait for patients in Japan to complete Part 1 in order to proceed to Part 2
- #3 Internal unblinded data review at the end of Part 1 Japan: an internal review committee will review in a blinded fashion the aggregate safety data from Part 1 in Japan before Part 2 can start in Japan. This committee will also assess PK similarity between Japanese and non-Japanese patients. The analysis and review for Japanese patients will be performed when all Japanese patients in Part 1 have completed 4 weeks of dosing. PK similarity between Japanese and non Japanese will be determined based on PK data available by the time all patients have completed 4 weeks of treatment

The internal review committees for #2 and #3 data reviews are comprised of individuals not directly involved in day to day study operational execution and whose purpose is to review data (such as safety, tolerability, and/or clinical endpoints). Note that since the responsibilities of these committees are different, they may include different individuals from different functions.

To protect the overall integrity of this study, specific steps, as further described, will be taken to maintain the blind of the study to all those involved in the conduct of the study and/or the data review.

### 3. TIMING AND PURPOSE OF DATA REVIEWS AND INTERIM ANALYSES

# 3.1 Internal blinded safety data review (Part 1)

The internal review committee will review blinded TEAE/SAEs and other available individual patient safety data from all the patients in each cohort before dosing to the subsequent cohort can occur.

The blinded safety data review in Part I will occur up to 4 times during the conduct of the study:

- When all patients from non-Japanese Cohort 1 have completed the first 4 week course of therapy
- When all patients from non-Japanese Cohort 2 have completed the first 4 week course of therapy
- When all patients from Japanese Cohort 1 have completed the first 4 week course of therapy
- When all patients from Japanese Cohort 2 have completed the first 4 week course of therapy

Review of the blinded safety data will be conducted by the internal review committee. A decision on the next higher dose will be made jointly by the GSO and CSD and documented in safety data review meeting minutes. In addition, the CSD will send communication to sites that the next cohort may move to dosing of IMP. Should safety concern(s) arise, these will be brought through the standard internal safety governance process for review.

Decisions for Dose Escalation will be based on the following blinded data:

- All fatal or life-threatening AEs
- Any SAE or  $\geq$  CTCAE Grade 3 event considered related to the study drug
- Any other safety-related issues identified by the Sponsor's Medical Monitor (Clinical Study Director) or Global Safety Officer that pose a medical concern
- New or worsening lens opacity or cataract

If at least 2 patients within the same cohort develop the same SAE or AE (≥Grade 3), the treatment blind will be broken for the concerned patients. If 2 patients or more were receiving GZ/SAR402671, dosing within the cohort will be stopped. Otherwise, GZ/SAR402671 administration per protocol will continue as planned after reviewing all data and the internal review committee determine that it is safe to do so.

For safety purposes, the treatment of a specific patient may be unblinded before the next dose level is administered.

Depending on the safety/tolerability profile observed in the dose level Cohort "n" as well as of the safety/tolerability data observed in the dose level Cohort "n-1" if applicable, one of the following decisions will be taken for Cohort "n+1":

- Continuation of dose escalation as scheduled
- Discontinuation of Part 1 of the study

# 3.2 Internal unblinded data review at the end of Part 1 non-Japan

An internal review committee will review safety, pharmacodynamics and pharmacokinetic data from Part 1 before Part 2 can occur. This committee consisting of individuals not associated with ongoing clinical operational execution of the study will also select the dose for Part 2 (this does not apply to Japanese Part 1).

The data review will occur when all patients from non-Japanese Part1 have completed the first 4 week course of therapy.

A decision to proceed to Part 2 will be made by the Internal Review Committee at the end of Part 1 based on the following unblinded data:

- Safety:
  - AEs
  - laboratory results
  - ECG
  - Vital signs
  - Examination (neurological, ophthalmologic, physical)
- Pharmacodynamic:
  - In CSF: GL1.
- Pharmacokinetic:
  - CSF parameters:
    Week 4: Concentration at any time within 2 to 4 hours after administration of GZ/SAR402671
  - Plasma parameters (optional): Ctrough, Cmax, AUC0-24

In Part 2, the GZ/SAR402671 dose will be the highest dose determined to be safe and well tolerated in Part 1. Moreover, CSF exposure must be known. If there is no CSF exposure of GZ/SAR402671 at the highest safe dose, the study will be stopped.

Depending on the above data in the different dose levels, one of the following decisions will be taken (this does not apply to Japanese Part 1):

- Continuation of study to Part 2 with dose GZ/SAR402671 15 mg
- Continuation of study to Part 2 with dose GZ/SAR402671 8 mg
- Continuation of study to Part 2 with dose GZ/SAR402671 4 mg
- Discontinuation of the study.

## 3.3 Internal data review at the end of Part 1 Japan

The internal review committee will review blinded TEAE/SAEs and other available individual patient safety data from all the Japanese patients before Part 2 can start in Japan. This committee will also assess PK similarity between Japanese and non-Japanese patients. The data review will occur when all Japanese patients from Part1 have completed the first 4 week course of therapy.

PK similarity between Japanese and non-Japanese patients will be assessed by an independent unblinded pharmacokineticist:

- Venglustat Plasma PK parameters (Day 1 and week 4) Cmax and AUC0-24 and/or AUC0-48 as applicable will be determined using non compartmental analysis of observed plasma concentrations and nominal time data. The mean (and range) values of these parameters will be compared with the corresponding values obtained previously for Part-1 ROW data
- Venglustat CSF concentrations (mean and range at week 4) will be determined for Japanese patients and compared with the corresponding values obtained previously for Part-1 ROW data

At the end of Japanese Cohort 3, one of the following decisions will be taken:

- Continuation of study to Part 2 in Japan at the dose selected for Part 2 in non-Japanese patients
- Discontinuation of study in Japan

### 4. KEY RESPONSIBILITIES FOR ACT14820 INTERNAL REVIEW COMMITTEES:

Different internal review committees (IRC), comprised of individuals not involved directly in study conduct will be identified for Internal unblinded data review at the end of Part 1 (non-Japan). The ACT14820 IRC will consist of the minimal number of representatives needed from each of the required R&D functions (ie, Clinical, Pharmacovigilance, Biostatistics & Programming, Pharmacokinetics, etc.) to analyze and report the interim data for the ACT14820 study.

These people are all experienced professionals accustomed to operating under a strict measure of confidentiality, and they will not have any further role in the blinded data review or conduct of the ongoing ACT14820 study.

### 5. PROCESS FOR ANALYZING DATA FOR ACT14820

Process for internal blinded safety data review (Part 1)

No statistical analysis will be performed for the purpose of internal blinded data review. The data review will be based on blinded individual patient data (eg. patient profiles and any available

CIOMs). The conclusion and decision of the blinded safety data review will be documented in the meeting minutes and through notification to sites that administration of IMP at the next dosing level may occur.

Process for internal unblinded data review at the end of Part 1 non-Japan (when all non-Japanese patients from Part 1 have completed 4 weeks of dosing)

A Statistical Analysis Plan (SAP) for Part 1 will be prepared by the ACT14820 study statistician prior to the soft data base lock for Internal data review at the end of Part 1. This SAP will detail all the statistical analyses planned for the interim and final analysis of Part 1 of the study. This SAP will be approved before the internal data review of Part 1 data is performed.

Two reports including descriptive statistical tables, listings, graphs and text summary when applicable will be prepared by the statistician and programmer in the IRC (for safety and pharmacodynamics data listed in Section 3.2) and by the pharmacokineticist in the IRC (for PK data described in Section 3.2). Both reports will be password protected and sent to the members of the IRC at end of Part 1. The lead of the ACT14820 IRC will combine these two reports and include an overall summary with recommendation regarding the continuation of the study to Part 2, including dose recommendation for Part 2.

The required validated statistical programs for producing safety and pharmacodynamics datasets and report outputs will be prepared by the study statisticians and programmers. Biomarker data containing unblinded results will be sent directly to the independent statisticians and programmers in the ACT14820 IRC team by unblinded teams. Once the snapshot is taken, unblinding randomization list and treatment kit de-codes will be supplied directly to the independent statisticians and programmers in the ACT14820 IRC by the IVRS vendor (Perceptive) and sanofi Randomization Code Administrator. Randomization list, treatment kit de-codes, unblinded analysis data sets and all unblinded outputs will be stored in a secure, restricted electronic location only accessible to the independent statistician and programmer in the IRC, and off-limits to the rest of sanofi and in particular to those individuals involved in the ACT14820 clinical study team.

The ACT14820 clinical study team members will continue to work with the blinded data only; procedures for managing and processing data in the ongoing, blinded trial will be followed according to Sanofi standards and good clinical practice. Data will not be frozen as we do not expect a database lock but a snapshot for internal data review. Data will continue to be added, updated or deleted after the internal data review.

Process for internal data review at the end of Part 1 Japan (when all Japanese patients from Part 1 have completed 4 weeks of dosing)

The safety data review will be based on blinded individual patient data (eg. patient profiles and any available CIOMs).

For PK similarity between Japanes and non-Japanese, a short text summary will be prepared by the independent pharmacokineticist and sent to the IRC to provide information on PK comparison between Japanese and non-Japanese patients (including mean values and/or reporting fold

difference to make sure the blind is maintained). Since only the mean values/fold difference in PK will be described, summary may be shared with other team members as needed.

### 6. PREPARATION AND DISTRIBUTION OF INTERNAL DATA ANALYSIS RESULTS

No formal Key Results Memo (KRM) or Clinical Study Report (CSR) will be prepared.

After the data review at the end of Part 1 (non-Japan), the IRC will prepare the text of the internal data review report or interim analysis report (this does not apply to data review prior to dose escalation). Internal data review report will be a password protected file. The password will be determined by the lead of the ACT14820 IRC.

The results will not be distributed to investigators, patients, ACT14820 clinical study members or others within or external to the organization, thus minimizing any chance of future bias.

No public release of the interim results is anticipated at the time this document is being prepared. However, if the information is considered as material and prompt disclosure is required by law, the company may choose to disclose the topline results and will try the best effort to protect the study integrity.

This procedure will be followed in conjunction with the QSOP -009231 for bioanalysis and pharmacokinetic analysis, "Process of maintaining the blind during bioanalysis and pharmacokinetic analysis for clinical studies within DSAR".